## **Statistical Analysis Plan**

**Study ID:** 208090

**Official Title of Study:** Reporting and Analysis Plan Amendment 1 for A Phase III, randomized, multicenter, open-label, non-inferiority study evaluating the efficacy, safety and tolerability of switching to dolutegravir/lamivudine fixed dose combination in HIV-1 infected adults who are virologically suppressed

**Date of Document:** 29-Sep-2022

#### The GlaxoSmithKline group of companies

| Division | : | Worldwide Development |
|---|---|---|
| Information Type | : | Reporting and Analysis Plan (RAP) |
| Title | : | Reporting and Analysis Plan Amendment 1 for A Phase III, randomized, multicenter, open-label, non-inferiority study evaluating the efficacy, safety and tolerability of switching to dolutegravir/lamivudine fixed dose combination in HIV-1 infected adults who are virologically suppressed |
| <b>Compound Number</b> | : | GSK1349572+GR109714 (GSK3515864) |
| <b>Effective Date</b> | : | Refer to Document Date |

## **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 208090 (SALSA).
- This RAP will be provided to the study team members to convey the content of the 208090 Statistical Analysis Complete (SAC) deliverables for the reporting effort up to Week 52.
- This version of the RAP amendment 1 (to the originally approved RAP dated 03-Nov-2020) is to provide details on the Final End of Study (EOS) analysis.

### RAP Author(s):

| Author | Date |
|---------------------------------------|-------------|
| Lead | |
| PPD | 14-Sep-2022 |
| Associate Statistician, Biostatistics | |

Copyright 2022 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

# RAP Team Review Confirmations (Method: E-mail)

| Reviewer | Date |
|-------------------------------------------------|-------------|
| PPD | 19-Sep-2022 |
| Medicine Development Leader, ViiV | 19-Sep-2022 |
| PPD | 21-Sep-2022 |
| PPD , ViiV | |
| PPD | 16-Sep-2022 |
| Manager, Data Management, GSK | |
| PPD | 20-Sep-2022 |
| Clinical Development Manager, GSK | |
| PPD | 21-Sep-2022 |
| PPD , GSK | |
| PPD | 16-Sep-2022 |
| PPD , GSK | |
| PPD | 20-Sep-2022 |
| , Clinical Development, ViiV | |
| PPD | 20-Sep-2022 |
| Clinical Development Investigator, ViiV | |
| PPD | 19-Sep-2022 |
| , Global Health Outcomes Teams, ViiV | |
| PPD | 21-Sep-2022 |
| Principal Programmer, Clinical Programming, GSK | |
| PPD | 20-Sep-2022 |
| Clinical Development Leader, ViiV | |

# Clinical Statistics & Clinical Programming Line Approvals (Method: Pharma eTMF eSignature)

| Approver | Date |
|---------------------------------------|--------------------|
| Principal Statistician, Biostatistics | 29-Sep-2022 |
| PPD , Clinical Progr | amming 29-Sep-2022 |

The main changes included in RAP Amendment 1 are listed in Section 15.16 Appendix 16 – Final (End of Study) Analysis

## **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| 1. | INTR | ODUCTION | 6 |
| 2. | SLIMI | MARY OF KEY PROTOCOL INFORMATION | 6 |
| ۷. | 2.1. | Changes to the Protocol Defined Statistical Analysis Plan | |
| | 2.1. | Study Objective(s) and Estimand(s) / Endpoint(s) | |
| | 2.3. | Study Objective(s) and Estimand(s) / Endpoint(s) | |
| | 2.4. | Statistical Hypotheses / Statistical Analyses | |
| | 2.4. | Statistical Hypotheses / Statistical Arialyses | 9 |
| 3. | | INED ANALYSES | |
| | 3.1. | Interim Analyses | |
| | 3.2. | Final Analyses | 10 |
| 4. | ANAL | YSIS POPULATIONS | 11 |
| | 4.1. | Protocol Deviations | 12 |
| 5. | CON | SIDERATIONS FOR DATA ANALYSES AND DATA HANDLING VENTIONS | |
| | 5.1. | Study Treatment & Sub-group Display Descriptors | |
| | 5.2. | Baseline Definitions | |
| | 5.3. | Multicentre Studies | |
| | 5.4. | Examination of Covariates, Other Strata and Subgroups | 14 |
| | | 5.4.1. Covariates and Other Strata | |
| | | 5.4.2. Examination of Subgroups | |
| | 5.5.<br>5.6. | Multiple Comparisons and Multiplicity Other Considerations for Data Analyses and Data Handling Conventions | |
| 6. | STUE | DY POPULATION ANALYSES | 19 |
| | 6.1. | Overview of Planned Study Population Analyses | |
| 7. | FFFI( | CACY ANALYSES | 21 |
| • | 7.1. | | |
| | | 7.1.1. Endpoint / Variables | |
| | | 7.1.2. Summary Measure | |
| | | 7.1.3. Population of Interest | |
| | | 7.1.4. Strategy for Intercurrent (Post-Randomization) Events | |
| | | 7.1.5. Statistical Analyses / Methods | |
| | 7.2. | Secondary Efficacy Analyses | |
| | | 7.2.1. Endpoint / Variables | |
| | | 7.2.2. Summary Measure | |
| | | 7.2.3. Population of Interest | |
| | | 7.2.4. Strategy for Intercurrent (Post-Randomization) Events | |
| | | 7.2.5. Statistical Analyses / Methods | |
| | 7.3. | Exploratory Efficacy Analyses | |
| 8. | SVEE | ETY ANALYSES | 30 |
| O. | 8.1. | Adverse Events Analyses | |
| | 8.2. | Adverse Events Analyses | |
| | 8.3. | Clinical Laboratory and Biomarker Analyses | |
| | U.J. | Omnoai Laboratory and Diomainer Alialyses | |

### CONFIDENTIAL

| | | 8.3.1. | Lipid Parameters Analyses | 35 |
|---|---|---|---|---|
| | | 8.3.2. | HOMA-IR and HbA1c Analyses | 37 |
| | | 8.3.3. | Bone Biomarkers Analyses | 39 |
| | | 8.3.4. | Renal Biomarkers Analyses | 40 |
| | | 8.3.5. | Inflammatory Biomarkers Analyses | 41 |
| | 8.4. | Other Sa | fety Analyses | |
| | | 8.4.1. | Weight and BMI Analyses | 45 |
| 9. | OTHE | | TICAL ANALYSES | |
| | 9.1. | | utcomes | |
| | | 9.1.1. | Overview of Planned Analyses | |
| | | 9.1.2. | Planned Health Outcomes Statistical Analyses | 46 |
| | 9.2. | | | 48 |
| | | 9.2.1. | Overview of Planned Analyses | |
| | | 9.2.2. | Planned Virology Statistical Analysis | 48 |
| 10. | PHAR | MACOKIN | IETIC ANALYSES | 50 |
| 11. | POPU | LATION F | PHARMACOKINETIC (POPPK) ANALYSES | 50 |
| 12. | PHAR | MACODY | NAMIC ANALYSES | 50 |
| 40 | DUAD | | IETIO / BUADAA CODYALAMIO ANALYOFO | |
| 13. | PHAR | MACOKIN | IETIC / PHARMACODYNAMIC ANALYSES | 50 |
| 4.4 | DEEE | DENCES | | E4 |
| 14. | KEFEI | KENCES. | | 51 |
| 15 | A DDE | VIDICES | | 52 |
| 15. | 15.1. | | c 1: Protocol Deviation Management and Definitions for Per | 55 |
| | 13.1. | | Population | 54 |
| | | | Exclusions from Per Protocol Population | |
| | 15.2. | | c 2: Schedule of Activities | |
| | 10.2. | | Protocol Defined Schedule of Events | |
| | 15.3. | | 3: Assessment Windows | |
| | 10.0. | | Definitions of Assessment Windows for Analyses | |
| | 15.4. | Annendiy | 4: Study Phases and Emergent Adverse Events | 63 |
| | 10.4. | 15.4.1. | Study Phases | |
| | | 15.4.2. | Combining Treatment Phases and States | |
| | | 15.4.3. | Emergent Flag for Adverse Events | |
| | 15.5. | | c 5: Data Display Standards & Handling Conventions | |
| | | 15.5.1. | Reporting Process | |
| | | 15.5.2. | Reporting Standards | |
| | 15.6. | | c 6: Derived and Transformed Data | |
| | | 15.6.1. | General | |
| | | 15.6.2. | Study Population | |
| | | 15.6.3. | Efficacy | |
| | | 15.6.4. | Safety | |
| | | 15.6.5. | Viral Genotyping and Phenotyping | |
| | | 15.6.6. | Health Outcomes | |
| | | 15.6.7. | Cut-off date for protocol deviations | |
| | | 15.6.8. | eCRF Baseline Third Agent Class Determination | |
| | 15.7. | | 7: Reporting Standards for Missing Data | |
| | | 15.7.1. | Premature Withdrawals | |
| | | 15.7.2. | Handling of Missing Data | |

### CONFIDENTIAL

| 15.8. | Appendix 8: Values of Potential Clinical Importance | .98 |
|---|---|---|
| 15.9. | Appendix 9: Population Pharmacokinetic (PopPK) Analyses | |
| 15.10. | Appendix 10: Time to Event Details | |
| | 15.10.1. TRDF Detailed Steps | 100 |
| | 15.10.2. TRDF Detailed Steps for the Kaplan-Meier plot | 105 |
| | 15.10.3. ERDF Detailed Steps | 801 |
| 15.11. | Appendix 11: Snapshot Algorithm Details | |
| 15.12. | Appendix 12: Modified Snapshot Algorithm Details | 114 |
| 15.13. | Appendix 13: Abbreviations & Trade Marks | 118 |
| | 15.13.1. Abbreviations | 118 |
| | 15.13.2. Trademarks | 119 |
| 15.14. | Appendix 14: Model Checking and Diagnostics for Statistical | |
| | Analyses | 120 |
| | 15.14.1. Statistical Analysis Assumptions | 120 |
| 15.15. | Appendix 15: Test of Homogeneity: Fleiss, Liu & Kelly Method1 | 121 |
| | 15.15.1. Statistical Analysis Method for Test of Homogeneity by | |
| | Fleiss, Liu & Kelly1 | |
| 15.16. | Appendix 16: Final (End of Study) Analysis | 122 |
| | 15.16.1. Study Phases | |
| | 15.16.2. Analysis Populations for the Continuation Phase | 123 |
| | 15.16.3. Study Population1 | 123 |
| | 15.16.4. Efficacy Analysis | 123 |
| | 15.16.5. Safety Analysis | 124 |
| | 15.16.6. Virology Analysis | 124 |
| | 15.16.7. COVID - 19 analysis1 | |
| | 15.16.8. Other Analyses (Health Outcomes) | |
| | 15.16.9. List of Data Displays for End of Study (EOS) Final Report1 | 125 |
| 15.17. | Appendix 17: List of Data Displays1 | |
| | 15.17.1. Data Display Numbering1 | |
| | 15.17.2. Mock Example Shell Referencing | |
| | 15.17.3. Deliverables | |
| | 15.17.4. Study Population Tables1 | |
| | 15.17.5. Study Population Figures1 | |
| | 15.17.6. Efficacy Tables1 | |
| | 15.17.7. Efficacy Figures1 | |
| | 15.17.8. Safety Tables1 | |
| | 15.17.9. Safety Figures1 | |
| | 15.17.10. Virology Tables | 152 |
| | 15.17.11.Pharmacokinetic Tables | |
| | 15.17.12. Pharmacokinetic Figures1 | 153 |
| | 15.17.13. Health Outcomes Tables | |
| | 15.17.14. Health Outcomes Figures | |
| | 15.17.15.ICH Listings | |
| | 15.17.16.Non-ICH Listings | 159 |
| 15.18. | Appendix 18: Example Mock Shells for Data Displays | 166 |

### 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for Protocol 208090. The RAP is based on the following 208090 protocol versions Amendment 04 (05May2020), Amendment 04/CHI-1(20May2020)

## 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

The following changes were made to the agreed upon sections in the protocol [(Dated: 14 NOV 2018)].

| Section # and Name | Description of Change and Rationale |
|---|---|
| Exploratory Objective/Endpoints: Protocol Section 3.0 | Addition of an exploratory objective/endpoints that were not specified in the protocol Section 3.0. Objective: To evaluate the effect of subject characteristics (e.g., demographic factors, Baseline CD4) on antiviral and immunological responses to DTG/3TC compared to CAR |
| | <ul> <li>Endpoints:</li> <li>Proportion of subjects by subgroups with plasma HIV-1 RNA</li> <li>&lt;50 c/mL using the Snapshot algorithm at Weeks 24 and 48</li> <li>Change from Baseline in CD4+ cell counts at Weeks 24 and 48 by patient subgroups</li> </ul> |

# 2.2. Study Objective(s) and Estimand(s) / Endpoint(s)

| Objectives | Estimands / Endpoints |
|---|---|
| Primary | Primary |
| To demonstrate the non-inferior antiviral activity of switching to DTG/3TC FDC once daily compared to continuation of CAR over 48 weeks in virologically suppressed adults living with HIV-1 | Proportion of subjects with plasma HIV-1 RNA ≥50 c/mL) endpoint as per FDA snapshot category at Week 48 using the Snapshot algorithm for the ITT-E population |
| Secondary | Secondary |
| To demonstrate the antiviral activity of switching to DTG/3TC FDC once daily compared to continuation of CAR over 48 weeks | Proportion of subjects with plasma HIV-1 RNA <50 c/mL at Week 48 using the Snapshot algorithm for the ITT-E population |
| To evaluate the antiviral activity of switching to DTG/3TC FDC once daily compared to continuation of CAR over 24 weeks | <ul> <li>Proportion of subjects with plasma HIV-1 RNA ≥50 c/mL) endpoint as per FDA snapshot category at Week 24</li> <li>Proportion of subjects with plasma HIV-1 RNA &lt;50 c/mL at Week 24 using the Snapshot algorithm for the ITT-E population</li> </ul> |

| Objectives | Estimands / Endpoints |
|---|---|
| To evaluate the immune effects of DTG/3TC FDC once daily compared to continuation of CAR To evaluate the safety and tolerability of | <ul> <li>Change from Baseline in CD4+ cell count and in CD4+/CD8+ cell counts ratio at Weeks 24 and 48</li> <li>Incidence of disease progression (HIV-associated conditions, AIDS, and death) through Weeks 24 and 48</li> <li>Incidence and severity of adverse events (AEs) and</li> </ul> |
| DTG/3TC FDC once daily compared to CAR over time | <ul> <li>laboratory abnormalities</li> <li>Proportion of subjects who discontinue treatment due to<br/>AEs</li> </ul> |
| To evaluate the safety and tolerability of DTG/3TC FDC once daily in those with creatinine clearance of between 30-49 mL/min/1.73m² compared to those with a creatinine clearance of ≥50 mL/min/1.73m² | <ul> <li>Incidence and severity of AEs and laboratory abnormalities</li> <li>Proportion of subjects who discontinue treatment due to AEs</li> </ul> |
| To evaluate the effects of DTG/3TC FDC once daily on fasting lipids over time compared to CAR | Change from Baseline in fasting lipids at Weeks 24 and 48 |
| To assess viral resistance in participants meeting Confirmed Virologic Withdrawal (CVW) Criteria | Incidence of observed genotypic and phenotypic resistance to ARVs for participants meeting CVW Criteria |
| To assess health related quality of life for participants treated with DTG/3TC FDC compared to CAR | Change from Baseline in health status using HIV TSQ at Weeks 24 and 48 (or Withdrawal from the study) and SDM at Weeks 24, 48 and every 24 weeks during the continuation phase (or Withdrawal from the study) |
| Tertiary/Exploratory | Tertiary/Exploratory |
| To assess willingness to switch for participants treated with DTG/3TC FDC compared to CAR | Reasons for Willingness to Switch at Day 1 |
| To evaluate renal (in urine and blood),<br>bone (in blood), inflammatory (in blood)<br>biomarkers and insulin resistance in<br>participants treated with DTG/3TC FDC<br>compared to CAR | Change from Baseline in renal, bone and inflammatory biomarkers and homeostasis model of assessment-insulin resistance (HOMA-IR) at Weeks 24 and 48 |
| To evaluate biomarkers of telomerase <sup>a</sup> function in participants treated with DTG/3TC FDC compared to CAR. | Change from baseline in biomarkers of telomerase function at Week 48 |
| <sup>a</sup> Separate RAP and report will be produced for b | piomarkers of telomerase |

## 2.3. Study Design



See study protocol for further details

## 2.4. Statistical Hypotheses / Statistical Analyses

This study is designed to show that the antiviral effect of switching to a simplified two-drug regimen of DTG/3TC FDC once-daily is non-inferior to continuation on CAR.

Non-inferiority in the proportion of subjects with plasma HIV-1 RNA  $\geq$  50 c/mL at Week 48 as measured by using the FDA (Food and Drug Administration) Snapshot algorithm (see Appendix 11), can be concluded if the upper bound of a two-sided 95% confidence interval for the difference in the proportion of subjects with plasma HIV-1 RNA  $\geq$  50 c/mL between the two treatment arms (DTG/3TC - CAR) is less than 5%. If  $r_d$  is the response rate on DTG/3TC and  $r_c$  is the response rate on CAR, then the hypotheses can be written as follows:

H<sub>0</sub>: 
$$r_d - r_c \ge 5\%$$
 H<sub>1</sub>:  $r_d - r_c < 5\%$ 

#### 3. PLANNED ANALYSES

# 3.1. Interim Analyses

An interim analysis will be performed at Week 24. To minimise bias, the results of the Week 24 results will not be shared with subjects and investigators or presented externally until after the last subject completes their Week 48 visit. Please refer to the Blinding Agreement for more details.

The planned analysis at Week 24 will be performed after the completion of the following sequential steps:

- Last subject has completed their visit at Week 24 as defined in the protocol, including any re-test as appropriate.
- All required database cleaning activities have been completed and, final database release and database freeze have been declared by Data Management.
- All criteria for unblinding<sup>1</sup> the randomization codes at Week 24 have been met.

No adjustment for multiplicity will be made as the Week 24 analyses will be secondary, however non-inferiority at Week 24 will be declared if the upper bound of a two-sided 95% confidence interval for the difference in HIV-1 RNA  $\geq$  50 c/mL rates between the two treatment arms is less than 5%<sup>2</sup>.

An IDMC is instituted to ensure external objective medical and/or statistical review of efficacy and safety to protect the ethical interests and well-being of subjects and to protect the scientific validity of the study. An ad-hoc review of data by the IDMC will be triggered whenever the number of confirmed virologic withdrawals (CVWs) exceeds thresholds pre-specified in the IDMC charter. Full details of the methods, timing, decision criteria and operating characteristics are pre-specified in the IDMC Charter. Details of the analyses and outputs provided to the IDMC are detailed in an IDMC RAP.

- 1. Note that analyses for time points will be performed when subjects complete visits relevant to that time point i.e. Week 24 analysis takes place when the last patient has completed their Week 24 visit..
- 2. Please refer to Section 7.1.5.1 for details and conditions for presentation of test for superiority

# 3.2. Final Analyses

The primary analysis is at Week 48. An additional analysis will be performed at the end of the continuation phase .

The planned analyses at Weeks 48 and end of continuation phase<sup>3</sup> will be performed after the completion of the following sequential steps:

- Last subject has completed their relevant visit at week 48 (or end of continuation) as defined in the protocol, including any re-test as appropriate.
- All required database cleaning activities have been completed and final database release and database freeze has been declared by Data Management.

• All criteria for unblinding the randomization codes at Week 48 have been met.

Further data cuts and analyses may be conducted as necessary in support of regulatory submissions and publications.

The Sub-study analyses will be covered by separate RAPs.

3. Note that analyses for time points will be performed when subjects complete visits relevant to that time point i.e. Week 48 analysis takes place when the last patient has completed their Week 48 visit, and not when they have completed their Week 48 and end of continuation phase.

## 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Screened | <ul> <li>Comprises Screened for inclusion in the study, including screen-failures.</li> <li>This population will be based on the treatment to which the subject was randomized. Screen-failures will be categorised as "Non-randomized".</li> </ul> | Study Population |
| Randomized | <ul> <li>The Randomized population will consist of all subjects who are randomized in the study</li> <li>Any subject who receives a treatment randomization number will be considered to have been randomized.</li> </ul> | Study Population |
| Intent-to-Treat<br>(ITT) | <ul> <li>Comprises all randomized subjects</li> <li>Subjects will be assessed according to the treatment to which the subject was randomized regardless of treatment they actually received.</li> <li>Any subject receiving a treatment randomization number will be considered to be randomized.</li> </ul> | Efficacy (sensitivity analyses) |
| Intent-To-Treat<br>Exposed (ITT-E) | <ul> <li>Comprises all randomized subjects who receive at least one dose of study treatment either DTG/3TC or CAR.</li> <li>This population will be based on the treatment to which the subject was randomized.</li> </ul> | Study Population,<br>Efficacy and Health<br>Outcomes |
| Per-Protocol (PP) | <ul> <li>This population will consist of subjects in the ITT-E Population with the exception of significant protocol violators.</li> <li>Protocol deviations that would exclude subjects from the PP population are defined in Section 4.1 (Protocol Deviations) and Appendix 1 (Protocol Deviation Management and Definition for Per-Protocol Population).</li> </ul> | Efficacy (Sensitivity<br>Analysis) |
| CVW | Comprises all subjects in the ITT-E population who have met the derived CVW criteria (see Section 15.6.3) | <ul><li>Genotypic</li><li>Phenotypic</li></ul> |

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| | | Efficacy |
| potential | Comprises subjects in the ITT-E population having | Genotypic |
| Precautionary<br>Virologic<br>Withdrawal<br>(pPVW) | 2 consecutive measurements between 50 and 200 c/mL. The current HIV-1 RNA values <u>must</u> be below 200 c/mL, but the previous HIV-1 RNA can <u>also</u> have been >=200 c/mL | Phenotypic |
| Safety | Comprises all subjects who receive at least one dose of study treatment either DTG/3TC or CAR. | Safety |
| | This population will be based on the treatment the subject actually received <sup>4</sup> . | |

#### 1. NOTES:

- Please refer to Appendix 17: List of Data Displays which details the population to be used for each display being generated.
- 4. As recorded on IVRS. If the randomized treatment is incorrect, the actual treatment will only be recorded in IVRS through sponsor intervention

## 4.1. Protocol Deviations

| Term | Definition |
|---|---|
| Study Deviation Rules Document | The document describing study deviations (and associated coding/naming conventions) that may be identified during a study and the frequency of study deviation reviews. |
| Protocol Deviation<br>(PD) | Any departure from study-specific requirements specified in a protocol. Subsets of protocol deviations are categorized as important or significant. |
| Important Protocol<br>Deviations | A subset of protocol deviations that may significantly impact the completeness, accuracy, and/or reliability of the study data or that may significantly affect a subject's rights, safety, or well-being. All important deviations have a Violation Flag in CTMS and are associated with a Rule Number. |
| Significant Protocol<br>Deviations | Considered a subset of important protocol deviations, typically impacting efficacy assessments, which lead to the exclusion from the per-protocol population. All significant deviations are captured in CTMS and are associated with a Rule Number. |

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management, patient assessment) will be summarised and listed.

Separately, important deviations which result in exclusion from analysis populations and events that results in exclusion from the analysis population will be summarised and listed (see Appendix 1).

The COVID-19 Pandemic has the potential to impact subject visit completion. This may result in PDs being reported which are related to COVID-19 rather than study non-compliance by subjects or sites. As a result, all COVID-19 specific PDs identified using "COVID-19" prefix as defined in the protocol deviations specification document will be summarised and listed.

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Deviation Rule Document.

- O Data will be reviewed prior to unblinding and freezing of the database with the aim of capturing and categorising all important deviations.
- This dataset will be the basis for the summaries and listings of protocol deviations.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

# 5.1. Study Treatment & Sub-group Display Descriptors

| Treatment Group Description | Order [1] |
|-----------------------------|-----------|
| DTG/3TC | 1 |
| CAR | 2 |

#### NOTES:

1. Order represents treatments being presented in TFL, as appropriate.

Treatment comparisons will be displayed as follows using the descriptors as specified:

1. DTG/3TC vs CAR

#### 5.2. Baseline Definitions

For all endpoints (unless otherwise stated) the baseline value will be the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. If time is not collected, Day 1 assessments are assumed to be taken prior to first dose and used as baseline.

Unless otherwise stated, if baseline data are missing no derivation will be performed and baseline will be set to missing.

Unless otherwise specified, the baseline definitions specified in the table below will be used for derivations for endpoints/parameters and indicated on summaries and listings.

| Definition | Reporting Details |
|---|---|
| Change from Baseline | = Post-Dose Visit Value – Baseline |
| % Change from Baseline | = 100 x [(Post-Dose Visit Value – Baseline) / Baseline] |

#### 5.3. Multicentre Studies

Data will be summarised for all centres combined. Country will be included as an exploratory subgroup for analyses of specific endpoints.

# 5.4. Examination of Covariates, Other Strata and Subgroups

#### 5.4.1. Covariates and Other Strata

- Table 1 presents the covariates that may be used in descriptive summaries and statistical analyses, some of which may also be used for subgroup analyses.
- Additional covariates of clinical interest may also be considered.

Table 1 List of Covariates for Descriptive Summaries and Statistical Analyses

| Details | Endpoints | | | | | |
|---|---|---|---|---|---|---|
| | Renal<br>Biomarkers | Bone<br>Biomarkers | Inflammatory<br>Biomarkers | HOMA-IR ,<br>HbA1c | Weight,<br>BMI/Lipids | HO (SDM and HIVTSQ) |
| Randomization is stratified by baseline third agent class: | Υ | Y | Υ | Υ | Υ | Υ |
| Baseline third agent class (PI, INI, NNRTI). for analysis purposes, randomization strata will be derived using eCRF data, even if this differs from the strata captured in IVRS (details of how this is derived can be found in Section 15.6.8) All statistical analyses will adjust for the above randomization strata, unless stated otherwise. Treatment-by-Strata interactions will be assessed as specified in the analysis sections. | | | | | | |
| Age (years): (Continuous) | Υ | Υ | Υ | Υ | Υ | Υ |
| Gender: Male & Female | Υ | Υ | Υ | Υ | Υ | Υ |
| Baseline CD4+ cell count (continuous) | Υ | Υ | Υ | Υ | Υ | |
| Race (White, Black or African American, Asian, Other) | Υ | Υ | Υ | Υ | Υ | Υ |
| BMI (continuous) | Υ | Υ | Υ | Υ | | |
| Smoking status (Never vs. Former vs. Current Smoker) | | Υ | Υ | | | |
| Diabetes mellitus (Yes vs. No) | Y | | | Y (for<br>HbA1c) | | |
| Hypertension (Yes vs. No) | Υ | | | Υ | | |
| HCV-coinfection (Yes vs. No) | | | Υ | | | |
| Baseline value of the endpoint* | Υ | Υ | Υ | Υ | Υ | Υ |

<sup>\*</sup> Baseline value will be continuous, and if the outcome is log-transformed the baseline value will be log-transformed as well

## 5.4.2. Examination of Subgroups

The list of subgroups may be used in descriptive summaries and statistical analyses. Additional subgroups of clinical interest may also be considered.

• If the percentage of subjects is small within a subgroup, then the subgroup categories may be refined prior to unblinding the trial.

If the category cannot be refined further, then descriptive rather than statistical comparisons may be performed for the particular subgroup.

| Subgroups |
|---|
| Randomization is stratified by baseline third agent class: |
| Baseline third agent class (PI, INI, NNRTI). |
| For analysis purposes, randomization strata will be derived using eCRF data, even if this differs from the strata captured in IVRS |
| All statistical analyses will adjust for the above randomization strata, unless stated otherwise. Treatment-by-Strata interactions will be assessed as specified in the analysis sections. |
| <ul> <li>Age (years): <ul> <li>&lt;35, 35 - 49, ≥50, and &lt;50 vs. ≥50</li> <li>&lt;60 and ≥60 may also be performed if specifically required for regulatory purposes</li> </ul> </li> <li>Gender: Male &amp; Female</li> <li>Race: <ul> <li>White, Black or African American, Asian, Other</li> <li>White, Non-White</li> </ul> </li> <li>Country <ul> <li>Baseline CD4+ cell count: <ul> <li>&lt;500, ≥500 cells/mm³</li> </ul> </li> <li>CDC HIV-1 classification <ul> <li>HIV infection stage 0</li> <li>HIV infection stage 1</li> <li>HIV infection stage 2</li> <li>HIV infection stage 3 (AIDS)</li> <li>HIV infection stage unknown</li> <li>Baseline Creatinine Clearance</li></ul></li></ul></li></ul> |

| Subgroup | Subgroups |
|---|---|
| | Baseline concerns with long-term side effects of their current ART (PCLTT): (Yes/No) * |

<sup>\*</sup> Subgroup is for Health outcome analysis. This is derived from Willingness to switch questionnaire with baseline response given as "Concerned about long-term side effects" as the reason for willingness to participate in a clinical study where their current HIV medication may be switched.

Subgroup analyses for endpoints will be presented as shown in the Table 2.

Table 2 List of Subgroup Variables for Descriptive Summaries and Statistical Analyses

| | Endpoint | | | | | |
|---|---|---|---|---|---|---|
| Subgroup | Proportion<br>of patients<br>with<br>plasma<br>HIV-1 RNA<br><50¹ c/mL² | Summary<br>of Study<br>Snapshot<br>outcomes<br>(Plasma<br>HIV-1<br>RNA ≥/<<br>50 c/mL) | CD4+ Cell<br>Count and<br>CD4+/CD8+<br>Ratio<br>Change<br>from<br>Baseline | AEs <sup>3</sup> | Clinical<br>Chemistry,<br>Hematology<br>and Liver<br>Chemistries | HO<br>(SDM<br>and<br>HIVTSQ) |
| Baseline third agent class (PI, INI, NNRTI,) | Y | Y | Y | Y | | Y |
| Age (years): <35, 35 - 49, ≥50 | Y | Y | Υ | Υ | | |
| Age (years): <50, ≥50 | Y | Y | | | | |
| Gender: Male & Female | Y | Y | Y | Υ | | |
| Country | Υ | Υ | | | | |
| Race: White, Black or African<br>American, Asian, Other | Y | Y | Y | Y | | |
| Race: White, non-white | Υ | Y | Υ | | | |
| Baseline CD4+ cell count: <500, ≥500 cells/mm3 | Y | Y | Y | Y | | |
| CDC HIV-1 classification:: HIV infection stage 0, 1, 2, 3 (AIDS), Unknown | Y | Y | Y | Y | | |
| Baseline Creatinine Clearance: 30-49 mL/min/1.73m², ≥50 mL/min/1.73m² | | | | Y | Y | |
| Baseline concerns about long-term side effects of their current HIV regimen (PCLTT): (Yes/No) | | | | | | Y |

<sup>1.</sup> A sensitivity analysis will also be performed for the following endpoint: HIV-1 RNA <40 c/mL and Target Not Detected Status. See Section 7.2.5 for more details.

<sup>2.</sup> Includes forest plot for unadjusted difference of patients with plasma HIV 1 RNA <50 c/mL between treatment arms.

3. Subgroup analyses will be presented for the following analyses: Adverse Events by System Organ Class (see Appendix 17 Full Data Displays for more information)

## 5.5. Multiple Comparisons and Multiplicity

The primary comparison of interest is the comparison between DTG/3TC and CAR for the primary endpoint in the ITT-E population. This analysis will be adjusted for by the actual stratification factor as determined from the eCRF data (not as recorded in IVRS) randomisation.

No adjustment for multiplicity is required as there is only one primary comparison of interest.

# 5.6. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

| Section | Component |
|---|---|
| Section 15.1 | Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population |
| Section 15.2 | Appendix 2: Schedule of Activities |
| Section 15.3 | Appendix 3: Assessment Windows |
| Section 15.4 | Appendix 4: Study Phases and Emergent Adverse Events |
| Section 15.5 | Appendix 5: Data Display Standards & Handling Conventions |
| Section 15.6 | Appendix 6: Derived and Transformed Data |
| Section 15.7 | Appendix 7: Reporting Standards for Missing Data |
| Section 15.8 | Appendix 8: Values of Potential Clinical Importance |
| Section 15.9 | Appendix 9: Population Pharmacokinetic (PopPK) Analyses |
| Section 15.10 | Appendix 10: Time to Event Details |
| Section 15.11 | Appendix 11: Snapshot |
| Section 15.12 | Appendix 12: Modified Snapshot |
| Section 15.13 | Appendix 13: Abbreviations & Trade Marks |
| Section 15.14 | Appendix 14: Model Checking and Diagnostics for Statistical Analyses |
| Section 15.15 | Appendix 15: Test of Homogeneity: Fleiss, Liu & Kelly Method |
| Section 15.16 | Appendix 16: Final (End of Study) analysis |
| Section 15.17 | Appendix 17: List of Data Displays |
| Section 15.18 | Appendix 18: Example Mock Shells for Data Displays |

# 6. STUDY POPULATION ANALYSES

# 6.1. Overview of Planned Study Population Analyses

The study population analyses will be based on the Intent-To-Treat Exposed (ITT-E) population, unless otherwise specified.

Table 3 provides an overview of the planned study population analyses, with full details of data displays being presented in Appendix 17: List of Data Displays.

Table 3 Overview of Planned Study Population Analyses

| Display Type | Data Displa | ys Generated |
|---|---|---|
| | Table | Listing |
| Randomization | | |
| Randomization | | Υ [1] |
| Misrandomized Strata or Treatment | Y | |
| Subject Disposition | | |
| Subjects Enrolled by Country and Site ID [2] | Y | Y |
| Subjects Enrolled by Country and Site ID relative to COVID-19 Pandemic measures | Υ | |
| Country Level Listing of Start Dates of COVID-19 Pandemic Measures | | Y |
| History of Rescreened Subjects [2] | | Y |
| Reasons for Screen Failure [2] | Υ | Y |
| Subject Disposition | Υ [3,4] | |
| Subject Status and Subject Disposition by Relationship to COVID-19 Pandemic | Υ | |
| Treatment Status and Reasons for Discontinuation of Study Treatment by relationship to COVID-19 Pandemic | Υ | |
| Reasons for Withdrawal by Visit | Y | Y |
| Study Visit Dates | | Y |
| Visits Impacted by COVID-19 Pandemic <sup>[11]</sup> | Υ | Y |
| Populations Analysed | | |
| Study Populations [2] | Y | Y |
| Protocol deviations | | |
| Important Protocol Deviations by Relationship to COVID-19 | Υ | Y |
| Deviations leading to exclusion from PP | Υ | Y |
| Inclusion and Exclusion Criteria Deviations | | Υ |

| Display Type | Data Displa | ys Generated |
|---|---|---|
| | Table | Listing |
| Non-Important Protocol Deviation Related to COVID-<br>19 | | Υ |
| Demography and baseline characteristics | | |
| Demographic Characteristics [5] | Υ | Y |
| Summary of Age Ranges | Y | |
| Race & Racial Combinations [6] | Y | Y |
| Hepatitis C Status | Υ | Υ |
| CDC Classification of HIV infection at Baseline | Y | Y |
| HIV Risk Factor | Y | Y |
| Cardiovascular Risk Assessments at Baseline | Y | Y |
| Distribution of CD4+ Cell Counts | Υ | |
| Distribution of HIV-1 RNA (c/mL) | Y | |
| Distribution of CD4+/CD8+ cell count ratio | Y | Y |
| Medical Conditions, Concomitant Medications & Ar | tiretroviral Therapy | |
| Medical Conditions (Current and Past) | Υ | Y |
| Medical Conditions: Sub-conditions (Current/Past) | Y | |
| Concomitant Medications (non-ART) | Υ [7] | Υ [8] |
| Prior and Concomitant ART Medications | Υ | Υ [9] |
| Baseline third agent class (Strata) [10] | Υ | Υ |
| Lipid Modifying agents (Baseline and Post-Baseline) | Υ | |
| Other | | • |
| History of Depression and Anxiety at Baseline | Y | |

#### 1. NOTES:

- Y = Display Generated, T = Tables, L = Listings, IP = Investigational Product
- 1. ITT-E. One listing of subjects randomized but not treated, and one listing of planned and actual treatment strata.
- 2. Screened population.
- 3. Subject Accountability by Phase (Overall, Randomized Phase, Continuation Phase)
- 4. Subjects who have not been recorded as withdrawing from the study in the respective phase will be categorized as "Ongoing at time of the analysis" for summary purposes.
- 5. Age, sex, ethnicity, weight, height, BMI (kg/m^2) and child-bearing potential collected at screening.
- 6. The five high level FDA race categories and designated Asian subcategories will be summarised along with all combinations of high level categories which exist in the data. The nine race categories collected will be summarised along with categories for mixed race. A by-subject listing of race will also be produced.
- 7. Summarised by Ingredient ATC Level 1
- 8. One listing for concomitant non-ART medications and one listing showing the relationship between verbatim text, ingredient and ATC Level 1.
- 9. One listing for Prior ART, one listing for concomitant ART and one listing showing the relationship between verbatim text, ingredient, combination and ATC Level 4.
- 10. Based on the actual third agent class that subjects were classified into according to data captured on the eCRF.
- 11. Visits impacted by COVID-19 Pandemic will also be presented by stacked bar chart

#### 7. EFFICACY ANALYSES

## 7.1. Primary Efficacy Analyses

The primary treatment effect to be estimated will be the effect on the composite virologic outcome at Week 48, using the FDA (Food and Drug Administration) Snapshot algorithm. The variable is the binary response indicating the virologic outcome category of plasma HIV-1 RNA ≥50 copies/mL (c/mL) at Week 48 and the summary measure is the difference in the percent of subjects with plasma HIV-1 RNA ≥50 c/mL at Week 48 between each treatment group. The population is all subjects in the Intent-to-Treat Exposed (ITT-E) population. The individual components of the estimand are detailed as follows.

## 7.1.1. Endpoint / Variables

The primary endpoint is the percent of subjects with plasma HIV-1 RNA ≥50 c/mL at Week 48 using the FDA Snapshot algorithm (see Section 15.11).

The primary endpoint is the binary response indicating the virologic outcome category of plasma HIV-1 RNA  $\geq$ 50 c/mL at Week 48 using the FDA Snapshot algorithm (See Appendix 11). The other Snapshot outcomes (HIV-1 RNA  $\leq$ 50 c/mL and no virologic data at Week 48 Window) will be collapsed into the non-response category.

#### 7.1.2. Summary Measure

Difference in the percent of subjects with plasma HIV-1 RNA  $\geq$ 50 c/mL at Week 48, defined by the FDA snapshot algorithm (see Appendix 11), between each treatment groups (DTG/3TC – CAR).

#### 7.1.3. Population of Interest

The primary efficacy analyses will be based on the Intent-To-Treat Exposed (ITT-E) population (defined in Section 4) unless otherwise specified.

### 7.1.4. Strategy for Intercurrent (Post-Randomization) Events

A treatment policy strategy will be used for intercurrent events such as discontinuations, missing plasma HIV-1 RNA samples and change in background regimen are handled using the Snapshot algorithm (see Section 15.11), which details how to assign each subject's virologic outcome.

#### 7.1.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 17: List of Data Displays and will be based on GSK data standards and statistical principles commonly applied in GSK HIV-1 trials.

Table 4 provides an overview of the planned efficacy analyses, with full details of data displays being presented in Appendix 17: List of Data Displays.

Table 4 Overview of Planned Primary Efficacy Analyses

| | Absolute | | | | | | |
|---|---|---|---|---|---|---|---|
| Endpoint | St | ats Analysi | S | Sum | mary | Individual | |
| | T | F | L | T | F | F | L |
| Percent of Subjects v | vith plasma | a HIV 1 RN | A ≥50 c/m | L at week | 48 – Snaps | hot | |
| Primary Analysis | Υ [1] | | Υ | | | | |
| Sparse Data | Y [2] | | | | | | |
| Analysis | I [2] | | | | | | |

- 1. NOTES:
- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- 2 [1] Generated using the 'Intent-to-Treat Exposed' (primary), 'Per-Protocol' and 'Intent-to-Treat' (sensitivity) populations.
- 3 [2] See methodology section for more information.

### 7.1.5.1. Statistical Methodology Specification

#### **Endpoint**

The binary response indicating the virologic outcome category of plasma HIV 1 RNA ≥50 c/mL at Week 48 using the FDA Snapshot algorithm (see Appendix 11).

#### **Model Specification**

The primary efficacy endpoint will be analysed using a stratified analysis for proportions with Cochran-Mantel-Haenszel (CMH) weights, adjusting for baseline third agent class (PI, INI, NNRTI). The CMH estimate of the adjusted treatment difference will be calculated as a weighted average of strata-specific estimates of the treatment difference calculated within each of the following three Baseline analysis strata:

- Baseline third agent: PI
- Baseline third agent: INI
- Baseline third agent: NNRTI

If  $n_k$  is the number of DTG/3TC treated subjects,  $m_k$  is the number of PI-, INI-, or NNRTI-based ART treated subjects, and  $N_k = n_k + m_k$  is the total number of subjects in the kth stratum, then the CMH estimate is given by:

$$\hat{d}_{cmh} = \frac{\sum W_k \hat{d}_k}{\sum W_k}$$

where,

$$W_k = \frac{n_k m_k}{N_k}$$

are CMH weights and  $d_k$  are estimates of the differences in proportions of subjects with plasma HIV-1 RNA  $\geq$ 50 c/mL between the two treatment arms,  $r_{DTG/3TC}$  - $r_{CAR}$ , for the kth strata.

The corresponding two-sided 95% CI will be calculated as

$$\hat{d}_{cmh} \pm 1.96 \times \sqrt{\hat{\text{var}}(\hat{d}_{cmh})}$$

Where the variance estimator (Sato ,1989) is consistent in both sparse data and large strata and is given below.

$$var(\hat{d}_{cmh}) = \frac{\hat{d}_{cmh}(\sum P_k) + \sum Q_k}{\left(\sum n_k m_k / N_k\right)^2} = \frac{\hat{d}_{cmh}(\sum P_k) + \sum Q_k}{\left(\sum W_k\right)^2}$$

where

$$P_k = \frac{n_k^2 y_k - m_k^2 x_k + n_k m_k (m_k - n_k)/2}{N_k^2}$$

$$Q_k = \frac{x_k (m_k - y_k) / N_k + y_k (n_k - x_k) / N_k}{2}$$

With  $x_k$  and  $y_k$  corresponding to the number of subjects with HIV-1 RNA  $\geq$ 50 c/mL at Week 48 as determined by the FDA Snapshot algorithm (See Appendix 11) for treatment and comparator, respectively, for the  $k^{th}$  stratum.

## **Model Checking & Diagnostics**

Not applicable

#### Model Results Presentation

Adjusted CMH estimate of the difference in the proportion of subjects with plasma HIV-1 RNA ≥ 50 c/mL between each treatment group (DTG/3TC – CAR) and corresponding 95% confidence interval will be presented.

Non-inferiority will be concluded if the upper bound of the two-sided 95% confidence interval (CI) for the CMH adjusted difference in the proportion of patients with plasma HIV-1 RNA  $\geq$  50 c/mL

between each treatment group (DTG/3TC – CAR) is less than 5%. The p-value for non-inferiority based on a non-inferiority margin of 5% will also be presented. 95% confidence intervals for the percent of subjects with virologic failure by treatment group.

If the analysis shows non-inferiority, then a superiority hypothesis will be tested at the two-sided 5% level of significance. Superiority favoring DTG/3TC will be declared if the upper bound of two-sided confidence interval is below 0%. If superiority is declared, the p-value for superiority will also be presented.

### **Subgroup Analyses**

Subgroup analyses will not be performed for this endpoint

#### Sensitivity and Supportive Analyses

- 1. Per-Protocol population analysis:
  - To assess the impact of significant protocol deviations, statistical analysis will be repeated using the Per-protocol population and compared for consistency with the results from the primary ITT-E population analysis. If both analyses show non-inferiority then the hypothesis that the antiviral effect of treatment with DTG/3TC is superior to treatment with CAR will be tested at the two-sided 5% level of significance.
- 2. Intent-to-Treat population analysis:
  - Statistical analysis will be repeated using the Intent-to-Treat population and compared for consistency with the results from the ITT-E and PP populations.
  - In this analysis, subjects randomized but not exposed to study treatment will be classified as "having no virologic data".
- 3. Separate supportive analyses will be performed to enable the assessment of the homogeneity of the treatment difference across strata.
  - The weighted least squares chi-squared statistic of [D'Agostino, 2008,Fleiss, 1981] will be used to test for one-way homogeneity of the treatment difference across the levels of each strata for baseline third agent class (PI, INI, NNRTI), with each categorical variable considered separately. Following Lui and Kelly [Lui, 2000], ½ will be added to each cell in any strata for which the stratum-specific rate estimates of either r<sub>DTG/3TC</sub> or r<sub>CAR</sub> are zero or one, and tests will be one-sided. Tests of homogeneity will be assessed at the one-sided 10% level of significance. For details see Appendix 15.

For each stratum in addition to the proportion of subjects with plasm HIV-1 RNA≥50 c/mL by treatment group and subgroup (with 95% CI type CI) as described in Appendix 15, the p-value from the test of homogeneity will also be reported for each categorical stratification variable.

These results will be used to assess the statistical assumption underlying the CMH stratified analysis procedure - namely the assumption on a common difference in unadjusted proportions across strata.

4. As the expected rate of HIV-1 RNA≥50 c/mL at week 48 is close to 0 (as a result of suppressed entry criteria), the 95% adjusted CI may be sensitive to the statistical method

used in its construction. Therefore, a sensitivity analysis using the Summary Score method (computed from the Miettinen-Nurminen CI limits of the stratum risk difference) will be performed to calculate the 95% CI of the adjusted treatment difference. This will be compared to the primary analysis method of CMH detailed above.

## 7.2. Secondary Efficacy Analyses

## 7.2.1. Endpoint / Variables

The secondary endpoints will include the following:

- The binary responses indicating the virologic outcome category of plasma HIV 1 RNA ≥50 c/mL at week 24 using the FDA Snapshot algorithm (see Appendix 11).
- The binary responses indicating the virologic outcome category of plasma HIV 1 RNA <50 c/mL at week 24 and Week 48 using the FDA Snapshot algorithm (see Appendix 11).
- CD4+ cell count at weeks 24 and 48.
- CD4+/CD8+ cell count ratio at weeks 24 and 48.
- Incidence of disease progression (HIV-associated conditions, AIDS, and death) through weeks 24 and 48

## 7.2.2. Summary Measure

- The number and percent of subjects with plasma HIV 1 RNA ≥50 c/mL at weeks 24 using the FDA snapshot algorithm (see Appendix 11).
- The number and percent of subjects with plasma HIV 1 RNA <50 c/mL at weeks 24 and 48 using the FDA snapshot algorithm (see Appendix 11).
- Change from baseline in CD4+ cell count at weeks 24 and 48.
- Change from baseline in CD4+/CD8+ cell count ratio at weeks 24 and 48.
- Incidence of disease progression (HIV-associated conditions, AIDS, and death) through weeks 24 and 48.

#### 7.2.3. Population of Interest

The secondary efficacy analyses will be based on the ITT-E population.

#### 7.2.4. Strategy for Intercurrent (Post-Randomization) Events

Intercurrent events such as discontinuations, missing plasma HIV-1 RNA samples and change in background regimen are handled using the FDA snapshot algorithm (see Appendix 11) which details how to assign each subject's virologic outcome. Intercurrent events will not be controlled for in disease progression and CD4+ cell count analyses.

## 7.2.5. Statistical Analyses / Methods

Table 5 provides an overview of the planned secondary efficacy analyses, with full details of data displays being presented in Appendix 17: List of Data Displays.

Table 5 Overview of Planned Secondary Efficacy Analyses

| Endpoints | Absolute | | | | | | | | | Chang | je from | Base | line | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Stats Summary Individual Analysis | | | Stats<br>Analysis | | | Summary | | Individual | | | | |
| | Т | F | L | T | F | F | L | Т | F | L | Т | F | F | L |
| Percent of Subjects | with F | Plasn | na H | IV-1 RN | <b>IA</b> ≥/ | <50 c/ | mL- S | nap | shot | | | | | |
| Plasma HIV-1<br>RNA ≥50 c/mL<br>analysis at Week<br>24 | Y | | | | | | | | | | | | | |
| Plasma HIV-1<br>RNA <50 c/mL<br>analysis at Week X | Υ[11] | | | <b>Y</b> [10] | | | | | | | | | | |
| Study Outcomes<br>(Plasma HIV-1<br>RNA ≥/ < 50 c/mL)<br>based on the<br>Snapshot at Week<br>X <sup>[6]</sup> | | | | Y | | | Y | | | | | | | |
| Plasma HIV-1<br>RNA <50 c/mL<br>analysis By Visit<br>through Week X [6] | | | | Y | | | | | | | | | | |
| Plasma HIV-1<br>RNA ≥50 c/mL<br>analysis By Visit<br>through Week X <sup>[6]</sup> | | | | Υ | | | | | | | | | | |
| Plasma HIV-1<br>RNA <50 c/mL<br>analysis by<br>subgroup at Week<br>X <sup>[6]</sup> | | | | Y | <b>Y</b> [1] | | | | | | | | | |
| Study Outcomes<br>(Plasma HIV-1<br>RNA ≥/ < 50 c/mL)<br>based on the<br>Snapshot by<br>subgroup at Week<br>X <sup>[6]</sup> | | | | Y | | | | | | | | | | |

| Endpoints | Absolute | | | | | | | | Change from Baseline | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stats<br>Analysis | | 3 | Summary | | Individual | | Stats<br>Analysis | | Summary | | Individual | | |
| | Т | F | L | Т | F | F | L | Т | F | L | Т | F | F | L |
| Percent of Subjects with Plasma HIV-1 RNA ≥/ <50 c/mL- Modified Snapshot | | | | | | | | | | | | | | |
| Study Outcomes<br>(Plasma HIV-1<br>RNA ≥/ < 50 c/mL)<br>at Week x <sup>[6]</sup> | | | | Y | | | Y | | | | | | | |
| Confirmed Virologic | Confirmed Virologic Withdrawal (CVW) | | | | | | | | | | | | | |
| HIV-1 RNA<br>distribution at time<br>of suspected and<br>confirmed Virologic<br>withdrawal | | | | Y | | | Y | | | | | | | |
| Potential Precautionary Virologic Withdrawal (pPVW) | | | | | | | | | | | | | | |
| pPVW by Visit | | | | | | | Υ | | | | | | | |
| Plasma HIV-1 RNA | over tir | ne – | Obs | served | | | | | | | | | | |
| By Visit through<br>Week X <sup>[6]</sup> | | | | | | | <b>Y</b> [2,9] | | | | Y [5] | | | |
| CD4+ Cell Counts [3 | 3] | | | | | | | | | | | | | |
| By Visit through Week X [6] | | | | | | Y<br>[2] | Υ | | | | Υ | | | Y |
| By Subgroup at Week X <sup>[6]</sup> | | | | | | | | | | | Y | | | |
| CD4+/CD8+ Cell Co | unt Ra | tio <sup>[3]</sup> | | | | | | | | | | | | |
| By Visit through<br>Week X [6] | | | | | | Y<br>[2] | Y | | | | Υ | | | Y |
| By Subgroup at Week X <sup>[6]</sup> | | | | | | | | | | | Υ | | | |
| Post-baseline HIV-1 | Disea | se Pi | rogr | ession | [4] | | | | | | | | | |
| HIV Conditions including Recurrences at Week X [6,7] | | | | Υ | | | Υ | | | | | | | |
| HIV Conditions<br>excluding<br>Recurrences at<br>Week X [6,7] | | | | Υ | | | | | | | | | | |
| HIV Disease<br>Progressions at<br>Week X <sup>[6,8]</sup> | | | | Υ | | | | | | | | | | |

## 1. NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.

  Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.

- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
  - 1. Plot of 95% confidence intervals for unadjusted treatment difference in the proportion of subjects below 50 c/mL with overall and by subgroup.
  - 2. Individual plasma HIV-1 RNA and CD4+ profiles only for subjects with at least one HIV-1 RNA levels ≥ 50 c/mL observed including at Day 1 and through withdrawal visit.
  - 3. Using observed case (OC) data which contains the data that is available at a particular time point, with no imputation for missing values.
  - 4. HIV disease progressions categories: CDC Category Stage 1 at enrolment to Stage 3 event; CDC Category Stage 2 at enrolment to Stage 3 event; CDC Category Stage 3 at enrolment to New Stage 3 Event; CDC Category Stage 0, 1, 2 or 3 at enrolment to Death.
  - 5. Descriptive summary of the log10 change from baseline HIV-1 RNA by visit presented.
  - 6. Week X refers to Week 24 and Week 48.
  - 7. Stage 3 only.
  - 8. Progression to Stage 3 or death.
  - 9. Includes target detected/not detected flag see Section 15.6.3 for more information.
  - 10. Repeated on the following endpoint: <40 c/mL and Target Not Detected Status.
  - 11. Repeated on the following endpoints: 1) <40 c/mL only, 2) <40 c/mL and Target Not Detected Status.

### 7.2.5.1. Statistical Methodology Specification

#### **Endpoint**

- The binary responses indicating the virologic outcome category of plasma HIV 1 RNA ≥50 c/mL at week 24 using the FDA Snapshot algorithm (see Appendix 11).
- The binary responses indicating the virologic outcome category of plasma HIV 1 RNA <50 c/mL at week 24 and Week 48 using the FDA Snapshot algorithm (see Appendix 11).
- The analysis approach will follow the methods as described for the primary endpoint.

#### **Model Specification**

Specification will be same as described for the primary endpoint

### **Model Checking & Diagnostics**

Same as described for the primary endpoint

#### **Model Results Presentation**

- Model presentation will be the same as described for the primary endpoint.
- Percent of subjects with plasma HIV 1 RNA ≥50 c/mL will be analysed at Weeks 24. Percent subjects with plasma HIV 1 RNA <50 c/mL will be analysed at Week 24 and Week 48.</li>
- For Percent of subjects with plasma HIV-1 RNA <50 c/mL endpoint, non-inferiority of switching to DTG/3TC compared to continuation of CAR (as per FDA snapshot algorithm) will be assessed using a -12% non-inferiority margin. Non-inferiority will be concluded if the lower bound of a 2-sided 95% confidence interval for the difference in success rates between the two treatment arms is greater than -12%.

#### **Subgroup Analyses**

Subgroup analyses will be performed for the percent of patients with plasma HIV 1 RNA <50 c/mL, study outcomes and unadjusted difference in proportion of patients with plasma HIV 1 RNA <50 c/mL between treatment arms at Week 24 and Week 48 endpoints (see Section 5.4.2).</li>

#### **Supportive Analyses**

- 1. Supportive analysis based on the <50 HIV-1 RNA endpoint will be performed based on the same analysis for the following endpoints:
  - Percent of Subjects with Plasma HIV-1 RNA <40 c/mL at Week 24 and Week 48</li>
  - Percent of Subjects with Plasma HIV-1 RNA <40 c/mL and Target Not Detected Status at Week 24 and Week 48
  - Percent of Subjects with Plasma HIV-1 RNA <40 c/mL and Target Not Detected Status at Week 24 and Week 48 by Baseline Third Agent Class
- 2. Proportion of subjects without virologic (ERDF) or virologic/tolerability (TRDF) failure:
  - Estimated using the Kaplan-Meier nonparametric method based on the time to Confirmed Virologic Withdrawal (CVW) criteria met or treatment-related (i.e. drug-

- related AE, protocol defined safety stopping criteria, or lack of efficacy)/efficacy related discontinuation (i.e. lack of efficacy).
- The detailed algorithm for TRDF (and ERDF) is listed in Appendix 10. The estimate of the standard error used to derive confidence intervals for the difference in proportions between treatment groups will be based on Greenwood's formula [Kalbfleisch, 1980]
- The estimated proportion of subjects without Confirmed Virologic Withdrawal and not discontinued due to treatment-related/efficacy-related reasons at Week 24 and at Week 48 will be presented by treatment group, along with estimated difference in proportions between treatment groups and its associated two-sided 95% CI.
- 3. Modified snapshot algorithm for study outcomes at Week 24 and Week48:
  - Snapshot study outcomes will be repeated using the modified snapshot algorithm. The
    modified snapshot includes additional sub-reasons under "HIV-1 RNA≥50 c/mL" and "No
    Virologic Data" snapshot categories that are further divided by relationship to COVID-19.
    For details see Section 15.12.

## 7.3. Exploratory Efficacy Analyses

- Subjects with plasma HIV-1 RNA <50 c/mL using the Snapshot algorithm at Week 24 and 48 by subgroup, based on the ITT-E population.
- Change from baseline CD4+ and CD4+/CD8+ ratio cell counts at Week 24 and 48 by subgroup.

These analyses have been specified in previous sections.

### 8. SAFETY ANALYSES

The safety analyses will be based on the Safety population, unless otherwise specified.

## 8.1. Adverse Events Analyses

Adverse events analyses including the analysis of adverse events (AEs), Serious (SAEs) and other significant AEs will be based on GSK Core Data Standards. The details of the planned displays are provided in Appendix 17: List of Data Displays.

Emergent AEs will be tabulated by treatment group and a total column. For AEs captured more than once, the most severe intensity will be included in summaries, and all events will be included in listings. For the purposes of summarising AE data, unless stated otherwise, the summaries will include post-baseline data.

For Week 24 and 48 analyses, outputs will be presented for the Randomized Phase unless otherwise specified. Safety data presented through weeks 24 and 48, will comprise all available safety data collected at that time point. For example, if some earlier recruiting subjects have reached Week 36 and have available safety data, this will be presented for the Week 24 analysis.

Table 6 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 17: List of Data Displays.

Table 6 Overview of Planned Safety Analyses

| Endpoint | Absolute | | | |
|---|---|---|---|---|
| | Sumi | mary | Individual | |
| | Т | F | F | L |
| Exposure | | | | |
| Extent of Exposure | Υ | | | Υ [1] |
| Adverse Events [2] | | | | |
| All AEs by SOC and PT <sup>[2, 7]</sup> | Υ | | | Υ |
| All AEs by Maximum Grade [2] | Υ | | | Υ [3] |
| Common AEs by Frequency [4] | Υ | Υ [5] | | |
| Common Grade 2-5 AEs [4] by Frequency | Υ | | | |
| Drug-Related AEs by SOC and PT | Υ | | | Y |
| All Drug-Related AEs by SOC and Maximum Grade | Υ | | | |
| Common non-Serious AEs by SOC and PT (subjects and number of occurrences) | Υ | | | |
| Common Drug-related Grade 2-5 AEs [4] | Υ | | | |
| Drug-Related AEs leading to withdrawal from study | Υ | | | |
| AEs Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment <sup>[8]</sup> | Υ | | | Υ |
| Serious and Other Significant AEs | | | | |
| All SAEs by SOC | Υ | | | |
| All Drug-Related SAEs by SOC | Υ | | | |
| Serious AEs by SOC and PT | Υ | | | |
| Reason for Considering as a Serious Adverse Event | | | | Υ |
| Possible Suicidality-Related Adverse Event (PSRAE) | | | | Y [6] |
| Cardiovascular events | | | | Y |
| Incidence of COVID-19 as reported as an AE and SAE <sup>[9]</sup> | Y | | | Y |
| Incidence of treatment discontinuation due to AE of COVID-19 infection <sup>[9]</sup> | Y | | | Y |
| Impact of Covid-19 on Assessment of Safety Base | d on COVID- | 19 eCRF | | |
| All AEs of Suspected, Probable, Confirmed for COVID-19 Infection | T | | | L |
| COVID-19 Diagnosis | T | | | L |

#### NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed data.

- 1. Includes reason for any dose change/interruption in both arms.
- 2. For AEs reported more than once by a subject, the most severe intensity will be included.
- 3. One listing of all AEs including verbatim text and preferred term, one showing the relationship between verbatim text, preferred term and SOC and another giving subject numbers for individual all treatment emergent AEs.
- 4. Common AEs are those with >=2% (or 0.5% for drug-related grade 2-5 AEs if there are no such AEs >=2%) incidence in either treatment group summarised by frequency.
- 5. Plots of incidence rates and relative risk with 95% CI for DTG/3TC vs. CAR.
- 6. Four PSRAE listings: Event and Description (Section 1- Section 2), Possible Cause (Section 3), Section 4 and Section 5-Section 8.
- 7. Repeated by subgroup (see Section 5.4.2).
- 8. Repeated by maximum grade as well.
- 9. Incidence of COVID-19 reported as an AE, SAE, treatment discontinuation due to AE of COVID-19 infection will be available in the adverse events summary tables/listings.

## 8.2. Adverse Events of Special Interest Analyses

A comprehensive list of MedDRA terms based on clinical review will be used to identify each type of event (see Section 15.6.4). Changes to the MedDRA dictionary may occur between the start of the study and the time of reporting and/or emerging data from ongoing studies may highlight additional adverse events of special interest, therefore the list of terms to be used for each event of interest and the specific events of interest will be based on the safety review team (SRT) agreements in place at the time of reporting. An overview of the planned adverse events of special interest analyses are presented in Table 7 and full details of the planned displays are provided in Appendix 17: List of Data Displays.

Table 7 Overview of Planned Adverse Events of Special Interest Analyses

| Endpoint | Absolut | е | | |
|---|---|---|---|---|
| | Sumi | mary | Individual | |
| | Т | F | F | L |
| Adverse Events of Special Interest[1] | | | | |
| Characteristics of Post<br>Baseline AESI | Y | | | |

<sup>1. 1</sup> See Section 15.6.4. for detail list of AESI

# 8.3. Clinical Laboratory and Biomarker Analyses

Laboratory evaluations will be based on GSK Core Data Standards. Table 8 provides an overview of the planned laboratory analyses, with full details of data displays being presented in Appendix 17: List of Data Displays.

Table 8 Overview of Planned Laboratory Analyses

| Endpoint | Absolute | | | | Change from Baseline | | | | | | Max Post BL | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Summary | | Individual | | Summary | | Individual | | Stats<br>Analysis | | Summary | | Individual | |
| | Τ | F | F | L | T | F | F | L | Т | F | Т | F | F | L |
| Laboratory Values C | ver T | ime | | | | | | | | | | | | |
| Clinical Chemistry <sup>[7]</sup> | Υ | | | <b>Y</b> [1] | Υ | | | | | | | | | |
| Fasted Lipid<br>(Triglycerides, LDL,<br>HDL and TC and<br>TC/HDL) <sup>[2]</sup> | <b>Y</b> [4] | | Υ[3,4] | <b>Y</b> [1] | Υ[4] | | | | Y | Y | | | | |
| NCEP shifts in lipids | | | | | Y[4] | Y[3,4] | | | | | | | | |
| Hematology [7] | Υ | | | <b>Y</b> [1] | Υ | | | | | | | | | |
| Urine Dipstick | | | | <b>Y</b> [1] | | | | | | | | | | |
| Urine Concentration | | | | <b>Y</b> [1] | | | | | | | | | | |
| Liver Chemistries | | | | | | | | | | | | Υ | | |
| Clinical Laboratory | and Bi | iomar | kers <sup>[8]</sup> | | • | | | | | | | | | |
| Bone Biomarkers | | | | Υ | Υ | | | Υ | Υ | Υ | | | | |
| Renal Biomarkers | | | | Υ | Υ | | | Υ | Υ | Υ | | | | |
| Inflammation<br>Biomarkers | | | | Y | Υ | | | Y | Y | Y | | | | |
| Change from<br>Baseline in HOMA-<br>IR, HbA1c at Week<br>24 and 48 | | | | Y | Υ | | | Y | Y | Υ | | | | |
| HOMA-IR, HbA1c by visit | Y | | | | Υ | | | | Y | Υ | | | | |
| HOMA-IR vs Weight<br>Scatter Plot | | | | | | | <b>Y</b> [5] | | | | | | | |
| HOMA-IR cut-off<br>(>=2, >=3 and<br>>=4) at Week 24<br>and 48 | | | | | Y | | | | Y | | | | | |
| <b>Emergent Laborator</b> | у Тох | icities | <b>;</b> | | | | | | | | | | | |
| Clinical Chemistry | Υ | | | | | | | | | | | | | |
| Hematology | Υ | | | | | | | | | | | | | |
| AST, ALT and Total<br>Bilirubin Maximum<br>Post-Baseline<br>Emergent Toxicity<br>by Baseline<br>Hepatitis C Status | | | | | | | | | | | Y | | | |

NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- 1. Listings for subjects with abnormalities for potential clinical concern/importance, defined as any Grade1-5 toxicity for Chemistry (Including Lipids), Hematology and Urinalysis.
- 2. Present both mmol/L and mg/DL.
- 3. Heatmap plot of NCEP categories in lipids over time.
- Subjects on lipid-lowering agents at baseline are not included in summaries. see Lipids. Section 15.6.4 for more details
- 5. A scatter plot of change in HOMA-IR (y-axis) vs change in weight (x-axis) at Weeks 24 and 48.
- 6. See Section 15.6.4 for more details.
- 7. Repeated by subgroup
- 8. Subjects from China will not be evaluated on Inflammatory Biomarkers, telomere length, Bone biomarkers and some Renal biomarkers (Retinol Binding Protein,Beta-2-Microglobulin, Urine RBP/creatinine and Urine B2M/creatinine)

## 8.3.1. Lipid Parameters Analyses

#### **Statistical Analyses**

#### **Endpoints**

 Change from Baseline in Fasting Lipids (Triglycerides, LDL cholesterol, HDL cholesterol, Total Cholesterol and TC/HDL ratio) at Weeks 24 and 48

#### **Covariates & Factors**

- Baseline 3<sup>rd</sup> Line Agent
- CD4+ cell count (continuous)
- Age (continuous)
- Sex (Female vs. Male)
- Race (White, Black or African American, Asian, Other)

#### **Data Handling**

- Before model fitting, missing values are assigned in the Observed Case Dataset:
  - Non-fasting values will be set to missing.
  - Subjects initiated serum lipid-lowering therapy at baseline (see Section 15.6.4)
     will be excluded from the analysis.
  - All values after initiation of lipid-lowering agents will be set to missing
  - Missing scheduled visits do not need to be created (given all scheduled visits appear in the dataset)
  - Non-missing values will need to be natural logarithm (In) transformed (including baseline value when included in models)
  - Depending on data structure, transpose non-missing values by subject if necessary

#### **Model Specification**

- Multiple imputation technique will be used as described below;
  - Multiple imputations will be drawn from a multivariate normal imputation model (taking into account scheduled measurements prior to analysis timepoints) with a Markov Chain Monte Carlo (MCMC) approach to estimate posterior distributions. The MCMC method in the MI procedure in SAS calling SAS PROC MI will be used with multiple chains, 500 burn-in iterations, and a noninformative
prior. A random seed number of 208090 will be used in the SAS program. Where a subject has a monotone or non-monotone pattern of missingness, all of their missing observations can be imputed under this approach. The absolute value will be imputed before the change value is calculated. Imputations will be drawn separately for subsets of subjects according to their treatment group, i.e., based on means and variance-covariances from the same treatment group (Missing At Random (MAR) approach) conditioning on covariates (as defined above).

- The imputations will be carried out 1,000 times. An ANCOVA (Week 24)/ MMRM (Week 48), using the observed margins (OM) option, will be performed on each dataset produced adjusting for the covariates (listed above), treatment, and baseline value, regardless of their significance. PROC MI ANALYZE in SAS will be used to combine the 1,000 estimated least squares means and difference to produce one estimated mean with 95% CI and associated p-value for the adjusted mean difference between each treatment group at Week 24 and Week 48.
- Interactions between treatment and covariates will not be assessed.

# **Model Checking & Diagnostics**

Refer to Appendix 14: Model Checking and Diagnostics for Statistical Analyses.

#### **Model Results Presentation**

Given that data is log transformed, estimated adjusted ratio (Week 24/Baseline or Week 48/Baseline) for each treatment and geometric mean ratio ((DTG/3TC/ CAR)) together with corresponding 95% CI will be presented. Results of the ratio are also expressed as percent change in adjusted mean and percent treatment difference respectively where percent change is derived as 100\* [Exp(model parameter estimate) -1].

#### Sensitivity Analyses - ANCOVA (Week 24)

- Sensitivity Analysis with Analysis of Covariance (ANCOVA) will be performed on the original data without multiple imputation techniques to deal with the missing data.
- ANCOVA will use the observed margins (OM) option, adjusting for treatment, covariates (listed above) and baseline value.
- Type III tests for the least-squares (LS) means will be used for the statistical comparison; the 95% CI will also be reported. Treatment group comparisons at Week 24 will be reported.
- Adjusted least squares means and corresponding standard errors (SEs) of adjusted least squares means will be presented for each treatment, together with estimated treatment difference (DTG/3TC – CAR) and corresponding 95% confidence interval and p-value.
- Note: if any lipid parameter is not normally distributed then the geometric mean and a 95% CI of geometric mean will be presented for each treatment, as well as geometric mean ratios and corresponding 95% CI and a p-value.

# Sensitivity Analyses – MMRM( Week 48)

- Sensitivity Analysis with Mixed Model Repeated Measures (MMRM) will be performed on the original data without multiple imputation techniques to deal with the missing data.
- MMRM will use the observed margins (OM) option, adjusting for treatment, covariates (listed above) and baseline value, with visit as the repeated factor.
- The model will make no further assumptions about the correlations within-subject scores (the correlation matrix for within-subject errors will be unstructured).
- The repeated measures analysis will assume that the treatment difference can vary between visits (i.e., a treatment\*visit interaction will be included in the model). The model will also assume that the effect of baseline score for the endpoint can vary between visits (i.e., baseline score\*visit interaction will be included in the model).
- The Kenward-Roger method will be used to estimate the denominator degrees of freedom. Type III tests for the least-squares (LS) means will be used for the statistical comparison; the 95% CI will also be reported. Treatment group comparisons at Week 24 and Week 48 will be reported.
- Adjusted least squares means and corresponding standard errors (SEs) of adjusted least squares means will be presented for each treatment, together with estimated treatment difference (DTG/3TC – CAR) and corresponding 95% confidence interval and p-value.
- Note: if any lipid parameter is not normally distributed then the geometric mean and a 95% CI of geometric mean will be presented for each treatment, as well as geometric mean ratios and corresponding 95% CI and a p-value.

# 8.3.2. HOMA-IR and HbA1c Analyses

#### **Statistical Analyses**

#### **Endpoints**

 Change from baseline in HOMA-IR, HbA1c at Weeks 24 and 48 (refer to 15.6.4 for details of derivation)

#### **Covariates & Factors**

- Baseline 3<sup>rd</sup> Line Agent
- CD4+ cell count (continuous)
- Age (continuous)
- Sex (Female vs. Male)
- Race (White, Black or African American, Asian, Other)
- BMI (continuous)
- Presence of diabetes mellitus (DM) (Yes vs no): Applicable for HbA1c only
- Hypertension (Yes vs no)
- Baseline value(continuous)

#### **Data Handling**

No multiple imputation techniques will be used to deal with the missing data.

# **Model Specification**

- If change in HOMA-IR or HbA1c is not normally distributed the data will be log transformed and geometric means will replace arithmetic means, a 95% CI will replace the standard deviations and mean changes from baseline will be presented as geometric mean ratios.
- Change from baseline will be analysed for the comparison between DTG/3TC and CAR.
- Using OC dataset, the Mixed Model Repeated Measures (MMRM), using the observed margins (OM) option, will adjust for treatment, covariates (listed above) and baseline value as a covariate, with visit as the repeated factor.
- The model will make no further assumptions about the correlations between a subject's value (the correlation matrix for within-subject errors will be unstructured).
- The repeated measures analysis will assume that the treatment difference can vary between visits (i.e. a treatment\*visit interaction will be included in the model), and separate estimates and 95% confidence intervals will be produced at each visit. The model will also assume that the effect of baseline value for the endpoint can vary between visits (i.e. baseline value\*visit interaction will be included in the model).
- Interactions between treatment and each of the covariates will not be assessed.

# **Model Checking & Diagnostics**

Refer to Appendix 14: Model Checking and Diagnostics for Statistical Analyses.

#### **Model Results Presentation**

- Adjusted least squares means and corresponding standard errors (SEs) of adjusted least squares means will be presented for each treatment, together with estimated treatment difference (DTG/3TC – CAR) and corresponding 95% confidence interval and p-value.
- Note: If change from baseline in HOMA-IR or HbA1c data are not normally distributed, the geometric mean and a 95% CI of geometric mean will be presented for each treatment, as well as geometric mean ratios and corresponding 95% CI and a p-value.

## **Sensitivity Analyses**

- Line plots of LS means with 95% confidence intervals for Adjusted Mean Change from Baseline will be generated for each treatment group by visit
- A logistic regression model will be performed on the proportion of subjects with HOMA-IR cut-off (>=2, >=3 and >=4) at Week 24 and Week 48 adjusting for the same covariates as specified in the MMRM analysis (without visit or interaction terms). Odds ratios, standard errors, confidence intervals and p-values will be presented for all covariates specified in the model. This analysis will be repeated on the proportion of subjects with HOMA-IR cut-off (>=2, >=3 and >=4) at Week 24 and Week 48. Upon delivery of data, an assessment regarding the amount of missing data will be made. If it's considered the amount of missing HOMA-IR outcome data at Week 24 and Week 48 as a result of COVID-19 is substantial, the logistic regression analysis may not be performed.

# **Subgroup Analyses**

Not applicable

## 8.3.3. Bone Biomarkers Analyses

#### **Statistical Analyses**

#### **Endpoints**

 Change from baseline in bone biomarkers (bone specific alkaline phosphatase, procollagen type I N-terminal propeptide, type I collagen cross-linked C-telopeptide, osteocalcin) at Weeks 24 and 48

#### **Covariates & Factors**

- Baseline 3<sup>rd</sup> Line Agent
- CD4+ cell count (continuous)
- Age (continuous)
- Sex (Female vs. Male)
- Race (White, Black or African American, Asian, Other)
- BMI (continuous)
- Smoking status (Never vs. Former vs. Current Smoker)
- Baseline value(continuous)

#### **Data Handling**

No multiple imputation techniques will be used to deal with the missing data.

# Model Specification - ANCOVA (Week 24)

- It is anticipated that at least some biomarkers will not be normally distributed and for those, the data will be log transformed and geometric means will replace arithmetic means, a 95% CI will replace the standard deviations and mean changes from baseline will be presented as geometric mean ratios.
- Change from baseline will be analysed for each bone biomarker for the comparison between DTG/3TC and CAR.
- An Analysis of Covariance (ANCOVA), using the observed margins (OM) option, will adjust for treatment, covariates (listed above) and biomarker value at baseline as a covariate. The OC dataset will be used for ANCOVA model.

# Model Specification - MMRM (Week 48)

- It is anticipated that at least some biomarkers will not be normally distributed and for those, the data will be log transformed and geometric means will replace arithmetic means, a 95% CI will replace the standard deviations and mean changes from baseline will be presented as geometric mean ratios.
- Change from baseline will be analysed for each bone biomarker for the comparison between DTG/3TC and CAR.
- Mixed Model Repeated Measures (MMRM), using the observed margins (OM) option, will
  adjust for treatment, covariates (listed above) and biomarker value at baseline as a
  covariate, with visit as the repeated factor. The OC dataset will be used for MMRM model.
- The model will make no further assumptions about the correlations between a subject's value (the correlation matrix for within-subject errors will be unstructured).
- The repeated measures analysis will assume that the treatment difference can vary between visits (i.e. a treatment\*visit interaction will be included in the model) and separates estimates and 95% confidence intervals will be produced at each visit. The model will also assume that the effect of baseline value for the endpoint can vary between visits (i.e. baseline value\*visit interaction will be included in the model).

Interactions between treatment and each of the covariates will not be assessed.

#### **Model Checking & Diagnostics**

• Refer to Appendix 14: Model Checking and Diagnostics for Statistical Analyses.

#### Model Results Presentation

- Adjusted least squares means and corresponding standard errors (SEs) of adjusted least squares means will be presented for each treatment, together with estimated treatment difference (DTG/3TC – CAR) and corresponding 95% confidence interval and p-value.
- Note: For biomarkers that are not normally distributed, the geometric mean and a 95% CI of geometric mean will be presented for each treatment, as well as geometric mean ratios and corresponding 95% CI and a p-value.

# **Sensitivity Analyses**

 Line plots of LS means with 95% confidence intervals for Adjusted Mean Change from Baseline will be generated for each treatment group by visit

## **Subgroup Analyses**

Not applicable

# 8.3.4. Renal Biomarkers Analyses

### **Statistical Analyses**

#### **Endpoints**

Change from baseline in renal biomarkers (serum Cystatin C, Urine Beta-2 Microglobulin /Urine Creatinine ratio (mg/mmol), urine albumin/creatinine ratio, urine protein/creatinine ratio, urine phosphate, eGFR (based on CKD-EPI-creatinine and CKD-EPI-cystatin C), serum creatinine and Urine Retinol Binding Protein 4/Urine Creatinine ratio (ug/mmol)) at Weeks 24 and 48

#### **Covariates & Factors**

- Baseline 3<sup>rd</sup> Line Agent
- CD4+ cell count (continuous)
- Age (continuous)
- Sex (Female vs. Male)
- Race (White, Black or African American, Asian, Other)
- BMI (continuous)
- Presence of diabetes mellitus (DM) (Yes vs no)
- Presence of Hypertension (Yes v no)
- Baseline value(continuous)

#### **Data Handling**

• No multiple imputation techniques will be used to deal with the missing data.

## Model Specification - ANCOVA (Week 24)

- It is anticipated that at least some biomarkers will not be normally distributed and for those, the data will be log transformed and geometric means will replace arithmetic means, a 95% CI will replace the standard deviations and mean changes from baseline will be presented as geometric mean ratios.
- Change from baseline will be analysed for each bone biomarker for the comparison between DTG/3TC and CAR.

 An Analysis of Covariance (ANCOVA), using the observed margins (OM) option, will adjust for treatment, covariates (listed above) and biomarker value at baseline as a covariate. The OC dataset will be used for ANCOVA model.

# Model Specification – MMRM (Week 48)

- It is anticipated that at least some biomarkers will not be normally distributed and for those, the data will be log transformed and geometric means will replace arithmetic means, a 95% CI will replace the standard deviations and mean changes from baseline will be presented as geometric mean ratios.
- Change from baseline will be analysed for each renal biomarker for the comparison between DTG/3TC and CAR.
- Using OC dataset, the Mixed Model Repeated Measures (MMRM), using the observed margins (OM) option, will adjust for treatment, covariates (listed above) and baseline renal biomarker value at baseline as a covariate, with visit as the repeated factor.
- The model will make no further assumptions about the correlations between a subject's value (the correlation matrix for within-subject errors will be unstructured).
- The repeated measures analysis will assume that the treatment difference can vary between visits (i.e. a treatment\*visit interaction will be included in the model), and separate estimates and 95% confidence intervals will be produced at each visit. The model will also assume that the effect of baseline value for the endpoint can vary between visits (i.e. baseline value\*visit interaction will be included in the model).
- Interactions between treatment and each of the covariates will not be assessed.

# **Model Checking & Diagnostics**

Refer to Appendix 14: Model Checking and Diagnostics for Statistical Analyses.

#### **Model Results Presentation**

- Adjusted least squares means and corresponding standard errors (SEs) of adjusted least squares means will be presented for each treatment, together with estimated treatment difference (DTG/3TC – CAR) and corresponding 95% confidence interval and p-value.
- Note: For biomarkers that are not normally distributed, the geometric mean and a 95% CI of geometric mean will be presented for each treatment, as well as geometric mean ratios and corresponding 95% CI and a p-value.

### **Sensitivity Analyses**

- Line plots of LS means with 95% confidence intervals for Adjusted Mean Change from Baseline will be generated for each treatment group by visit
- A sensitivity analysis will be performed for urine albumin/creatinine ratio and urine protein/creatinine ratio by imputing albumin, protein and creatinine values that are below the limit of quantitation. See Appendix 7.

# **Subgroup Analyses**

Not applicable

# 8.3.5. Inflammatory Biomarkers Analyses

#### **Statistical Analyses**

#### **Endpoints**

Change from baseline in inflammatory biomarkers (Interleukin-6 (IL-6), High-sensitivity C reactive protein (hs-CRP), D-dimer, Soluble CD14 (sCD14), Soluble CD163 (sCD163)) at Weeks 24 and 48

#### **Covariates & Factors**

- Baseline 3<sup>rd</sup> Line Agent
- CD4+ cell count (continuous)
- Age (continuous)
- Sex (Female vs. Male)
- Race (White, Black or African American, Asian, Other)
- BMI (continuous)
- Smoking status (Never vs. Former vs. Current Smoker)
- HCV-coinfection (Yes vs. No)
- Baseline value(continuous)

# **Data Handling**

No multiple imputation techniques will be used to deal with the missing data.

# Model Specification - ANCOVA (Week 24)

- It is anticipated that at least some biomarkers will not be normally distributed and for those, the data will be log transformed and geometric means will replace arithmetic means, a 95% CI will replace the standard deviations and mean changes from baseline will be presented as geometric mean ratios.
- Change from baseline will be analysed for each bone biomarker for the comparison between DTG/3TC and CAR.
- An Analysis of Covariance (ANCOVA), using the observed margins (OM) option, will adjust for treatment, covariates (listed above) and biomarker value at baseline as a covariate. The OC dataset will be used for ANCOVA model.

# Model Specification - MMRM (Week 48)

- It is anticipated that at least some biomarkers will not be normally distributed and for those, the data will be log transformed and geometric means will replace arithmetic means, a 95% CI will replace the standard deviations and mean changes from baseline will be presented as geometric mean ratios.
- Change from baseline will be analysed for each inflammatory biomarker for the comparison between DTG/3TC and CAR.
- Using OC dataset, the Mixed Model Repeated Measures (MMRM), using the observed margins (OM) option, will adjust for treatment, covariates (listed above) and baseline inflammatory biomarker value at as a covariate, with visit as the repeated factor.
- The model will make no further assumptions about the correlations between a subject's value (the correlation matrix for within-subject errors will be unstructured).
- The repeated measures analysis will assume that the treatment difference can vary between visits (i.e. a treatment\*visit interaction will be included in the model), and separate estimates and 95% confidence intervals will be produced at each visit. The model will also assume that the effect of baseline value for the endpoint can vary between visits (i.e. baseline value\*visit interaction will be included in the model).
- Interactions between treatment and each of the covariates will not be assessed.

#### **Model Checking & Diagnostics**

Refer to Appendix 14: Model Checking and Diagnostics for Statistical Analyses.

#### **Model Results Presentation**

- Adjusted least squares means and corresponding standard errors (SEs) of adjusted least squares means will be presented for each treatment, together with estimated treatment difference (DTG/3TC – CAR) and corresponding 95% confidence interval and p-value.
- Note: For biomarkers that are not normally distributed, the geometric mean and a 95% CI of geometric mean will be presented for each treatment, as well as geometric mean ratios and corresponding 95% CI and a p-value.

# **Sensitivity Analyses**

 Line plots of LS means with 95% confidence intervals for Adjusted Mean Change from Baseline will be generated for each treatment group by visit

# **Subgroup Analyses**

Not applicable

# 8.4. Other Safety Analyses

The analyses of non-laboratory safety test results will be based on GSK Core Data Standards, unless otherwise specified. An overview of other safety analyses is presented in Table 9 and full details of the planned displays are presented in Appendix 17: List of Data Displays. Note that ECGs and vital signs are only collected at screening, so will only be listed.

Table 9 Overview of Other Safety Analyses

| Endpoint | | Α | bsolu | ite | | Chan | ge fro | m Ba | seline | | ı | Max P | ost Bl | _ |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Sum | mary | Indiv | vidual Summary | | Indiv | ndividual Sta<br>Anal | | | | mary | Individual | | |
| | Т | F | F | L | Т | F | F | L | Τ | F | Т | F | F | L |
| Other Safety Analys | es | | | | | | | | | | | | | |
| ECG at screening | | | | Υ | | | | | | | | | | |
| Vital Signs | | | | Υ | | | | | | | | | | |
| Liver Assessment | Υ | | | Υ | | | | | | | | | | |
| Hepatobiliary<br>Abnormality criteria | Y | | | <b>Y</b> [3] | | | | | | | | | | |
| eC-SSRS | Υ | | | <b>Y</b> [1] | | | | | | | | | | |
| Subjects who became Pregnant | | | | Υ | | | | | | | | | | |
| Patient Profiles | | | | <b>Y</b> [2] | | | | | | | | | | |
| Pharmacokinetics<br>Listings for Subjects<br>with Liver Stopping<br>Events | | | | Y | | | | | | | | | | |

| Endpoint | | Α | bsolu | ıte | | Chan | ge fro | m Ba | seline | | Max Post BL | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Summary | | Individual | | Sum | Summary | | Individual | | ats<br>lysis | Summary | | Individual | |
| | Т | F | F | L | Т | F | F | L | Т | F | Т | F | F | L |
| Weight and BMI | | | | | | | | | | | | | | |
| Change from<br>baseline in BMI at<br>Weight at Week 24<br>and 48 | | | | Y | Y | | | Y | Y | Υ | | | | |
| BMI <sup>[4]</sup> and Weight by Visit | Y | | | | Υ | | | | Y | Y | | | | |
| BMI shift Table | Υ | | | | | | | | | | | | | |

- 1. Includes Baseline and lists all visits for a subject who reports any ideation or behaviour at any visit.
- 2. Patient profiles for subjects meeting protocol defined liver stopping criteria and for patients with HIV-1 RNA ≥ 50 c/mL. Patient profiles can also be provided for any other subjects.
- 3. All post-baseline abnormalities meeting Hepatobiliary Abnormality Criteria.
- 4. Heatmap plot of BMI categories over time.

### 8.4.1. Weight and BMI Analyses

#### **Statistical Analyses**

# **Endpoints**

Change from baseline in weight (kg) and BMI (kg/m2) at Weeks 24 and 48

#### **Covariates & Factors**

- Baseline 3<sup>rd</sup> Line Agent
- CD4+ cell count (continuous)
- Age (continuous)
- Sex (Female vs. Male)
- Race (White, Black or African American, Asian, Other)
- Baseline value(continuous)

# **Data Handling**

No multiple imputation techniques will be used to deal with the missing data.

#### **Model Specification**

- If the change from baseline in weight (BMI for BMI analysis) is not normally distributed, the
  data will be log transformed and geometric means will replace arithmetic means, a 95% CI
  will replace the standard deviations and mean changes from baseline will be presented as
  geometric mean ratios.
- Change from baseline will be analysed for the comparison between DTG/3TC and CAR.
- Using OC dataset, the Mixed Model Repeated Measures (MMRM), using the observed margins (OM) option, will adjust for treatment, covariates (listed above) and baseline weight (BMI for BMI analysis) value as a covariate, with visit as the repeated factor.
- The model will make no further assumptions about the correlations between a subject's weight (BMI for BMI analysis) (the correlation matrix for within-subject errors will be unstructured).
- The repeated measures analysis will assume that the treatment difference can vary between visits (i.e. a treatment\*visit interaction will be included in the model), and separate estimates and 95% confidence intervals will be produced at each visit. The model will also assume that the effect of baseline weight (BMI for BMI analysis) can vary between visits (i.e. baseline value\*visit interaction will be included in the model).
- Interactions between treatment and each of the covariates will not be assessed.

# **Model Checking & Diagnostics**

• Refer to Appendix 14: Model Checking and Diagnostics for Statistical Analyses.

#### Model Results Presentation

- Adjusted least squares means and corresponding standard errors (SEs) of adjusted least squares means will be presented for each treatment, together with estimated treatment difference (DTG/3TC – CAR) and corresponding 95% confidence interval.
- Note: If change in weight is not normally distributed, the geometric mean and a 95% CI of geometric mean will be presented for each treatment, as well as geometric mean ratios and corresponding 95% CI and p-values.

#### **Sensitivity Analyses**

• Line plots of LS means with 95% confidence intervals for Adjusted Mean Change from Baseline will be generated for each treatment group by visit.

#### Subgroup Analyses

Not applicable

# 9. OTHER STATISTICAL ANALYSES

# 9.1. Health Outcomes

# 9.1.1. Overview of Planned Analyses

The Health Outcomes analyses will be based on the Intent-To-Treat (Exposed) population, unless otherwise specified.

Table 10 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 17: List of Data Displays.

Table 10 Overview of Planned Health Outcome Analyses

| Endpoints | | Absolute | | | | | | | Char | nge | from | Baseli | ne | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stat | Stats Analysis Summary Individual S | | | Stats | Analys | is | Sum | mary | Individual | | | | |
| | Т | F | L | Т | F | F | L | Т | F | L | T | F | F | L |
| Symptom Distress Module (SDM) | | | | | | | | | | | | | | |
| Symptom Count (at Week 24 and 48) | | | | Υ | | | Υ | | | | Y | | | |
| Symptom Bother<br>Score (at Week 24<br>and 48) | | | | Υ | | | Υ | <b>Y</b> [3] | Y[1] | | Y | | | |
| Willingness to swit | ch | | | | | | | | | | | | | |
| Willingness to switch survey | | | | Υ | | | | | | | | | | |
| Treatment satisfact | tion | | | | | | | | | | | | | |
| HIVTSQ individual item scores by Visit | | | | Υ | | | Y | | | | | | | |
| HIVTSQ (at Week 24 and 48) | <b>Y</b> [2] | | | <b>Y</b> [2] | | | | Υ[2,3] | Υ[1,2] | | Υ[2] | | | |

<sup>1.</sup> Line Plot of Adjusted Mean (95% CI) and Line Plot of Difference (95% CI) in Adjusted Mean Change from Baseline over time.

# 9.1.2. Planned Health Outcomes Statistical Analyses

# Statistical Analyses

#### **Endpoints**

- Change from baseline in Overall Symptom Bother score at Week 24 and 48
- Change from baseline in HIVTSQ total score at Week 24 and 48
- Change from baseline in HIVTSQ general satisfaction/clinical sub-score at Week 24 and 48
- Change from baseline in HIVTSQ lifestyle/ease sub-scores at Week 24 and 48

<sup>2.</sup> Separate summaries for Total score (questionnaire items 1-10), General Satisfaction/Clinical sub-score (questionnaire items and ) and Lifestyle/ease sub-score (questionnaire items and ).

<sup>3.</sup> Repeat by subgroups (see Section 5.4.2).

#### **Covariates & Factors**

- Baseline 3<sup>rd</sup> Line Agent
- Age (continuous)
- Sex (Female vs. Male)
- Race (White, Black or African American, Asian, Other)
- Baseline score

#### **Data Handling**

No multiple imputation techniques will be used to deal with the missing data.

### **Model Specification**

- If the endpoint is not be normally distributed then, the data will be log transformed and geometric means will replace arithmetic means, a 95% CI will replace the standard deviations and mean changes from baseline will be presented as geometric mean ratios.
- Change from baseline will be analysed for the comparison between DTG/3TC and CAR
- Using OC dataset, Mixed Model Repeated Measures (MMRM), using the observed margins (OM) option, will adjust for treatment, covariates (listed above) and baseline score value as a covariate, with visit as the repeated factor.
- The model will make no further assumptions about the correlations between a subject's score (the correlation matrix for within-subject errors will be unstructured).
- The repeated measures analysis will assume that the treatment difference can vary between visits (i.e. a treatment\*visit interaction will be included in the model) and separates estimates and 95% confidence intervals will be produced at each visit. The model will also assume that the effect of baseline score for the endpoint can vary between visits (i.e. baseline score\*visit interaction will be included in the model).
- Interactions between treatment and each of the covariates will not be assessed.

#### **Model Checking & Diagnostics**

Refer to Appendix 14: Model Checking and Diagnostics for Statistical Analyses.

#### **Model Results Presentation**

- Adjusted least squares means and corresponding standard errors (SEs) of adjusted least squares means will be presented for each treatment, together with estimated treatment difference (DTG/3TC – CAR) and corresponding 95% confidence interval and p-value.
- Note: if SDM bother score is not normally distributed, the geometric mean and a 95% CI of geometric mean will be presented for each treatment, as well as geometric mean ratios and corresponding 95% CI and a p-value.

# **Sensitivity Analyses**

 Line plots of LS means with 95% confidence intervals for Adjusted Mean Change from Baseline will be generated for each treatment group by visit

### **Subgroup Analyses**

 Subgroup analyses will be performed for change from baseline in Overall Symptom Bother score and HIVTSQ total score at Week 24 and 48. Analysis will be performed as described above and will adjust for the covariates listed above, treatment, baseline score, subgroup, baseline score\*visit and treatment\*subgroup interaction term regardless of their significance (Subgroups are defined in Section 5.4.2).

#### Endpoint(s)

Willingness to switch survey

# Model Specification/Analysis Methodology

- Assess the reason(s) for their participation and facilitate an understanding of subject's willingness to switch
- A single item question prior to randomisation.
- 7 reasons for willingness to participate in a clinical study where the current HIV medication may be switched check all that apply
- Any missing values will remain missing

#### **Model Results Presentation**

Summary statistics will be presented by treatment group

# 9.2. Virology

# 9.2.1. Overview of Planned Analyses

### 9.2.2. Planned Virology Statistical Analysis

The virology analyses of genotype and phenotype data will be based on the CVW and pPVW resistance populations. Please see Section 15.6.3 for details of the derivation of CVW. Please see Section 15.6.3 for details of the derivation of pPVW.

The CVW population will be based on subjects who have experienced a CVW at any point. Summary tables will present CVWs up to and including the time point of interest. CVWs must be confirmed within the phase in which they are reported. Listings will present CVWs occurring at any point. Summary tables will present CVWs at the time point of SVW (or first elevation if this was >=50 c/mL and <200 c/mL).'

Table 11 provides an overview of the planned virology analyses, with full details of data displays being presented in Appendix 17: List of Data Displays.

Table 11 Overview of Planned Virology Analyses

| Endpoint | Absolute | | | |
|---|---|---|---|---|
| | Sumn | nary | Indivi | dual |
| | T | F | F | L |
| HIV-1 Subject Genotypic/Phenotypic Data A | HIV-1 Subject Genotypic/Phenotypic Data Accountability | | | |
| Genotypic Accountability | <b>Y</b> [2] | | | |
| Phenotypic Accountability | <b>Y</b> [2] | | | |
| Genotypic resistance | | | | |
| Genotypic resistance at time of CVW <sup>[1]</sup> | <b>Y</b> [2] | | | <b>Y</b> [4] |
| Genotypic resistance for subjects on treatment non-CVW time point <sup>[1]</sup> | <b>Y</b> [2] | | | Υ |
| Phenotypic resistance <sup>[5]</sup> | | | | |
| Phenotypic resistance at time of CVW <sup>[1]</sup> | <b>Y</b> [3] | | | <b>Y</b> [4] |

| Endpoint | | Abso | olute | |
|---|---|---|---|---|
| | Sumr | mary | Indivi | dual |
| | T | F | F | L |
| Phenotypic resistance for subjects on treatment at non-CVW time point <sup>[1]</sup> | <b>Y</b> [2] | | | Υ |
| INI and RT/PR replication capacity at time of CVW <sup>[1]</sup> | | | | <b>Y</b> [4] |
| INI and RT/PR replication capacity at time of non-CVW[1] | | | | <b>Y</b> [4] |
| Fold Change at CVW | Υ | | | |
| Net Assessment for Overall Susceptibility S | core | | | |
| Overall Susceptibility Score (OSS) | | | | Y |

- 1. NOTES:
- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data
- Individual = Represents FL related to any displays of individual subject observed raw data.
- 1. Sample used for resistance testing is taken at the time suspected virologic withdrawal criteria are met, and only tested once virologic withdrawal criteria are confirmed at a subsequent visit.
- 2. Separate outputs for INI and NRTI/NNRTI/PI mutations
- 3. Separate outputs by phenotypic cut-off and by number of drugs to which subjects are resistant.
- 4. Produce for CVW and pPVW resistance populations.
- 5. Phenotypic data are not available at Baseline because Genosure archive assay being used only provides genotype and not phenotype

# 10. PHARMACOKINETIC ANALYSES

There are no pharmacokinetic analyses planned for this study.

# 11. POPULATION PHARMACOKINETIC (POPPK) ANALYSES

There are no population pharmacokinetic analyses planned in this study.

# 12. PHARMACODYNAMIC ANALYSES

There are no pharmacodynamic analyses planned for this study.

# 13. PHARMACOKINETIC / PHARMACODYNAMIC ANALYSES

There are no pharmacokinetic / pharmacodynamic (PK/PD) analyses planned in this study.

# 14. REFERENCES

D'Agostino R.B., Vasan R.S., Pencina M.J., Wolf P.A., Cobain M., Massaro J.M. Kannel W.B. General Cardiovascular Risk Profile for Use in Primary Care: The Framingham Heart Study. *Epidemiology*. 2008; 117:743-753.

Fleiss J.L. Statistical Methods for Rates and Proportions. 2nd ed. New York: John Wiley; 1981.

Grundy S.M., et al. Executive summary of the third report of the National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation and Treatment of High Blood Cholesterol in Adults (Adult Treatment Panel III). *JAMA*. 2001;285

Inker LA, Schmid CH, Tighiouart H, et al; Estimating Glomerular Filtration Rate from Serum Creatinine and Cystatin C. *N Engl J Med.* 2012;367:20-9.

Johnson VA, Calvez V, Gunthard HF, et. al. Special Contribution. Update of the Drug Resistance Mutations in HIV-1: March 2013. IAS-USA Topics in Antiviral Medicine. Available at: https://www.iasusa.org/sites/default/files/tam/21-1-6.pdf. Accessed Octover 24, 2016.

Justice A, Holmes W, Gifford A, et al. Development and validation of a self completed HIV symptom index. Journal of Clinical Epidemiology. 2001; 54:S77-S90

Kalbfleisch JD, Prentice RL. The Statistical Analysis of Failure Time Data. *New York: Wiley*, 1980

Klingenberg. A new and improved confidence interval for the Mantel-Haenszel risk difference. *Statistics in Medicine*. 2014; 2968-2983.

Levey AS, Stevens LA, Schmid CH, et.al. A new equation to estimate glomerular filtration rate. *Ann Int Med.* 2009;150:604-12.

Liu TF, Shafer RW. Web Resources for HIV type 1 Genotypic-Resistance Test Interpretation. *Clin Infect Dis.* 2006;42 (11):1608-1618.

Lui K.J., Kelly C. A Revisit on Tests for Homogeneity of the Risk Difference, *Biometrics*, 2000;56:309-315.

Miettinen O, Nurminen M. Comparative Analysis of two rates. *Statistics in Medicine*. 1985; 4:213-226.

Posner K, Oquendo MA, Gould M, Stanley B, Davies M. Columbia Classification Algorithm of Suicide Assessment (C-CASA): classification of suicidal events in the FDA's pediatric suicidal risk analysis of antidepressants. *Am J Psychiatry*. 2007;164:1035–43.

Sato T. On the variance estimator for the Mantel-Haenszel risk difference. *Biometrics*. 1989;42:311-323.

Woodcock A, Bradley C . Validation of the HIV treatment satisfaction questionnaire (HIVTSQ). Qual Life Res. 2001;10(6):517-531.

Woodcock A, Bradley C. Validation of the revised 10-item HIV Treatment Satisfaction Questionnaire status version and new change version. Value Health. 2006;9(5):320-333.

# 15. APPENDICES

| Section | Appendix |
|---|---|
| RAP Section 4: | Analysis Populations |
| Section 15.1 | Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population |
| RAP Section 5 : 0 | General Considerations for Data Analyses & Data Handling Conventions |
| Section 15.2 | Appendix 2: Schedule of Activities |
| Section 15.3 | Appendix 3: Assessment Windows |
| Section 15.4 | Appendix 4: Study Phases and Emergent Adverse Events |
| Section 15.5 | Appendix 5: Data Display Standards & Handling Conventions |
| Section 15.6 | Appendix 6: Derived and Transformed Data |
| Section 15.7 | Appendix 7: Reporting Standards for Missing Data |
| Section 15.8 | Appendix 8: Values of Potential Clinical Importance |
| Section 15.9 | Appendix 9: Population Pharmacokinetic (PopPK) Analyses |
| Section 15.10 | Appendix 10: Time to Event Details |
| Section 15.11 | Appendix 11: Snapshot Algorithm details |
| Section 15.12 | Appendix 12: Modified Snapshot Algorithm details |
| Other RAP Appe | ndices |
| Section 15.13 | Appendix 13: Abbreviations & Trade Marks |
| Section 15.14 | Appendix 14: Model Checking and Diagnostics for Statistical Analyses |
| Section 15.15 | Appendix 15: Test of Homogeneity: Fleiss, Liu & Kelly Method |
| Section 15.16 | Appendix 16: Final (EoS) Analysis |
| Section 15.17 | Appendix 17: List of Data Displays |
| Section 15.18 | Appendix 18: Example Mock Shells for Data Displays |

# 15.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population

# 15.1.1. Exclusions from Per Protocol Population

A subject meeting any of the following criteria (Significant Protocol Deviations) will be excluded from the Per Protocol population:

| Number | Exclusion criteria |
|---|---|
| 01 | Subject deviates from any inclusion or exclusion criteria, as recorded in the eCRF |
| 02* | Subject took/received incorrect IP, i.e., other than the one to which they were randomized for greater than 10% of the total time On-treatment |
| 03* | Interruption of IP for greater than 10% of the total time On-treatment, for reasons other than treatment-related adverse events/laboratory abnormalities, based on eCRF IP exposure forms or eCRF CONMEDS forms in case commercial supply is used before study completion. |
| 04 | HIV immunotherapeutic vaccines used |
| 05 | Concurrent use of drugs that may decrease DTG concentration for >7 days: (Carbamazepine, Oxycarbamazapine, Phenobarbital, Phenytoin, St. John's wort (Hypericum perforatum), rifampin |
| 06 | Concomitant use of rifapentin |
| 07 | Other experimental agents, antiretroviral drugs not otherwise specified in the protocol, cytotoxic chemotherapy, or radiation therapy used |
| 08 | Systemically administered immunomodulators used through Week 48 visit |
| 09 | HCV therapy based on interferon or any other medications that have a potential for adverse drug-drug interactions with study treatment |
| 10 | Concomitant use of acetaminophen in subjects with acute viral hepatitis |
| 11 | Dofetilide or pilsicainide used concurrently |

| Number | Exclusion criteria |
|---|---|
| | with DTG |
| 12 | Subject's change (i.e., substitution or dose modification) of DTG, 3TC or component of CAR (except protocol allowed switches, e.g. switch of booster) but was not withdrawn from the study |
| 13 | Subject became pregnant while on study |
| 14 | Permanent discontinuation of IP/withdrawal due to a reason of "Protocol Deviation" (as recorded in the eCRF) |

<sup>\*</sup>Programmatically derived protocol deviations (PD), which are defined in a separate protocol deviations specification document. Please refer to Section 15.6.7 regarding cutoff dates regarding protocol deviations leading to exclusion from the per protocol set.

# 15.2. Appendix 2: Schedule of Activities

# 15.2.1. Protocol Defined Schedule of Events

| Procedures | g Visit <sup>a</sup> | Randomized Phase | | | | | | | Continuation<br>Phase <sup>c</sup> | drawal | Follow-up <sup>d</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening Visita | Baseline/<br>Day 1 | 4 | 12 | 24 | 36 | 48 <sup>b</sup> | 52 | Every 12<br>Weeks<br>After<br>Week 52 | Withdrawal | Follow |
| Clinical and Other Assessments | | | | | | | | | | | |
| Written informed consent | Χ | | | | | | | | | | |
| Inclusion/Exclusion criteriae | Χ | Х | | | | | | | | | |
| Demography | Χ | | | | | | | | | | |
| Prior ART history | Χ | | | | | | | | | | |
| Medical history <sup>f</sup> | Χ | | | | | | | | | | |
| Menopause historyg | Χ | Х | | | | | | Χ | | Х | |
| Current medical conditions | Χ | | | | | | | | | | |
| Cardiovascular risk assessment including vital signs <sup>h</sup> | Х | | | | | | | | | | |
| Body Weight (BMI will be calculated within the eCRF) <sup>i</sup> | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| HIV risk factors and mode of transmission | | Х | | | | | | | | | |
| CDC HIV-1 classification | Χ | Х | | | | | | | | | |
| HIV associated conditions | | Х | Х | Х | Х | Х | Х | Χ | Χ | Х | |
| Columbia Suicidality Severity Rating Scale | | Xk | Х | Х | Х | Х | Χ | Х | Χ | Х | |
| Concomitant medication | Χ | Х | Х | Х | Х | Х | Χ | Х | Χ | Х | Х |
| Symptom Directed Physical Exam <sup>l</sup> | Χ | Х | Х | Х | Х | Х | Χ | | Χ | Х | Х |

| Procedures | g Visit <sup>a</sup> | | | Rand | omized I | Phase | | | Continuation<br>Phase <sup>c</sup> | awal | pdn-/ |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening Visit <sup>a</sup> | Baseline/<br>Day 1 | 4 | 12 | 24 | 36 | 48 <sup>b</sup> | 52 | Every 12<br>Weeks<br>After<br>Week 52 | Withdrawal | Follow-up <sup>d</sup> |
| 12-lead ECG <sup>m</sup> | Х | | | | | | | | | | |
| Adverse events | | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ |
| Serious adverse events | Xn | Χ | Χ | Х | Χ | Χ | Х | Χ | X | Χ | Χ |
| Willingness to Switcho | | Χo | | | | | | | | | |
| HIV TSQ <sup>p</sup> | | Χ | Χ | | Χ | | Х | | | Χ | |
| Symptom Distress Module <sup>p</sup> | | Χ | Χ | | Χ | | Х | | X (every 24 weeks) | Χ | |
| Laboratory Assessments | | | | | | | | | | | |
| Quantitative plasma HIV-1 RNAq | X | Χ | Χ | Χ | Χ | Χ | Χ | | X | Χ | |
| Lymphocyte subset <sup>r</sup> | X | Χ | Χ | Χ | Χ | Χ | Χ | | | Χ | |
| Plasma for storages | Х | Χ | Χ | Χ | Χ | Χ | Χ | | X | Χ | |
| Clinical chemistry <sup>t</sup> | Χ | Χ | Χ | Χ | Χ | Χ | Х | | | Χ | Χ |
| Hematology | Χ | Χ | Χ | Χ | Χ | Χ | Χ | | | Χ | Χ |
| PT/INR (for Child-Pugh) | Χ | | | | | | | | | | |
| Fasting lipids and glucose <sup>u</sup> | | Χ | | | Χ | | Х | | | Χv | |
| Urinalysis and spot urine for protein analysis <sup>w</sup> | | Х | | | Х | | Х | | | Χ | Х |
| Pregnancy test <sup>x, y</sup> | S | U/S <sup>z</sup> | S | S | S | S | S | S | S | S | |
| HBsAg, anti-HBc, Anti-HBs, and HBV DNA <sup>aa</sup> | Х | | | | | | | | | | |
| HCV antibody | Х | | | | | | | | | | |
| RPR | Х | | | | | | | | | | |

| Procedures | g Visita | | | Rande | | Continuation<br>Phase <sup>c</sup> | rawal | pdn- | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening | Baseline/<br>Day 1 | 4 | 12 | 24 | 36 | 48 <sup>b</sup> | 52 | Every 12<br>Weeks<br>After<br>Week 52 | Withdrawal | Follow-up <sup>d</sup> |
| Renal, bone and inflammatory marker analytes (blood/urine) and HbA1c, insulin and glucosebb | | Х | | | Х | | Х | | | Х | |
| Whole Blood (Virology) <sup>∞</sup> | | Х | | | | | Х | | | Х | |
| Whole Blood (Telomere Length)dd | | Х | | | | | Х | | | Xee | |
| PBMCsff | | X | | | Χ | | Χ | | | <b>X</b> 99 | |
| Study Treatment | | | | | | | | | | | |
| IVRS/IWRShh | X | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ |
| Dispense IP | | Х | Χ | Χ | Χ | X | Χ | Χ | Χ | | |
| IP accountability (pill counts) | 20 | | Х | X | Χ | X | Χ | :1.500 | X | X | |

ART - antiretroviral therapy, BMI - body mass index, CDC - centers for disease control and prevention, DNA - deoxyribonucleic acid, ECG - electrocardiogram, eCRF - electronic case report form, HBV - hepatitis B virus, HCV - hepatitis C virus, INR - international normalized ratio, IP - investigational product

- a. As soon as all Screening results are available, randomization may occur.
- b. Participants with plasma HIV-1 RNA ≥50 c/mL at Week 48 (primary endpoint) must have HIV-1 RNA level re-assessed by a second measurement performed 2-4 weeks later, occurring prior to Week 52.
- c. All participants on the DTG/3TC FDC arm who complete through Week 52 will have the opportunity to enter the Continuation Phase. The Continuation Phase is not applicable for participants in Sweden and Denmark. For participants who will not continue past Week 52, do not dispense study intervention. Participants completing the Continuation Phase must return to the clinic for an End of Continuation Phase visit when transitioning to commercial supplies or to an alternate ART regimen, if appropriate. At this visit, conduct study assessments as specified for all Continuation Phase visits except for dispensing study intervention.
- d. An in-clinic Follow-Up visit will be conducted 4 weeks after the last dose of study intervention for participants with the following conditions at the last on-study visit: ongoing AEs, serious adverse events (SAEs) regardless of attributability, and any laboratory abnormalities that are considered to be AEs or potentially harmful to the participant. However, the investigator, in consultation with the medical monitor, should follow-up with the participant until the event is resolved, stabilized, otherwise explained, or the participant is lost to follow-up

- e. Inclusion/exclusion criteria will be assessed fully at the Screening visit. Changes between the Screening visit and the Day 1 visit should be considered to ensure eligibility, including review of additional assessments performed at Day 1. Genotypic resistance testing results if available MUST be provided to ViiV after screening and before randomization.
- f. Full medical history will be conducted prior to randomization and include assessments of cardiovascular, metabolic (e.g., Type I or II diabetes mellitus), psychiatric (e.g., depression), renal (e.g., nephrolithiasis, nephropathy, renal failure), and bone disorders.
- g. Menopause history will include date of last menstrual period (collected at Day 1, Week 52 or withdrawal) and menopausal status (collected at Screening, Week 52 or withdrawal) based on the criteria in the Protocol Section 11.4.1. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause.
- h. Assessment for cardiovascular risk will include height, weight, blood pressure, smoking status and history, pertinent medical conditions (e.g., hypertension, diabetes mellitus), and family history of premature cardiovascular disease. BMI will be calculated within the eCRF.
- i. The same scale should be used to measure body weight at each visit.
- j. Based on the participant's current CDC status in the past 6 months.
- k. On Day 1, the electronic Columbia Suicidality Severity Rating Scale (eC-SSRS), participant completed questionnaire is to be administered prior to the first dose.
- I. Limited physical examination to include blood pressure at Day 1 (recorded in eCRF) for Framingham score assessment. Blood pressure to be measured after resting in a semi-supine position for at least 5 minutes.
- m. A 12-lead ECG will be performed in a semi-supine position after resting for at least 5 minutes.
- n. Only SAEs related to study participation or to a concomitantly administered ViiV/GSK product will be collected between obtaining informed consent and administration of study intervention at Day 1.
- o. Willingness to Switch Survey must be done prior to randomization.
- p. Questionnaire/Surveys are recommended to be administered at the beginning of the visit before any other assessments are conducted. Only conduct questionnaires/surveys at Withdrawal if occurring prior to Week 48, except the Symptom Distress Module which should also be collected if Withdrawal occurs during the Continuation Phase.
- q. See Virologic Withdrawal and Stopping Criteria Section of protocol (Section 7.1.1).
- r. Lymphocyte subset will include collection of CD4 and CD8 for calculation of Cd4:CD8 ratio. CD8 will also be reported to sponsor.
- s. Plasma samples for storage will be collected at each visit starting at Day 1, including unscheduled visits (e.g. for HIV-1 RNA levels and immunological parameters). These samples will be used when needed such as when samples are lost, arrive at the laboratory unevaluable, or for genotypic and/or phenotypic analyses when participants meet Suspected and Confirmed Virologic Withdrawal criteria.
- t. See Protocol Appendix 7 for a list of clinical chemistry labs.
- u. An overnight fast is preferred; however, a minimum of a 6-hour fast is acceptable.
- v. Collect fasting lipids and glucose if the Withdrawal visit occurs at Weeks 24 or 48.
- w. A morning specimen is preferred. To assess renal biomarkers: urine albumin/creatinine ratio; urine protein/creatinine ratio; and urine phosphate.
- x. Women of childbearing potential only. S=serum, U=urine. Pregnancy events will be captured starting at Day 1 following exposure to study intervention.
- y. Remind females of reproductive potential of the need to avoid pregnancy while in study and adherence to the study's contraception requirements.
- z. Local Pregnancy result must be available **prior to randomization** on Day 1. Local serum pregnancy test on Day 1 is allowed if it can be done, and results obtained, within 24 hours **prior to randomization**.
- aa. HBV DNA testing will be performed for participants with positive anti-HBc and negative HBsAg and negative anti-HBs (past and/or current evidence). Participants must return to the clinic to provide a sample for HBV DNA testing prior to randomisation.
- bb. Blood sample for HbA1c, insulin, glucose, renal, bone and inflammation biomarker assessments: **Renal**: Cystatin C, Beta-2-Microglobulin (urine), Retinol Binding Protein (RBP; urine), urine B2M/creatinine ratio, urine RPB/creatinine ratio, urine albumin/creatinine ratio, urine protein/creatinine ratio, urine phosphate, serum creatinine; **Bone**: bone specific

#### **CONFIDENTIAL**

208090

- alkaline phosphatase, procollagen type 1-N-propeptide, type 1 collagen cross-linked C-telopeptide, osteocalcin; **Inflammation:** Interleukin-6 (IL-6), High-sensitivity C reactive protein (hs-CRP), D-dimer, Soluble CD14 (sCD14), Soluble CD163 (sCD163); insulin and glucose for HOMA-IR calculation
- cc. Where local country or laboratory practices allow, whole blood (Virology) may be used for virologic analyses as described in the protocol.
- dd. Where local country or laboratory practices allow, whole blood will be used for telomere length evaluation.
- ee. Collect sample for these assessments ONLY if the Withdrawal visit occurs at Week 48.
- ff. Where local country or laboratory practices allow, PBMC collection samples may be used for virologic analyses as described in Protocol Section 8.10.
- gg. Collect sample only if Withdrawal visit occurs at Weeks 24 or 48.
- hh. At Screening, a subject number will be generated.

# 15.3. Appendix 3: Assessment Windows

Laboratory data, health outcomes, vital signs, e-CSSRS and genotypic and phenotypic data will be assigned to assessment windows according to actual dates rather than the nominal visit labels as recorded on the eCRF or in the laboratory database.

A window around a target Study Day will typically include all days from the midpoints between it and the target Study Days of the previous and the proceeding visits. In general, the nominal target study day for week w is (7\*w)+1.

# 15.3.1. Definitions of Assessment Windows for Analyses

| Analysis Set | Parameter (if | Target | Analysi | s Window | Analysis |
|---|---|---|---|---|---|
| / Domain | applicable) | | Beginning<br>Timepoint | Ending<br>Timepoint | Timepoint |
| Efficacy,<br>Labs and<br>Health<br>outcomes<br>(not collected<br>at Week 52) | Laboratory Assessments<br>(including HIV-1 RNA,<br>lipids and biomarkers),<br>HIVTSQ, SDM | | | | |
| | | -28 | □-4 | □-4 | Screening |
| | | 1 | -3 | 1 | Day 1 |
| | | 29 | 2 | 56 | Week 4 |
| | | 85 | 57 | 126 | Week 12 |
| | | 169 | 127 | 210 | Week 24 |
| | | 253 | 211 | 294 | Week 36 |
| | | 337 | 295 | 378 | Week 48 |
| | | 449 | 379 | 490 | Week 64 |
| | | 7*w+1 | 7*w-41 | 7*w+42 | Week w,<br>w=76, 88, |
| | | Study Day<br>of last dose<br>+ 28 | >Study Day<br>of last dose<br>+1 | >Study Day of last dose +1 | Follow-up |
| Efficacy and<br>Safety Data<br>collected at<br>Week 48 and<br>Week 52) | Weight, BMI, eCSSRS | | | | |
| | | -28 | <b>[]-4</b> | []-4 | Screening |
| | | 1 | -3 | 1 | Day 1 |
| | | 29 | 2 | 56 | Week 4 |
| | | 85 | 57 | 126 | Week 12 |
| | | 169 | 127 | 210 | Week 24 |
| | | 253 | 211 | 294 | Week 36 |

| Analysis Set | Parameter (if | Target | Analysi | Analysis | |
|---|---|---|---|---|---|
| / Domain | omain applicable) | | Beginning<br>Timepoint | Ending<br>Timepoint | Timepoint |
| | | 337 | 295 | 350 | Week 48 |
| | | 365 | 351 | 406 | Week 52 |
| | | 449 | 407 | 490 | Week 64 |
| | | 7*w+1 | 7*w-41 | 7*w+42 | Week w, w= 76, 88, |
| | | Study Day<br>of last dose<br>+ 28 | >Study Day<br>of last dose<br>+1 | >Study Day of last dose +1 | Follow-up |
| | • | • | • | • | |

# 1. NOTES:

- For parameters which are not scheduled to be assessed at particular visits, the all-inclusive windows defined will still be used.
- Assessments at unscheduled visits will be included for 'any time On-treatment' time points and in data listings, as well as algorithms that make use of additional data (e.g., Snapshot).
- In the event a baseline value is missing, the latest pre-dose value prior to baseline will be used, notwithstanding this date occurring more than 3 days prior to baseline.

# 15.4. Appendix 4: Study Phases and Emergent Adverse Events

## 15.4.1. Study Phases

Data collected from both arms up to and including the date of the Week 52 visit will be considered to be during the Randomized Phase of the study.

For subjects randomized to DTG/3TC, data collected after Week 52 will be considered to be during the Continuation Phase of the study. For subjects randomized to the CAR arm, Continuation Phase of the study is not applicable.

| Phase | Randomized<br>Arm | Start | End |
|---|---|---|---|
| Randomized<br>Phase | DTG/3TC | IP start date | Week 52 DOV |
| Filase | | | or Withdrawal date before Week 52 DOV |
| | CAR | Day 1 DOV | Week 52 DOV |
| | | | or Withdrawal date before Week 52 DOV |
| Continuation Phase | DTG/3TC | Week 52<br>DOV+1 | IP end date or Withdrawal date |
| | CAR | Not applicable | Not applicable |

15.4.1.1. Study Phases for for Laboratory, HIV Associated Conditions, Vital Signs, Health Outcomes and Genotypic and Phenotypic Data

| Treatment State | Definition |
|---|---|
| Pre-Treatment | Date ≤ Study Treatment Start Date |
| On-Treatment | Study Treatment Start Date < Date ≤ Study Treatment Stop Date + 1 |
| Post-Treatment | Date > Study Treatment Stop Date +1 |

#### 1. NOTES:

If the study treatment stop date is missing then the assessment will be considered to be On-Treatment

#### 15.4.1.2. Study Phases for Adverse Events

For adverse events, partial AE start date will use imputation as described in Section 15.7.2.1. In the case of a completely missing start date, the event will be considered to have started On-treatment unless an end date for the AE is provided which is before start of study treatment; in such a case the AE is assigned as Pre-treatment.

| Treatment State | Definition |
|---|---|
| Pre-Treatment | AE Start Date < Study Treatment Start Date |
| On-Treatment | If AE onset date is on or after treatment start date & on or before treatment stop date. |
| | Study Treatment Start Date ≤ AE Start Date ≤ Study Treatment Stop Date |
| Post-Treatment | If AE onset date is after the treatment stop date. |
| | AE Start Date > Study Treatment Stop Date |
| Onset Time Since 1st Dose (Days) | If Treatment Start Date > AE Onset Date = AE Onset Date - Treatment Start Date |
| | If Treatment Start Date ≤ AE Onset Date = AE Onset Date - |
| | Treatment Start Date +1 |
| | Missing otherwise. |
| Duration (Days) | AE Resolution Date – AE Onset Date + 1 |
| Drug-related | If relationship is marked 'YES' on eCRF. |

#### NOTES:

- Partial AE start date will use imputation as described in Section 15.7.2.1
- In the case of a completely missing start date, the event will be considered to have started On-treatment
  unless an end date for the AE is provided which is before start of investigational product; in such a case the AE
  is assigned as Pre-treatment.
- If the IP Stop Date is missing, then any event with a start date on or after IP Start Date will be considered to be On-treatment.
- If the start date of the AE is after IP Stop Date but has been recorded as potentially related to IP, then it will be
  classified as On-treatment.

#### 15.4.1.3. Study Phases for Concomitant Medication

- Prior medications: Those taken (i.e., started) before the start date of investigational product.
- Concomitant medications: Those taken (i.e., started or continued) at any time between the start date and stop date of study treatment, inclusive. Prior medications that were continued during this period are also considered as concomitant medications.
- Post treatment medications: Those started after the stop date of study treatment. Concomitant medications that were continued during this period are also considered as post-treatment medications.

It will be assumed that medication has been taken on the date in which it is reported as started or stopped. For any medication starting on the same date as study treatment, it will be assumed that the medication was taken after the subject started taking study treatment.

Duration of episodes of concomitant medication will be calculated as medication stop date – medication start date, so long as the medication is defined as concomitant according to the rules above (and presented below in the scenario matrix). Durations will be left blank if stop date is missing.

ART medications will also be classified as prior to screening, concomitant to screening and/or post-treatment according with the following modifications:

- ART starting on study treatment stop date will be considered as only posttreatment and not concomitant. It is expected that after discontinuation of study treatment, a subject may immediately begin taking another ART.
- ART stopping on study treatment start date will only be considered as prior and not concomitant.
- Any ART entered on the Prior ART eCRF with partial end date will be assumed to have finished before Screening.
- ART stopped prior to screening includes all ART that has stopped prior to screening. All ingredients from any regimen that is switched to another regimen prior to the screening visit e.g. from TDF-based to TAF-based ART will be presented as having stopped.
- ART Medications received at or after Screening includes all ART that is either being received at the screening visit or is introduced at a later date. Note, for CAR patients this could be pre- or post- randomization and for DTG/3TC patients this can be pre-randomization only; at randomization and beyond for DTG/3TC patients, ART is recorded as 'study treatment' and not recorded via ART-specific concomitant medication pages.
- ART Medications Received at Screening includes all ART that is ongoing at the screening visit only.

| | Pre-treatment | | On-treatment | | | Post-treatment | Prior | Concomitant | Post |
|---|---|---|---|---|---|---|---|---|---|
| (a) | X | | | | | | Y | N | N |
| (b) | X | | ———х | | | | Υ | Y | N |
| (c) | X | | | | | ———х | Υ | Y | Υ |
| (d) | | | X | | | | N | Υ | N |
| (e) | | Q) | Χ | a) | 7 | х | N | Υ | Υ |
| (f) | | IP Start Date | | Stop Date | IP Stop Date+1 | X | N | N | Υ |
| (g) | ?x | art | | do | D d | | Υ | N | N |
| (h) | ? | St | х | S. | Sto | | Y* | Υ | N |
| (i) | ? | <u> </u> | | <u> </u> | ₫. | ———х | Υ* | Y* | Υ |
| (j) | X | | | | | ? | Υ | Y** | Y** |
| (k) | | | X | | | ? | N | Υ | Y** |
| (I) | | | | | | x? | N | N | Υ |
| (m) | ? | | | | | ? | Y*** | Y*** | Y*** |
| (n) | X | Х | | | | | Υ | Υ | N |
| (o) | ? | х | | | | | Y* | Υ | N |
| (p) | | Х | ———х | | | | N | Υ | N |
| (q) | | Х | | х | | | N | Y | N |
| (r) | | | | х | | ———х | N | Y | Υ |
| (s) | | | | х | | ? | N | Y | Y** |
| (t) | | | | | х | ———х | N | N | Υ |
| (u) | | | | | х | ? | N | N | Υ |
| (v) | | | Χ | | Х | | N | Y | Υ |

- 1. x = start/stop date of medication
- 2. ? = missing start/stop date of medication
- 3. \* If a medication is stopped On-treatment or Post-treatment and no start date is recorded it will be assumed that the medication was ongoing from the Pre-treatment phase
- 4. \*\* If a medication is started Pre-treatment or On-treatment and no stop date is recorded then usage will be assumed to be ongoing for the remainder of the study
- 5. \*\*\* If a medication has no start or stop date it will be assumed that the medication was ongoing from the Pre-treatment phase to the Post-treatment phase
- 6.

# 15.4.2. Combining Treatment Phases and States

On-treatment and Post-treatment assessments and events will be classified as occurring during the Randomized or Continuation Phase of the study as follow:

- If a subject did not enter the Continuation Phase, then any Post-treatment data will be assigned to the Randomized Phase.
- For subjects who did enter the Continuation Phase, any Post-treatment data will be assigned to the Continuation Phase.

For concomitant medication, if there is a duration overlapping any period then this should be reflected such that a concomitant medication (at time of the data cut):

- Starting and ending before treatment start then phase is set to missing
- Is taken at any point during the randomized phase only then phase is set to "Randomized Phase"
- Is taken at any point during the continuation phase only then phase is set to "Continuation Phase"
- Is taken at any point across the randomized and continuation phases then phase is set to "Randomized and Continuation Phase"

# 15.4.3. Emergent Flag for Adverse Events

| Flag | Definition |
|---|---|
| Emergent | Emergent refers to AE Severity/ Lab toxicity that develops or increases in intensity after baseline |

For adverse events, partial AE start date will use imputation as described in Section 15.7.2.1. In the case of a completely missing start date, the event will be considered to have started On-treatment unless an end date for the AE is provided which is before start of investigational product; in such a case the AE is assigned as Pre-treatment.

For laboratory data, there will be no imputation of dates, which are expected to be fully complete and available in SDTM transfers. Any laboratory dates that are partially missing will be queried.

#### 15.5. **Appendix 5: Data Display Standards & Handling Conventions**

# 15.5.1. Reporting Process

| Software | |
|---|---|
| The currently supporte | ed versions of SAS software and any other statistical reporting software required for the analysis and reporting will be used. |
| Reporting Area | |
| HARP Server | uk1salx00175 |
| HARP Compound | :\ARPROD\GSK3515864\mid208090\reporting_effort_number |
| Analysis Datasets | |
| Analysis datasets will | be created according to CDISC standards (SDTM IG Version 3.2 & ADaM IG Version 1.1 or above) |

- Analysis datasets will be created according to CDISC standards (SDTM IG Version 3.2 & ADaM IG Version 1.1 or above).
- For creation of ADaM datasets (ADCM/ADAE), the same version of dictionary datasets will be implemented as SDTM.

#### **Generation of RTF Files**

RTF files will be generated for all reporting efforts.

# 15.5.2. Reporting Standards

#### General

- The current GSK Statistical Display Standards Library will be applied for reporting, unless otherwise stated (Library Location: https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics
- Do not include subject level listings in the main body of the GSK Clinical Study Report. All subject level listings should be located in the modular appendices as ICH or non-ICH listings
- All data displays will use the term "subjects" rather than "participants".

#### **Formats**

GSK Statistical Display Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.

#### General

- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the GSK Standard statistical Display Principles but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Actual time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to GSK Standard Statistical Display Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.

#### **Unscheduled Visits**

- Unscheduled visits will be assigned to a study visit using the all-inclusive windows defined in Section 15.3.
- However, data summaries will only report visits that are planned assessment time points for each parameter (according to the Time and Events table).
- Assessments at unscheduled visits will be included for 'any time On-treatment' time points and in data listings, as well any algorithms that make use of additional data (e.g., Snapshot).

| 400 01 Manual (0.3.) 011 policy | |
|---|---|
| Descriptive Summary Statistics | |
| Continuous Data | Refer to GSK Standard Statistical Display Principle 6.06.1 |
| Categorical Data N, n, frequency, % | |
| Graphical Displays | |
| Refer to GSK Statistical Display Standard Statistical Principals 7.01 to 7.13. | |

# 15.6. Appendix 6: Derived and Transformed Data

#### 15.6.1. General

#### **Multiple Measurements at One Time Point**

- If there are multiple assessments within Screening window, the last assessment before Day 1 will be used
- If there are multiple assessments within Day 1 window, the latest pre-dose assessment will be used
- With the exception of the Snapshot endpoints, if after window assignment (see Section 15.3), there are multiple valid assessments of a parameter within the same window, then the following hierarchy will be used to determine the value to be used for summary statistics of observed values:
  - the assessment closest to the window target Study Day;
  - if there are multiple assessments equidistant from the target Study Day, then for continuous variables the mean of these values will be used and for categorical variables the worse assessment. For HIV-1 RNA, the geometric mean of the number of copies will be used as opposed to the arithmetic mean
- Assessments not chosen for use in summary statistics by this algorithm will still appear in
  the associated listings. Also, such valid assessments will be used when determining values
  of potential clinical concern for the 'any time On-treatment' time point, and for any algorithm
  that has specific rules for which observation to use (e.g., SNAPSHOT).
- In the event of laboratory re-tests being performed the last re-test in the visit window will be used. For example:
- If a subject had a week 24 viral load and then two re-tests (i.e. three viral loads labeled as week 24, unscheduled 1 unscheduled 2). and the first two viral loads were within the upper bound of the week 24 visit (Day 210) but the last re-test was slotted to week 36 then the last re-test would not be used for the week 24 snapshot.
- If a subject had a week 24 viral load but the re-test was performed on Day 220 (week 36) then the re-test viral load would not be used for the week 24 snapshot.

#### Study Day

- Calculated as the number of days from initial study treatment start date:
  - Ref Date = Missing → Study Day = Missing
  - Ref Date < Treatment Start Date → Study Day = Ref Date Treatment Start Date
  - Ref Data ≥ Treatment Start Date → Study Day = Ref Date (Treatment Start Date) +

Note that Treatment Start Date is considered to be on Study Day 1 and the day before this is Study Day -1; i.e., there is no Study Day 0.

#### Post-baseline

Post-baseline refers to the combined time periods of On-treatment and Post-treatment.
 Post-baseline may be further specified according to phase of the study: Randomized Phase and Continuation Phase.

# **Study Drug**

Study Drug refers to either Investigational Product DTG/3TC or CAR.
## 15.6.2. Study Population

#### **Demographics**

#### Age

- Age, in whole years, will be calculated with respect to the subject's Screening visit where year
  of birth is collected.
- GSK Statistical Display Standard algorithms will be used for calculating age where birth date will be imputed as follows:
  - o For all subjects, the missing date and month will have this imputed as '30th June'.
  - For analysis purposes, if a subject did not fail to meet inclusion criteria #1 (aged 18 years or older), then set any age imputed as <18 by the GSK Statistical Display Standard algorithm to 18. If the subject failed to meet inclusion criteria #1 then the imputed age will not be reset.
- Birth date will be presented in listings as 'YYYY'.
- Completely missing dates of birth will remain as missing, with no imputation applied. Consequently, the age of the subject will not be calculated and will remain missing.

## Framingham Risk Equation

The predicted probability,  $\widehat{p}$ , of having a cardiovascular disease (CVD) within the next 10-years according to the Framingham formula [D'Agostino, 2008] is

for females:

$$\widehat{p}_F = 1 - S_0(t) \exp\{2.32888 \times \log(\text{age}) + 1.20904 \times \log(TC) - 0.70833 \times \log(HDL) + 2.76157 \times \log(SBPu) + 2.82263 \times \log(SBPt) + 0.52873 \times I_S + 0.69154 \times I_d - 26.1931\}.$$

for males:

$$\widehat{p}_{M} = 1 - S_{0}(t) \exp\{3.06117 \times \log(\text{age}) + 1.12370 \times \log(TC) - 0.93263 \times \log(HDL) + 1.93303 \times \log(SBPu) + 1.99881 \times \log(SBPt) + 0.65451 \times I_{S} + 0.57367 \times I_{d} - 23.9802\},$$

where

$$S_0(t) = \begin{cases} 0.95012, \text{ females} \\ 0.88936, \text{ males} \end{cases}$$

TC = total serum cholesterol (mg/dL),

HDL = serum HDL cholesterol (mg/dL),

SBPu = systolic blood pressure (mmHg) if subject is not treated for high blood pressure (note that if a subject is treated for high blood pressure then log(SBPu) = 0)

SBPt = systolic blood pressure (mmHg) if subject is treated for high blood pressure (note that if a subject is not treated for high blood pressure then log(SBPt) = 0)

$$I_s = \begin{cases} 1, & \text{current smo} \text{ ker} \\ 0, & \text{otherwise} \end{cases}$$

$$I_d = \begin{cases} 1, \ diabetic \\ 0, \ otherwise \end{cases}$$

#### **Demographics**

- A subject will be considered as treated for high blood pressure if at Screening/Day 1 visit the subject receives any medication for hypertension (need to check whether any of the terms "HYPERTENSION", "HYPERTENTION", "HIPERTENSION" or similar is included in the description of SDTM.CM.CMINDC variable)
- Smoking status is collected on Screening/Day 1 visit as "Never smoked", "Current smoker", "Former smoker". For "Current smoker"  $I_s$  should be set to 1 and for "Never smoked" and "Former Smoker"  $I_s$  should be set to 0.
- A subject is classified as diabetic if "Current" or "Past" has been selected in the medical history eCRF
  page completed on Screening/Day 1 visit; if "Not assessed" has been selected then the subject will be
  considered diabetic if the subject receives any medication for diabetes on Screening/Day 1 visit (need to
  check whether any of the terms "DIABETES" or "DIABETIC" is included in the description of
  SDTM.CM.CMINDC variable).
- The 10-year probability of CVD will not be calculated for subjects who have indicated "Current "or "Past" myocardial infarction in the medical history eCRF page completed on Screening/Day 1 visit. These subjects will not be included in summary statistics (e.g. mean, sd, median) of 10-year CVD risk in 'Summary of Baseline Cardiovascular Risk Assessments Table', but will be counted in the highest category of risk (i.e. >20%) in the summary by category.

#### Extent of Exposure

- Exposure to DTG/3TC will be calculated from the IP eCRF pages. Exposure to CAR will be calculated from the CONART eCRF pages.
- Subjects who were randomized to DTG/3TC but did not report a IP start date will be categorised
  as having zero days of exposure.
- Subjects who were randomized to CAR but withdrew on Day1 will be categorised as having zero days of exposure
- Missing Treatment Stop Date will be imputed, for purposes of calculating exposure, as the date
  of last visit or the recorded date of withdrawal/completion, whichever is earlier.
- Actual exposure will be calculated where the duration of any dosing interruptions based on eCRF data will be subtracted from the result above.
- The ratio (percentage) of the actual exposure to the overall exposure (i.e. study treatment stop date – study treatment start date+1) will be used to define protocol deviation leading to exclusion from PP Population due to study treatment interruption (i.e. >10%).

#### **Strata**

- For analysis purposes, randomization strata will be used from that derived using eCRF data, even if this differs from the strata captured in IVRS.
- For patients randomized to DTG/3TC, baseline third agent class is collected on the prior ART history form. For patients randomized to current CAR, baseline third agent class is collected on the concomitant ART form.
- Third agent class is identified using terms from the GSK Drug Dictionary

## 15.6.3. Efficacy

#### **HIV-1 RNA**

## **Snapshot**

- It is intended to be primarily a virologic assessment of the endpoint, and as such follows a "virology first" hierarchy.
- Plasma HIV1-RNA < 50 c/mL or plasma HIV1-RNA ≥ 50 c/mL within an analysis window is typically determined by the last available plasma HIV-1 RNA measurement in that window while the subject is On-treatment.
- When no HIV-1 RNA data is available within a window, a subject cannot be classified under HIV1-RNA < 50 c/mL. Depending on the reason for lack of data, the subject will be classified as a HIV1-RNA ≥ 50 c/mL or reported as 'No Virologic Data at Week X'; in the latter case, the algorithm further classifies the nature of the missing data. Typically, a subject withdrawn (i) due to AE or, (ii) for another reason yet was suppressed at the time, will be counted as 'No Virologic Data at Week X'. Should a subject withdraw for reasons other than AE and was not suppressed at the time, they will be a HIV1-RNA ≥ 50 c/mL.</p>
- For each scheduled assessment time, the snapshot response rate for a given threshold (e.g.,
   <50 c/mL) is defined as:</li>

Snapshot Rate= Number of responders in that analysis window
Number of subjects in the analysis population

 Full details of the algorithm, including the handling of special cases, are included in Section 15.11 of note, the date at which the subject 'discontinue/withdrawn from the study' in the Snapshot algorithm is the date of treatment discontinuation, rather than the date of study withdrawal.

## Plasma HIV-1 RNA

- For summaries and analyses which use HIV-1 RNA level as a continuous measure, the logarithm to base 10 of the value will be used.
- HIV-1 RNA results may be provided as censored values, such as <40 or >9,999,999 c/mL. For the purposes of summary statistics, such values will be replaced by the next value beyond the limit of detection, e.g., 39 or 10,000,000 c/mL, respectively, for the given examples. Data listings will show the censored values as provided.
- Qualitive measures (i.e. "target detected" and "target non-detected") may also be provided by
  the laboratory vendor for values <40 c/ml. When a measurement of plasma HIV-1 RNA is below
  the limit of quantification (i.e. 40 c/mL) and is qualitatively observable that will be denoted as a
  "Target Detected" measure, while HIV-1 RNA below the limit of quantification that is not
  qualitatively observable that will be denoted as "Target Not Detected". Any measurements <40
  c/mL characterised as "Target Non-Detected" or "Target Detected" will be captured in the
  database.</li>

Confirmed Virologic Withdrawal (CVW), Suspected Virologic Withdrawal (SVW) and Precautionary Virologic Withdrawal (PVW) and potential Precautionary Virologic Withdrawal (pPVW)

Please refer to the protocol, Section 7.1.1 for more details of the derivation of CVW, PVW, pPVW and SVWs.

#### **HIV-1 RNA**

#### PVW (leading to discontinuation)

- May be met after two consecutive assessments with HIV-1 RNA >=50 and <200 c/mL without an identifiable, non-virologic cause (immunization, illness, nonadherence) and after discussion with Medical Monitor, OR
- Will be met with three consecutive on treatment assessments with HIV-1 RNA >=50 and <200 c/mL</li>

#### pPVW

 Will be met after two consecutive assessments with HIV-1 RNA >=50 and <200 c/mL. The current HIV-1 RNA values <u>must</u> be below 200 c/mL, but the previous HIV-1 RNA can <u>also</u> have been >=200 c/mL

#### <u>SVW</u>

 One assessment with HIV-1 RNA >= 200 c/mL after Day 1 with an immediately prior HIV-1 RNA <50 c/mL.</li>

#### CVW

 One assessment with HIV-1 RNA >= 200 c/mL after Day 1 with an immediately prior HIV-1 RNA >=50 c/mL

#### **General Considerations**

- The subsequent HIV-1 RNA sample taken after SVW will be used for the determination of CVW.
- Based on the protocol specific conditions outlined in the protocol, derivation of SVW and CVW will
  use nominal visits and unscheduled visits.
- Visit windowing will not be applied.
- The condition of 2-4 weeks between the suspected and confirmatory re-test (as described in protocol Section 7.1) will not be used when programmatically identifying CVW.
- A patient can only be classified as CVW for the analyses if the patient has not withdrawn IP at the
  time of the HIV-RNA re-test value (at CVW value), where Treatment Start < HIV-1 RNA sample date</li>
   = Treatment Stop Date + 1 (if Treatment Stop date exists). Note: study drug interruptions will not
  be taken into account when programmatically identifying CVW.
- Similarly, viral loads above criteria cut-offs resulting in SVW, CVW, PVW and pPVW need to have occurred post-Day 1 in order for the criteria to be met. For example an SVW can occur at Week 4 if Week 4 HIV-1 RNA >=200 i.e. the viral load above SVW criterion occurred post-Day 1.
- Additional guidelines specified in the protocol related to patient management only and will not be taken into account when programmatically identifying CVW.
- The SVW can become a pPVW, and then later a PVW, if the confirmatory viral loads are between 50 and 200 c/mL
- Please refer to Section 7.1.1 of the protocol for details of the derivation.

#### CDC HIV-1 Classification and HIV-associated conditions

 HIV associated conditions will be assessed according to the 2014 CDC Revised Classification System for HIV Infection in Adults (see protocol Section 11.12).

#### **HIV-1 RNA**

 Any 'other' conditions reported in the eCRFs will be identified programmatically before being sent for clinical review to determine whether they should be classed as stage 3 associated conditions. Review will be ongoing and as a minimum will take place prior to each reporting effort.

#### 15.6.4. Safety

#### **Extent of Exposure**

 Exposure to DTG/3TC will be calculated from the IP eCRF pages. Exposure to CAR will be calculated from the CONART eCRF pages. Number of days of exposure to study drug will be calculated as:

Duration of Exposure in Days = (Treatment Stop Date –Treatment Start Date) + 1

For subjects randomized to DTG/3TC or CAR at Day 1:

- For Randomized Phase:
  - For patients completing the Randomized Phase Exposure = IP Start Date to (Week 52 DOV -1)
  - If a subject discontinues prior to Week 52, the IP Stop Date recorded in the eCRF will be used. A partial or missing IP stop date is handled as described in Section 15.7.2.1.
  - o A Day 1 Date of Visit will be used for partial or missing IP start date.
- The overall exposure is calculated as
  - Exposure = IP Stop Date IP Start Date + 1
- Duration of dosing in subject years will be calculated as the sum of subject duration of dosing in days (across all subjects)/365.25
- Subjects who were randomized to DTG/3TC but did not report a IP start date will be categorised
  as having zero days of exposure.
- Subjects who were randomized to CAR but withdrew on Day1 will be categorised as having zero days of exposure.
- Missing Treatment Stop Date will be imputed, for purposes of calculating exposure, as the date
  of last visit or the recorded date of withdrawal/completion, whichever is earlier.
- An alternative calculation of exposure will be performed where the duration of any dosing interruptions based on eCRF data will be subtracted from the result above.
- The ratio (percentage) of the actual exposure to the overall exposure (i.e. study treatment stop date – study treatment start date+1) will be used to define protocol deviation leading to exclusion from PP Population due to study treatment interruption (i.e. >10%).

#### **Adverse Events**

#### AE Severity - DAIDS Grading

 The DAIDS grading (VERSION 2.1, March 2017) for severity of clinical adverse events will be performed.

#### **Extent of Exposure**

See protocol for DAIDS grading criteria.

#### **Adverse Events of Special Interest (AESI)**

The preferred terms for each AESI will be review by safety and clinical team and updated before each formal analysis in a separate document. The following table below shows the AESI categories.

#### **AESI**

Anxiety

Depression and hypomania

Drug Hypersensitivity

Insomnia

Nightmare/Abnormal Dreams

Rash

Sleep disorder

Suicidality and self-injury

## **Laboratory Parameters**

- Additional non-protocol specified laboratory assessments performed at the institution's local laboratory that are databased will not be included in the listings or analyses/summaries. All analyses will be based on central laboratory assessments only. If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of significant digits in the observed values will be used to determine how much to add or subtract in order to impute the corresponding numeric value.
  - Example 1: 2 Significant Digits = '< x ' becomes x 0.01
  - Example 2: 1 Significant Digit = '> x' becomes x + 0.1
  - Example 3: 0 Significant Digits = '< x' becomes x 1

#### Lab Toxicities - DAIDS Grading

- Toxicities will be based on the Division of AIDS (DAIDS) grading system, as specified in the protocol.
- Toxicity grades provided by the central laboratory do not distinguish between abnormally high or low criteria, when both are relevant for a particular parameter.
- When summarising toxicity grades for such parameters, they will be categorised as to whether they are above or below the midpoint of normal range.

| Parameter | Below Midpoint | Above Midpoint |
|----------------|----------------|----------------|
| Calcium | Hypocalcaemia | Hypercalcaemia |
| Fasted glucose | Hypoglycaemia | Hyperglycaemia |
| Sodium | Hyponatremia | Hypernatremia |
| Potassium | Hypokalemia | Hyperkalemia |

## **Lipid-Modifying Agents**

- The following ATC codes correspond to lipid-modifying agents:
  - o ATC Level 2: C10
  - ATC Level 3: C10A, C10B (if Level 2 is not available)

#### **Laboratory Parameters**

- ATC Level 4: C10AA, C10AB, C10AC, C10AD, C10AX, C10BA, C10BX (if level 2, 3 are not available)
- Subjects are considered to have used a lipid modifying agent at baseline if they were taking the
  medication at the time of their baseline laboratory assessment or if they stopped their lipid
  modifying medication within 12 weeks of their baseline lipid testing date.

## National Cholesterol Education Program (NCEP) Lipids Categories

• In addition to DAIDS toxicity scales (see protocol), lipid values will be categorized according to the 2001 NCEP Adult Lipid Guidelines [Grundy, 2001].

| Parameter | Value Range<br>(mmol/L) | Value Range<br>(mg/dL) | Category |
|---|---|---|---|
| Triglycerides | <1.70 | <150 | Normal |
| | 1.70 to <2.26 | 150 to <200 | Borderline High |
| | 2.26 to <5.65 | 200 to <500 | High |
| | ≥5.65 | ≥500 | Very High |
| Total Cholesterol | <5.18 | <200 | Desirable |
| | 5.18 to <6.21 | 200 to <240 | Borderline High |
| | ≥6.21 | ≥240 | High |
| HDL Cholesterol | <1.04 | <40 | Low |
| | 1.04 to <1.56 | 40 to <60 | Normal |
| | ≥1.56 | ≥60 | High |
| LDL Cholesterol | <2.59 | <100 | Optimal |
| | 2.59 to <3.37 | 100 to <130 | Near/Above Optimal |
| | 3.37 to <4.14 | 130 to <160 | Borderline High |
| | 4.14 to <4.92 | 160 to <190 | High |
| | ≥4.92 | ≥190 | Very High |

#### Total Cholesterol / HDL Cholesterol Ratio

 When both total cholesterol and HDL cholesterol results are available from the same date for a subject, then the ratio will be calculated by dividing the total cholesterol result by the HDL cholesterol result. The ratio can be classified as follows:

| Parameter | Value Range |
|-------------------------------|--------------|
| Total Cholesterol / HDL Ratio | < 3.5 |
| | 3.5 to < 4.4 |
| | 4.4 to < 5 |
| | ≥5 |

#### Glomerular Filtration Rate (GFR)

Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation [Levey et al.] will be
used by the central laboratory to provide an estimate of GFR, in mL/min per 1.73 m2, as follows
for the CKD-EPI creatinine equation:

$$GFR = 141 \times min \left(\frac{CRT_{mg/dL}}{\kappa}, 1\right)^{\alpha} \times max \left(\frac{CRT_{mg/dL}}{\kappa}, 1\right)^{-1.209} \times 0.993^{Age} \times [1.018 \text{ if Female}] \times [1.159 \text{ if Black}]$$

#### **Laboratory Parameters**

where age (in years) is at time of assessment,  $\kappa$  = 0.7 if female or 0.9 if male,  $\alpha$  = -0.329 if female and -0.411 if male, min() indicates the minimum of CRT/ $\kappa$  or 1, max() indicates the maximum of CRT/ $\kappa$  or 1, and CRTmg/dL is serum creatinine concentration in mg/dL. The serum creatinine concentration in mg/dL is obtained from GSK standard units of  $\mu$ mol/L as CRTmg/dL =0.0113x CRT $\mu$ mol/L.

#### **CKD-EPI Cystatin C Equation (2012)**

The following will be used for the CKD-EPI Cystatin C Equation:
eGFR = 133 x min(Scys/0.8, 1)-0.499 x max (Scys/0.8, 1)-1.328 x 0.996Age x 0.932 [if female]
Abbreviations / Units
eGFR (estimated glomerular filtration rate) = mL/min/1.73 m2
Scys (standardized serum cystatin C) = mg/l
min = indicates the minimum of Scys/0.8 or 1
max = indicates the maximum of Scys/0.8 or 1
age = years
Assays

#### **Hepatitis Status**

- Hepatitis C status will be determined using antibody (IgM or IgG) and/or hepatitis C virus (HCV)
   RNA assessments performed during screening.
- If both antibody and virus RNA assessments are available, then the latter will take precedence and positive/negative status will be based on whether HCV RNA is detectable (i.e., ≥43 IU/mL [≥1.63 log IU/mL]) or not
- Antibody (IgM or IgG) status with 'BORDERLINE' or 'REACTIVE' will be considered Positive
- A subject will be considered positive for hepatitis B virus (HBV) if they have a positive surface
  antigen or detectable HBV DNA result during screening. Subjects positive for HBV are not
  allowed to enter the study.

#### BMI

BMI classification is based on standard categories adopted by the WHO and FDA:

Underweight = BMI of < 18.5 kg/m2

Normal = BMI of 18.5 - 24.99 kg/m2

Overweight = BMI of 25 - 29.99 kg/m2

Obese = BMI of  $\geq$  30 kg/m2

#### **Other Safety Endpoints**

## Columbia Suicide Severity Rating Scale (C-SSRS)

- Missing data will not have any imputation performed.
- A positive alert is triggered if a subject has reported suicidal ideation/behaviour in categories 4-9.
- Questions in categories 3-5 will be triggered if suicidal ideation is reported in categories 1 or/and 2.
- Incomplete calls:
  - when no complete call is databased on the same day, the data from the incomplete call will be used
  - if a subject has only an incomplete call, and it resulted in a positive alert, the relevant pages in the eCRF should be completed, even though the call was incomplete
  - o when a complete call is databased on the same day, the data from the complete call will be used in the summaries.
- Duplicate calls, if they occur on the same day:
  - Both calls will be reported in the listings.
  - For summary tables, the entry with latest time record will be used.
  - o For summary tables at baseline, unscheduled repeat visits will not be summarised.
  - Relevant eCRF pages will be completed based on the latest entry (if it was a positive alert).
- Late Day 1 assessments
  - Late DAY 1 assessments will be summarised as representing baseline status (i.e., treated as true DAY 1 assessments). Where this leads to multiple DAY 1 assessments, 'complete' assessments will be used over 'incomplete' assessments to represent baseline status. Such assessments will be considered DAY 1 if they occur by Day 14.
- Day 1 assessments performed at later visits
  - DAY 1 assessments on (or close to) study day 1 will be accepted as DAY 1
    assessments (as above). For DAY 1 assessments performed at later visits, the
    'Lifetime' assessment observation will not be summarised but the 'Within the past 2
    months' assessment will be used as a surrogate for the later post-baseline visit
    assessment.

#### Homeostatic model assessment-Insulin Resistance (HOMA-IR)

- HOMA-IR = (fasting plasma insulin (mU/L) \* fasting plasma glucose (mmol/L)) / 22.5.
- HOMA-IR categories will be categorised as follows:
  - o <2
  - o 2 to <3
  - o 3 to <4
  - o >=4

All HOMA-IR analyses will be based on fasting values and only patients with post-baseline values will be included in analyses (i.e. patients with missing post-baseline HOMA-IR will not be included in summary tables or figures). Additionally, patients who are diabetic as captured on the medical history form at screening will be excluded from all HOMA-IR analyses. Finally, any patient who has taken an anti-diabetic medication (ATC code "A10" (DRUGS USED IN DIABETES)) as captured on the medical history form up to screening will be removed from the analysis.

## 15.6.5. Viral Genotyping and Phenotyping

## Genotype

## **Amino Acid Changes**

- A mutation is considered present whenever the encoded amino acid residue differs from the amino acid that would have been encoded by the wild-type (e.g., HXB2, NL43) comparator gene; e.g., Q148K.
- If the encoded amino acid is seen as a mixture of wild-type and mutant amino acid, e.g., Q148Q/K, the mutated amino acid is considered present at the codon of interest.
- If the encoded amino acid is seen as a mixture of two or more amino acids, which may or may
  not include wild type, e.g., Q184K/H or Q184K/H/Q, etc., for the purposes of calculating the
  number of mutated amino acids, only one mutation is considered to be present at the codon of
  interest.

#### **Representation of Amino Acid Changes**

| Mutations | Amino acid change |
|---|---|
| T69S | Single mutation from amino acid 'T' (vendor reference) to 'S' (sample) at codon '69' |
| Q148H/K/R | Mixture of amino acid mutations 'H', 'K' and 'R' (sample) from amino acid 'Q' |
| | (vendor reference) at codon '148' |
| _69_1T | First insertion of amino acid 'T' (sample) at codon '69' |
| _69_2S | Second insertion of amino acid 'S' (sample) at codon '69' |
| _69_3S/A | Third insertion of a mixture of amino acids 'S' and 'A' (sample) at codon '69' |
| L74L/- | Mixture of amino acid 'L' (sample) and a deletion at codon '74' |
| V75- | Single deletion of amino acid (sample) at codon '75' |

#### **Resistance Associated Mutations**

Known INI mutations associated with the development of resistance to RAL, EVG, BIC or DTG:

| Analysis Q148H/K/R, V151I/L/A, S153F/Y, N155H/S/T, E157Q, G163R/K, S230R, R263K, L68V/I*, L74I*, E138T*, V151I*, G193E* |
|---|
|---|

#### NOTES:

- Current listing includes INSTI mutations identified via the Stanford HIV Resistance database, or identified
  during in vitro passage of DTG\*, or as seen in a previous DTG studies in INI-experienced subjects\* (i.e.
  ING112574) and may be modified in case of additional substantive data availability. This table is updated
  only by Virologists.
- INI mutations listed taken from Stanford HIV Resistance Database (http://hivdb.stanford.edu/DR/cgi-bin/rules\_scores\_hivdb.cgi?class=INI cited 25 Oct 2019) and accessed on 28Oct/2020.
- Each INI mutation listed had a score of ≥15. INI substitutions listed above in bold had a score for EVG or RAL of =60.
- Major resistance mutations to other classes (i.e., NRTI, NNRTI, PI) as defined by the International Antiviral Society-USA (IAS-USA). The most up to date IAS-USA guidelines available at the time of DBF will be used in the analysis.

#### Genotype

## **Amino Acid Changes**

| Class | Mutations |
|---|---|
| NRTIs | M41L, A62V, K65R/E/N, D67N, 69 insert, K70E/R, L74V, V75I, F77L, Y115F, F116Y, Q151M, M184V/I, L210W, T215Y/F, K219Q/E |
| NNRTIs | L100I, K101E/P, K103N/S, V106A/M, V108I, E138/A/G/K/Q/R, V179L, Y181C/I/V, Y188C/L/H, G190S/A, H221Y, P225H, F227C, M230I/L, |
| Pls | D30N, V32I, M46I/L, I47A/V, G48V, I50V/L, I54M/L/V, Q58E, T74P, L76V, |
| | V82A/T/F/L/S, N83D, I84V, N88S, L90M |

Note: List generated from IAS\_USA Guideline, - 2019 Drug Resistance Mutations Update Volume 27, Issue 3, September /October 2019

#### **Susceptibility Scores**

## Stanford Genotypic Susceptibility Score (S-GSS)

- To establish genotypic susceptibility to ART treatment, a genotypic sensitivity score will be calculated.
- Genotypic sensitivity to each drug will be assessed using the HIVdb, the Integrated Genotypic Resistance Interpretation System [Liu, 2006].
- In the Stanford HIVdb system, each HIV-1 drug resistance mutation is assigned a drug penalty score. Also, for combination of specific mutations an extra penalty is assigned. The penalty scores for each drug resistance mutation and for combination of drug resistance mutations at different positions within each genomic region are available here

NNRTI: https://hivdb.stanford.edu/dr-summary/mut-scores/NNRTI/NRTI: https://hivdb.stanford.edu/dr-summary/mut-scores/NRTI/

PI: https://hivdb.stanford.edu/dr-summary/mut-scores/PI/

INSTI: https://hivdb.stanford.edu/dr-summary/mut-scores/INSTI/.

- Any mutations that are not included the Stanford database will contribute 0 to the GSS calculations.
- The drug resistance estimate is obtained by adding together the penalty scores from all mutations
  associated with resistance to that drug and by adding also the penalty for combinations of certain
  mutations, if present, and then a numeric score (S-GSS) is applied for each drug as shown in the Table
  below.
- When there's a mixture of two or more mutations at the same position, the mutation associated with the largest penalty is scored.
- The HIVdb S-GSS will be calculated for all subjects with genotypic data at all time points from when
  genotypic data are available for all drugs in the Stanford database. However, Tables will report S-GSS
  scores only for drugs that have been taken by at least one subject during the study. Listings will report S-GSS scores for all drugs in the Stanford database.
- Examples

<u>Example 1:</u> Assume a subject at a specific time point has the INSTI mutations G140S and Q148H. The following Table shows the calculation of drug resistance estimate score for drugs DTG and EVG.

| Genotype | | |
|----------------------------|-----------------|----------|
| Amino Acid Changes | no Acid Changes | |
| | Penalt | y Scores |
| INSTI mutations | DTG | EVG |
| G140S | 10 | 30 |
| Q148H | 25 | 60 |
| G140S + Q148H | 10 | 0 |
| Total | 45 | 90 |
| (drug resistance estimate) | | |

For DTG, mutation G140S has a penalty score of 10, mutation Q148H has a penalty score of 25. One need also to account for the penalty score for the combination of the two mutations which is 10. The sum of all penalties scores gives the drug resistance estimate score which is 45 in this case. Similar calculation for EVG applies.

<u>Example 2:</u> Assume a subject at a specific time point has the INSTI mutations: G140A/C/S (i.e. recorded as G140A, G140C and G140S in SDTM.PF) and Q148H/K/R. The following Table shows the calculation of drug resistance estimate score for DTG.

| | DTG | |
|---|---|---|
| | Individual Mutation | Penalty scores used for drug |
| INSTI mutations | Penalty Score | resistance calculation |
| G140A | 10 | |
| G140C | 10 | 10 |
| G140S | 10 | |
| Q148H | 25 | |
| Q148K | 30 | 30 |
| Q148R | 25 | |
| G140A/C/S + Q148H/K/R | 10 | 10 |
| Total | | 50 |
| (drug resistance estimate) | | |

For mixture of mutations at the same position, the mutation associated with the largest penalty is used, hence for Q148H/K/R the penalty score of 30 for Q148K is used. For G140A/C/S all mutations have the same score 10 so, 10 is used. The penalty score for the combination of mutations at codon positions 140 and 148 is 10. The sum of the three penalties scores gives the drug resistance estimate score which is 50.

 Scores for particular patterns of INSTI, NNRTI, NRTI and PI mutations have been calculated and are readily available here

NNRTI: https://hivdb.stanford.edu/dr-summary/pattern-scores/NNRTI/

 $NRTI: \ https://hivdb.stanford.edu/dr-summary/pattern-scores/NRTI/$ 

PI: https://hivdb.stanford.edu/dr-summary/pattern-scores/PI/

INSTI: https://hivdb.stanford.edu/dr-summary/pattern-scores/INSTI/

The drug resistance estimate is obtained by adding together the penalty scores from all
mutations associated with resistance to that drug and then a numeric score (S-GSS) is applied
for each drug as shown below. Any mutations that are not included the Stanford database will
contribute 0 to the GSS calculations. When there's a mixture of two or more mutations at the

#### Genotype

#### **Amino Acid Changes**

same position, the mutation associated with the largest penalty is scored. The sum scores are titrated to fall within the following ranges: susceptible, potential low-level resistance, low-level resistance, intermediate resistance, and high-level resistance (see table below).

•



 The HIVdb GSS will then be calculated for each subject defined as the sum of the resistance scores for each of their background drugs.

## Monogram Genotypic Susceptibility Score (M-GSS)

- Genotypic sensitivity to each drug will be assigned using the Monogram resistance score and will be reported in a listing for all drugs where Monogram resistance score is available in the database.
- Assays PSGT, GSIN, PSGTIN denote Genotypic Sensitivity as 'Sensitive' or 'Resistance' whereas assay GSARC as 'Sensitive', 'Resistance Possible' or 'Resistance'.
- Genotypic Sensitivity provided by Monogram based on assays PSGT, GSIN, PSGTIN is translated to a Genotypic Sensitivity Score (M-GSS) according to the table below.
- For the DTG/3TC arm a subject might have a M-GSS score of 0, 1 or 2, and in the CAR arm a subject might have a M-GSS score of 0, 1, 2, or 3 (since CAR is a 3-drug regimen).

| Sensitivity |
|-------------|

#### Phenotype

#### Phenotypic Susceptibility Scores (PSS)

- Phenotypic susceptibility to all licensed antiretroviral drugs and DTG will be determined using PhenoSense HIV
  assays from Monogram Inc. and will be reported as fold change (FC) in IC50 relative to wild-type control virus NL43, i.e., FC of sample virus = IC50 of sample virus/IC50 of control virus.
- Since the maximum assay limit for FC for each ART varies from subject to subject, FC values that are greater than the maximum assay limit (e.g., '>100') will be interpreted as having a value equal to the smallest maximum assay limit for that ART in the study population for data analysis. Censored values will be presented 'as is' in the listings.
- Phenotypic susceptibilities will be categorised according to FC (based on Monogram PhenoSense assay). Clinical
  cut-offs (where available) or biological cut-offs by PhenoSense will be used to define the phenotypic susceptibility
  of background treatment.
- Replication capacity is generated as part of standard phenotypic assays.

## Phenotype

To establish susceptibility to background treatment, a phenotypic sensitivity score will be calculated.
Phenotypic susceptibility to each drug in a subject's background regimen will be determined by
applying drug-associated cutoffs as defined by the PhenoSense algorithm to the phenotypic fold
resistance to that drug at a certain timepoint (e.g., Screening or Baseline). A numeric score will be
assigned to each background drug using two different methods: one with full sensitivity only (PSSf) and
one with partial sensitivity included (PSSp).

#### **PSS with Full Sensitivity Only (PSSf)**

| Fold Change | Score | Interpretation |
|--------------------------------------------|-------|----------------|
| > clinical lower cutoff or biologic cutoff | CCI | |
| clinical lower cutoff or biologic cutoff | | |

## **PSS with Partial Sensitivity Included (PSSp)**

| Fold Change | Score | Interpretation |
|---|---|---|
| > clinical higher cutoff | CCI | |
| ≤ clinical higher cutoff and > clinical lower cutoff | | |
| ≤ clinical lower cutoff | | |

• Both PSSf and PSSp will be calculated separately for each subject defined as the sum of the resistance scores for each background drug.

| Drug | Abbreviation | Class | PhenoSense cutoff |
|-----------------|--------------|-------|-------------------|
| Abacavir | ABC | NRTI | $(4.5 - 6.5)^a$ |
| Lamivudine | 3TC | NRTI | 3.5 a |
| Didanosine | ddl | NRTI | (1.3 – 2.2) a |
| Stavudine | d4T | NRTI | 1.7 a |
| Zidovudine | AZT (ZDV) | NRTI | 1.9 |
| Emtricitabine | FTC | NRTI | 3.5 |
| Tenofovir | TDF | NRTI | (1.4 – 4) a |
| Delavirdine | DLV | NNRTI | 6.2 |
| Efavirenz | EFV | NNRTI | 3 |
| Nevirapine | NVP | NNRTI | 4.5 |
| Etravirine | ETR | NNRTI | (2.9-10) a |
| Rilpivirine | RPV | NNRTI | 2.0 |
| Fosamprenavir/r | FPV/r | PI | (4-11) a |
| Atazanavir/r | ATV/r | PI | 5.2 a |
| Indinavir/r | IDV/r | PI | 10 a |
| Lopinavir/r | LPV/r | PI | (9 – 55) a |
| Nelfinavir | NFV | PI | 3.6 |
| Saquinavir/r | SQV/r | PI | (2.3 – 12) a |

| Phenotype | | | |
|--------------------------|---------------------------|-----|-------------|
| Tipranavir/r | TPV/r | PI | (2 – 8) a |
| Darunavir/r | DRV/r | Pl | (10 – 90) a |
| Ritonavir | RTV | Pl | 2.5 |
| Enfuvirtide | T20 | Fl | 6.48 |
| Raltegravir | RAL | INI | 1.5 |
| Elvitegravir | EVG | INI | 2.5 |
| Dolutegravir | DTG | INI | (4-13) a |
| Bictegravir | BIC | INI | (2.5-10) |
| a clinical cutoff (lower | r cutoff – higher cutoff) | · | |

## Phenotypic Susceptibility Score (PSS)

## Net Assessment and Overall susceptibility of ARTs

- Net assessment is an assessment of antiviral activity of ARTs using both genotypic and phenotypic test results interpreted through a proprietary algorithm (from Monogram Biosciences) and provides the overall susceptibility of the drug (Note: partially sensitive and resistant calls are considered resistant in this analysis).
- For determining overall susceptibility of ARTs (OSS), a binary scoring system (0= color), 1=colors) for each antiretroviral agent was used and will be provided in the Monogram dataset. OSS will be calculated as the sum of the net assessment scores of ARTs comprising the subject's ART and categorised as 0, 1, 2, or 3. OSS values will be calculated only for the time of CVW when net assessment is available.

#### **Phenotype**

#### Decision tree approach for Monogram resistance data analyses

- We might have resistance data that come from mixed datasets: PSGT, PSIN, GSIN (primary assays)
   vs PSGT+IN (secondary assay)
- If one of the primary assay does not work for a specific timepoint, we might report the secondary assay if data is available. If all primary assays for a specific timepoint work then we report primary. For example, for baseline if the same assay section (PSGT, PSIN, GSIN) worked then we report primary. If at least one of PSGT or PSIN or GSIN didn't work then we report secondary PSGT+IN.
- Secondary assay testing results might not always be available.

#### **Background:**

- PSGT provides both geno and pheno data for PRO/RT (NRTI and NNRTI) only, with pheno
  including PRO/RT Replication Capacity (RC)
- PSIN Provides pheno data on Integrase only, with pheno including IN RC
- GSIN Provides geno data on Integrase only, This assay provides NO RC data.
- PSGT+IN Secondary assay used if PSGT or GSIN assay fails; it provides both geno and pheno data on PRO, RT and Integrase
- If one of the primary assays does not work for a specific timepoint, we might report the data from the secondary assay, if available. If all primary assays for a specific timepoint work, then we use the data from the primary assays, as secondary assay analysis is not performed. If at least one of PSGT or PSIN or GSIN haven't worked for a specific time point (e.g. Baseline, CVF or time of switch from DTG + 3TC FDC), then we use data from the secondary PSGT+IN and the data from any primary assay that worked from this time point are ignored.
- Secondary assay testing results might not always be available.
- The decision tree algorithm will be used for data summaries in Tables. Listings will report all data from all assays that worked at a specific time point.
- For examples please refer to decision tree below.

#### **Table Symbol Key:**

Y = assay test successful N = assay test failure 2<sup>nd</sup> = back up test performed **bold** = assay to use for analysis

#### How to make decisions:

<u>Scenario 1</u>: if primary PSGT, PSIN and GSIN assays all work for both Baseline and CVF or at time to switch due to Baseline resistance mutations samples, then PSGT+IN assay will not be performed and no PSGT+IN data should be generated.

| Assays | Baseline | CVF or Switch |
|--------|----------|---------------|
| PSGT | Υ | Υ |
| PSIN | Υ | Υ |
| GSIN | Υ | Υ |

#### Phenotype

Scenario 2: If PSGT, PSIN and GSIN all work for Baseline sample; PSGT works for CVF or at time of Switch sample but PSIN and GSIN fail, while PSGT+IN works, then use PSGT+IN (PR, RT and INSTI) for CVF/Switch and a PSGT, PSIN, GSIN for Baseline; do not use PSGT data at CVF/Switch.

| Assays | Baseline | CVF or Switch |
|-------------------------|----------|---------------|
| PSGT | Υ | Υ |
| PSIN | Υ | N |
| GSIN | Υ | N |
| 2 <sup>nd</sup> PSGT+IN | - | Υ |

Scenario 3: If PSGT works for Baseline, but PSIN and GSIN fail, then secondary PSGT+IN assay will be performed on Baseline sample. Similarly, if PSGT works for CVF or switch sample but PSIN and GSIN fail to work, in this scenario, use data generated from PSGT+IN assay on both Baseline and CVF/switch sample for analyses, regardless of obtained PSGT assay data. Same is the case if PSGT fails in both time points and PSIN and GSIN do not fail; the data from PSGT+IN from both time points will be used.

| Assays | Baseline | CVF or Switch |
|-------------------------|----------|---------------|
| PSGT | Υ | Υ |
| PSIN | N | N |
| GSIN | N | N |
| 2 <sup>nd</sup> PSGT+IN | Υ | Υ |

<u>Scenario 4</u>: If PSGT works but GSIN and PSIN both fail on Baseline sample, then 2<sup>nd</sup> PSGT+IN assay might be performed. If PSGT, PSIN and GSIN all work for CVF or Switch sample, then use Baseline PSGT+IN data from Baseline, regardless of PSGT Baseline data.

| Assays | Baseline | CVF or Switch |
|-------------------------|----------|---------------|
| PSGT | Υ | Υ |
| PSIN | N | Υ |
| GSIN | N | Υ |
| 2 <sup>nd</sup> PSGT+IN | Υ | - |

#### 15.6.6. Health Outcomes



#### **Treatment Satisfaction Score**

- Total Treatment Satisfaction Score is computed with items 1-10. Items 1-10 are summed to produce a score with a possible range of 0 to 60.
- Higher scores represent greater treatment satisfaction as compared to the past few weeks.
- A maximum of 5 items can be missing, which can be imputed to reflect the mean of the completed item scores. If 6 or more items are missing, then the treatment satisfaction scale score should not be computed.
- General Satisfaction/Clinical sub-score is computed with items and and . These items are summed to produce a score with possible range of 0 to 30
- Lifestyle/ease sub-score is computed with items and and and are summed to produce a score with possible range of 0 to 30.

#### **Individual Item Scores**

- Items are rated as 6 (very satisfied, convenient, flexible, etc.) to 0 (convenient)
- Higher scores represent greater satisfaction with each aspect of treatment
- For individual item scores outputs, missing scores will not be computed (according to Page 7 of the [HIVTSQ User Guidelines]).
- If multiple assessments equidistant from the target Study Day, the assessments with worst score will be used.

| Symptom Distress Module |
|---|
| Questionnaire (Questions 1-20 are scored CCI) CCI - This section contained Clinical Outcome Assessment data collection questionnaires or indices, which are protected by third party |
| CCI - This section contained Clinical Outcome Assessment data collection questionnaires or indices, which are protected by third party copyright laws and therefore have been excluded. |
| copyright laws and therefore have been excluded. |

- The Symptom Distress Module (also referred to as HIV Symptom Index) is a 20-item selfreported measure that addresses the presence and perceived distress linked to symptoms commonly associated with HIV or its treatment.
- The aggregate scores are derived from the individual scores:
  - symptom count: unweighted sum of the number of symptoms which are present;
  - symptom bother score: unweighted sum of the bother item scores for each symptom.
- These aggregate scores are considered assessable only if less than 10% of the symptom items
   (i.e. one or two symptom items) are missing. The missing items are then considered as the "I do
   not have this symptom" option as this would be interpreted as the symptom was either not
   applicable or unimportant to the subject.
- If more than two symptoms are missing, the aggregated scores (symptom bother score and symptom count) are set to missing.
- If multiple assessments equidistant from the target Study Day, the assessments with worst score will be used.

#### Symptom count

- The "symptom count" based on which of the 20 symptoms were present in the subject.
- The symptom count ranges from 0 to 20.

#### Symptom bother score

- The symptom bother score ranges from 0 to 80.
- If the subject ticked CCI This section contained Clinical, the bother score is 0
- If the subject gave a bother rating, then it is based on ranging from 1 CCI This section (CCI This section).

#### **Symptom Distress Module**

• If the subject ticked two boxes, the worst case is considered. In particular, if the option "I do not have this symptom" is ticked conjointly with a bother rating, the bother score is defined according to the bother rating.

#### Willingness to switch survey

## **Questionnaire (Questions 1-7)**

CCI - This section contained Clinical Outcome Assessment data collection questionnaires or indices, which are protected by third party copyright laws and therefore have been excluded.

- Assess the reason(s) for their participation and facilitate an understanding of subject's willingness to switch
- A single item question prior to randomisation.
- 7 reasons for willingness to participate in a clinical study where the current HIV medication may be switched check all that apply
- Any missing values will remain missing

## 15.6.7. Cut-off date for protocol deviations

#### **Cut-off date**

The following rules should be used to calculate cut-off date for protocol deviations up to and including Week 24:

- For subjects who have Week 24 viral load date (cut-off 1):
  - cut-off = Week 24 viral load date (used for snapshot algorithm) from LB (laboratory) dataset, or date of re-test date if patient had a re-test
- For subjects who do not have Week 24 viral load date (cut-off 2):
  - cut-off date = the earliest of (Day of Study Discontinuation from DS, date of Withdrawal Visit from SV, Study day of permanent treatment discontinuation from EX (for subjects randomized to DTG/3TC) or CM (for patients randomized to CAR), study treatment start date + 210\* -1).

\*upper bound of week 24 window

Additional Statistical Programming Checks to identify 'Subjects with study withdrawal due to a reason of "Protocol Deviation" (as recorded in the eCRF) at or prior Week 24' will be performed.

- Consider subjects that have discontinued from the study prior or at Week 24 with 'Protocol deviation' as a reason in DS (study discontinuation).
- Cut-off date (cut-off 3):
- For subjects who have Week 24 viral load date -> cut-off = Week 24 viral load date (used for snapshot algorithm) from LB (laboratory) dataset.
- For subjects who withdrawn before Week 24 Snapshot HIVRNA sample taken or if missing data during week 24 window but on study-> cut-off = IP start date + 210\* - 1
- Compare the PD occurrence date (Day of Study Discontinuation from DS) to cut-off date (see paragraph above, please note: cut-off rules 1 and 2 defined above do not apply here)
- If cut-off date ≥ PD occurrence date, then deviations will result in exclusion from the per protocol set.

Similar rules will be followed for Week 48 and subsequent time points and will be detailed in a separate Protocol Deviation specification document. Please refer to latest version of the Protocol Deviation specification document prior to the analysis for full details of protocol deviation identification.

<sup>\*</sup>upper bound of week 24 window

## 15.6.8. eCRF Baseline Third Agent Class Determination

Baseline third agent will be determined as the third agent ingredient:

- still being taken at randomization for CAR patients
- discontinued immediately prior to randomization for DTG/3TC patients.

## 15.7. Appendix 7: Reporting Standards for Missing Data

## 15.7.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | Subject study completion (i.e. as specified in the protocol) was defined as: Randomly assigned to either treatment group, completed the Randomized Phase including the Week 52 visit, and did not enter the Continuation Phase; |
| | <ul> <li>Subjects randomized to DTG/3TC treatment group, completed the Randomized Phase including the Week 52 visit, entered and completed the Continuation Phase, defined as remaining on study until: <ul> <li>DTG and 3TC FDC tablet is locally approved for use as a 2-drug regimen, and available through public health services or through the subject's usual health insurance payer, or</li> <li>the actual FDC tablet, if required by local regulations, is available, or</li> <li>the subject no longer derives clinical benefit, or</li> <li>the subject meets a protocol-defined reason for discontinuation, or</li> <li>development of the DTG/3TC dual regimen is terminated.</li> </ul> </li> <li>Withdrawn subjects will not be replaced in the study.</li> <li>All available data from subjects who were withdrawn from the study will be listed.</li> </ul> |

## 15.7.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Missing data occurs when any requested data are not provided, leading to blank fields on the collection instrument:</li> <li>These data will be indicated by the use of a "blank" in subject listing displays. Unless all data for a specific visit are missing in which case the data are excluded from the table.</li> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be missing data and should not be displayed as such.</li> </ul> |
| Snapshot | <ul> <li>In the Snapshot dataset, subjects without HIV-1 RNA data in the assessment<br/>window for the visit of interest (due to missing data or discontinuation of IP prior<br/>to the visit window) are classified as either 'HIV-1 RNA ≥50 c/mL') or 'No<br/>Virologic Data'. For full details of the Snapshot algorithm see Appendix 11</li> </ul> |
| Observed<br>Case (OC) | This dataset uses only the data that is available at a particular timepoint, with no imputation for missing values. |

## 15.7.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Partial dates will be displayed as captured in subject listing displays.</li> <li>Where necessary, display macros may impute dates as temporary variables for sorting data in listings only. In addition, partial dates may be imputed for 'slotting' data to study phases or for specific analysis purposes as outlined below.</li> </ul> |
| Exposure | <ul> <li>If study treatment stop date is missing, then for the purposes of calculating exposure, it will be imputed using the date of last visit or the recorded date of withdrawal/completion whichever is earlier.</li> <li>Partially Missing Stop Day: Last day of the month or last month of the year will be used, unless this is after the stop date of study treatment or withdrawal date; in this case the earliest of the two dates will be used. Note Study Treatment DTG/3TC is recorded on the Study Treatment eCRFs and CAR treatment is recorded on the CONART eCRFs.</li> </ul> |
| Adverse<br>Events and<br>Clinical<br>Events | <ul> <li>The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE and Clinical Event start and end dates; that is, the day of the month may be missing: <ul> <li>If the full date cannot be ascertained, the following conventions will be applied for calculating the time to onset and the duration of the event:</li></ul></li></ul> |

| Element | Reporting Detail |
|---|---|
| | case the study treatment start date will be used and hence the event is considered On-treatment as per Appendix 4: Treatment States and Phases O Partially Missing Stop Day: Last day of the month or last month of the year will be used, unless this is after the stop date of study treatment or withdrawal date; in this case the earliest of the two dates will be used. Otherwise, if patient hasn't withdrawn, last visit date will be used. The recorded partial date will be displayed in listings. |
| Concomitan<br>t<br>Medications | <ul> <li>Partial dates for any concomitant medications recorded in the eCRF will be imputed using the following convention: <ul> <li>If the partial date is a start date, the first day of the month will be used for the day and 'Jan' will be used for the month</li> <li>If the partial date is a stop date, last day of the month will be used for the day and 'Dec' will be used for the month.</li> <li>For medications recorded in the eCRF as prior ART, the earlier of this imputed date or the day before IP start will be used.</li> </ul> </li> </ul> |
| | The recorded partial date will be displayed in listings. |

# 15.8. Appendix 8: Values of Potential Clinical Importance

| Element | Reporting Detail |
|---|---|
| Laboratory<br>Values | The DAIDS grading for severity of laboratory toxicities and clinical adverse events is included in the protocol. |
| (Chemistry<br>(Including<br>Lipids), | The central laboratory will flag laboratory parameter toxicities directly in the provided datasets for subjects with any value outside normal range. |
| Hematology<br>and<br>Urinalysis) | <ul> <li>Abnormalities for potential clinical concern/importance will be defined as<br/>any Grade1-5 toxicity.</li> </ul> |

# **15.9. Appendix 9: Population Pharmacokinetic (PopPK) Analyses** There is no population pharmacokinetic analysis planned in this study.

## 15.10. Appendix 10: Time to Event Details

#### 15.10.1. TRDF Detailed Steps

#### **TRDF** Detailed steps

The steps below are for the derivation of TRDF at specific timepoints when the upper bound of the analysis window is used as a cut-off i.e. for the table only.

Randomized Period denotes period where subjects are still on their randomized treatment, prior to entering Continuation Phase for DTG/3TC subjects. This is also irrespective of blinding.

Final step of the derivation is made in following order:

- [1] When one EVENT (1.2, 2.2, 3.2, 4.2) criterion is satisfied, select. In situations where more than one EVENT criteria satisfied, select the earliest event. If the earliest event date satisfies more than one criteria (e.g. subject had CVW and discontinuation), select CVW.
- [2] When one CENSOR (1.1, 2.1, 3.1, 4.1, 5.x) criterion is satisfied, select. Else in situations where more than one CENSOR criteria satisfied, select the latest censor day. If the latest event date satisfies more than one criteria, apply the ordering below.

| Condition | Censor<br>Status | Event Description/AVAL |
|---|---|---|
| <ol> <li>Subjects met CVW event criteria during the randomized period.</li> <li>(Based on derived CVW confirmed prior to cutoff used for the analysis)</li> </ol> | | |
| Then set <b>tempAVAL</b> = Study Day of SVW immediately preceding CVW | | |
| 1.1 Initial elevation/SVW immediately preceding CVW event date is after the upper bound of the analysis visit window i.e tempAVAL > upper bound of the analysis visit window for Week X | CNSR=1 | EVNTDESC=Censored due to data cutoff. AVAL=Upper bound of analysis visit window. |

| TRDF Detailed steps | | |
|---|---|---|
| $1.2\ \text{Initial elevation/SVW immediately} \\ \text{preceding CVW event date is on or before the} \\ \text{upper bound of the analysis visit window} \\ \text{i.e tempAVAL} \leq \text{upper bound of the analysis} \\ \text{visit window for Week X} \\$ | CNSR=0 | EVNTDESC=CVW. AVAL= tempAVAL. |
| 2. Subjects with study withdrawal due to treatment related adverse events during the randomized period (defined as subjects that have reason for withdrawal =AE on disposition page and that the subject has at least one AE considered both: i) drug related (AEREL=Y) and ii) result in withdrawal from study (AEWD=Y)) Then set tempAVAL= Earliest of (Day of Study Discontinuation [from Disposition page]), date of Withdrawal Visit [from Study Visit domain], Study day of permanent treatment discontinuation [from Exposure and Concomitant ART domains]). Assumption: Study day of permanent treatment discontinuation is included in the definition to account for cases where discontinuation information is recorded later. This is a conservative approach consistent with treatment discontinuation preceding withdrawal. | | |
| 2.1 Study withdrawal is after the upper bound of the analysis visit window | CNSR=1 | EVNTDESC=Censored due to data cutoff. |
| i.e tempAVAL $>$ upper bound of the analysis visit window | | AVAL=Upper bound of analysis visit window. |
| 2.2 Study withdrawal is on or before the upper bound of the analysis visit window | CNSR=0 | EVNTDESC=Study Withdrawal Due to Treatment Related AE. |
| i.e tempAVAL $\leq$ upper bound of the analysis visit window | | AVAL= tempAVAL |

| TRDF Detailed steps | | |
|---|---|---|
| 3: Subjects met protocol defined stopping criteria during the randomized period., (Based on disposition page) | | |
| Then set <b>tempAVAL</b> =Earliest of (Day of Study Discontinuation [from Disposition page]), date of Withdrawal Visit [from Study Visit domain], Study day of permanent treatment discontinuation [from Study Treatment or CONART eCRF pages]). | | |
| 3.1 Protocol defined stopping criteria were met after the upper bound of the analysis visit window $ \label{eq:control_eq} \text{i.e tempAVAL} > \text{upper bound of the analysis } \\ \text{visit window} $ | CNSR=1 | EVNTDESC=Censored due to data cutoff. AVAL=Upper bound of analysis visit window. |
| 3.2 Protocol defined stopping criteria were met on or before the upper bound of the analysis visit window $ \text{i.e tempAVAL} \leq \text{upper bound of the analysis } \\ \text{visit window} $ | CNSR=0 | EVNTDESC=Study Withdrawal Due to Protocol Defined Criteria. AVAL=tempAVAL |
| 4: Subjects with study withdrawal due to lack of efficacy during the randomized period. (Based on disposition page) | | |
| Then set <b>tempAVAL</b> = Earliest of (Day of Study Discontinuation [from Disposition page]), date of Withdrawal Visit [from Study | | |

| TRDF Detailed steps | | |
|---|---|---|
| Visit domain], Study day of permanent treatment discontinuation [from Study Treatment or CONART eCRF pages]) | | |
| 4.1 Study withdrawal is after the upper bound of the analysis visit window | CNSR=1 | EVNTDESC=Censored due to data cutoff. |
| i.e tempAVAL $>$ upper bound of the analysis visit window | | AVAL=Upper bound of analysis visit window. |
| $\label{eq:continuous} 4.2 \text{ Study withdrawal is on or before the upper bound of the analysis visit window}$ $\text{i.e tempAVAL} \leq \text{upper bound of the analysis visit window}$ | CNSR=0 | EVNTDESC=Study Withdrawal Due to Lack of Efficacy AVAL= tempAVAL |
| If none of the above conditions met 5: Subjects with study withdrawal for other reasons during the randomized period. (Based on disposition page) | | |
| Then set <b>tempAVAL</b> = Earliest of (Day of Study Discontinuation [from Disposition page]), date of Withdrawal Visit [from Study Visit domain], Study day of permanent treatment discontinuation [from Study Treatment or CONART eCRF pages]) | | |
| 5.1 Study withdrawal is after the upper bound of the analysis visit window i.e tempAVAL > upper bound of the analysis visit window | CNSR=1 | EVNTDESC=Censored due to data cutoff. AVAL=Upper bound of analysis visit window. |
| 5.2 Study withdrawal is on or before the upper bound of the analysis visit window | CNSR=1 | EVNTDESC=Censored due to Study Discontinuation for Other Reasons. |

| TRDF Detailed steps | | |
|---|---|---|
| i.e $tempAVAL \! \leq \! upper$ bound of the analysis visit window | | AVAL=tempAVAL |
| 6: Subject completed the randomized period of the study. (Based on disposition page) | CNSR=1 | EVNTDESC= Censored as completed the Randomized Period. AVAL= Date of end of Treatment Phase |
| 7: Subject is ongoing in the study during the randomized period and have not yet completed the randomized period Assumption: this will only be in cases where the reporting effort/analysis is performed midway through the randomized period | CNSR=1 | EVNTDESC= Censored due to data cutoff. AVAL=Upper bound of analysis visit window. |

#### 15.10.2. TRDF Detailed Steps for the Kaplan-Meier plot

#### **TRDF Detailed steps**

The steps below are for the derivation of TRDF overall i.e. for the Kaplan-Meier plot only.

Final step of the derivation is made in following order:

- [1] When one EVENT (conditions 1-4) criterion is satisfied, select. In situations where more than one EVENT criteria satisfied, select the earliest event. If the earliest event date satisfies more than one criteria (e.g. subject had CVW and discontinuation), select CVW.
- [2] When one CENSOR (conditions 5.x) criterion is satisfied, select. Else in situations where more than one CENSOR criteria satisfied, select the latest censor day. If the latest event date satisfies more than one criteria, apply the ordering below.

| Condition | Censor<br>Status | Event Description/AVAL |
|---|---|---|
| Subjects met CVW event criteria during the randomized period. (Based on derived CVW confirmed prior to cut-off used for the analysis) | CNSR=0 | EVNTDESC=CVW. AVAL=Study Day of SVW immediately preceding CVW. |
| 2. Subjects with study withdrawal due to treatment related adverse events during the randomized period (defined as subjects that have reason for withdrawal =AE on disposition page and that the subject has at least one AE considered both: i) drug related (AEREL=Y) and ii) result in withdrawal from study (AEWD=Y)) | CNSR=0 | EVNTDESC=Study Withdrawal Due to Treatment Related AE. AVAL=Earliest of (Day of Study Discontinuation [from Disposition page]), date of Withdrawal Visit [from Study Visit domain], Study day of permanent treatment discontinuation [from Study Treatment or CONART eCRF pages]). |
| 3: Subjects met protocol defined stopping criteria during the randomized period., (Based on disposition page) | CNSR=0 | EVNTDESC=Study Withdrawal Due to Protocol Defined Criteria. AVAL=Earliest of (Day of Study Discontinuation [from Disposition page]), date of Withdrawal Visit [from Study |

| | | Visit domain], Study day of permanent treatment discontinuation [from Study Treatment or CONART eCRF pages]). |
|---|---|---|
| 4: Subjects with study withdrawal due to lack of efficacy during the randomized period. (Based on disposition page) | CNSR=0 | EVNTDESC=Study Withdrawal Due to Lack of Efficacy AVAL= Earliest of (Day of Study Discontinuation [from Disposition page]), date of Withdrawal Visit [from Study Visit domain], Study day of permanent treatment discontinuation [from Study Treatment or CONART eCRF pages]) |
| If none of the above conditions met | | |
| 5: Subjects with study withdrawal for other reasons on or before the end of randomized period. (Based on disposition page) | CNSR=1 | EVNTDESC=Censored due to Study Discontinuation for Other Reasons. AVAL=Earliest of (Day of Study Discontinuation [from Disposition page]), date of Withdrawal Visit [from Study Visit domain], Study day of permanent treatment discontinuation [from Study Treatment or CONART eCRF pages]) |
| 6: Subject completed the randomized period of the study. (Based on disposition page) | CNSR=1 | EVNTDESC= Censored as completed the Randomized Period. AVAL= Date of completion of randomized study period |
| 7: Subject is ongoing in the study during the randomized period and have not yet completed the randomized period | CNSR=1 | EVNTDESC= Ongoing in the Study. AVAL=Last visit date |

Notes:

#### CONFIDENTIAL

208090

- 1. Randomized Period = Randomized Phase
- 2. Efficacy visit windows should be used throughout for the upper bound of the analysis visit window
- 3. Subjects are considered to have completed the randomized period if they completed the Randomized Phase.
- 4. By definition, a subject must be on-treatment for a CVW to be recorded therefore inclusion of study date of treatment discontinuation in the derivation is not required
- 5. EVNTDESC, AVAL & CNSR variables created for the following timepoints:
  6. Week 24 or 48 for the table analysis
- 7. Overall for the Kaplan-Meier plot
#### 15.10.3. ERDF Detailed Steps

Similar algorithm will be applied for ERDF analyses and Kaplan-Meier figure, where condition 2 and 3 in Section 15.10.1 and Section 15.10.2 will not be considered.

#### 15.11. Appendix 11: Snapshot Algorithm Details

- Consider an analysis visit window, Week X (e.g. Week 24, Week 48). The Window for Week 24/48 visit is defined in Appendix 3. e.g. Week 48 (+/- 6 Week: 295 ≤ Study Day ≤ 378)
- Consider an HIV1-RNA threshold (e.g. 40, 50, 200 copies/mL ...) in analysis,
- The analysis window 'Week 48' and HIV1-RNA threshold of '50 c/mL' are used for the purpose of illustration. A subject's Snapshot response and reason at Week 48 are categorized as below.
  - o HIV1-RNA < **50** copies/mL
  - o HIV1-RNA ≥ 50 copies/mL

Data in window not below 50 Discontinued for lack of efficacy Discontinued for other reason while not below 50 Change in background therapy\*

No Virologic Data at Week 48 Window
 Discontinued study due to AE or death
 Discontinued study for other reasons
 On study but missing data in window

\* Note: since changes in ART or dose modification are not permitted in this protocol, all such subjects who change ART during Randomized Phase will be considered 'HIV1-RNA ≥ 50 c/mL'. if the change in ART is made prior to an analysis timepoint. For subjects on CAR, a switch from a PI boosted with ritonavir to the same PI boosted with cobicistat (and vice versa) is permitted per protocol and a switch from lamivudine to emtricitabine and vice versa will not be considered 'HIV1-RNA ≥ 50 copies/mL' due to 'change in ART'.

The steps in determining response and reasons are indicated in Table below, in the order stated.

#### **Detailed steps**

- Please note that the following scenarios will NOT be penalized Per Snapshot algorithm (i.e. please excluding these scenarios from **Condition** 1-4).
- Dose reduction, dropping a component, or change in formulation (e.g. 'Tivicay + Kivexa' to 'Triumeq' with the identical ingredients)
- Permitted Change (if a decision date is not collected in eCRF) / decision to permitted change is made prior to/on the first on-treatment viral load result
- Permitted change is made after the first on-treatment viral load result AND last ontreatment viral load prior to/on the date of change is <50 c/mL</li>

| Cond | | Response | Reasons |
|---|---|---|---|
| _ \ | k 48' indicates Week 48 window) | | |
| to | non-permitted change in background therapy prior Week 48 | HIV1-RNA ≥<br>50 | Change in background therapy |
| ۱<br>t | <b>permitted</b> change in background therapy <b>prior to</b> Neek 48 AND the latest on-treatment VL prior to/on he date of change is ≥ 50 c/m [a] | HIV1-RNA ≥ 50 | Change in background therapy |
| | <i>non-permitted</i> change in background therapy<br><i>uring</i> Week 48 | | |
| • | 3.1 Last on-treatment VL during Week 48 prior to/on the date of change ≥ 50 c/mL | HIV1-RNA ≥<br>50 | Data in window<br>not below 50 |
| • | 3.2 Last on-treatment VL during Week 48 prior to/on the date of change <50 c/mL | HIV1-RNA < 50 | |
| • | 3.3 No VL during Week 48 prior to/on the date of change | HIV1-RNA ≥ 50 | Change in background therapy |
| W | <b>permitted</b> change in background therapy <b>during</b> leek 48 AND the last on-treatment VL prior to/on the late of change is $\geq$ 50 c/mL [a] | | |
| 4. | 1 this last on-treatment VL occurs prior to Week 48 | HIV1-RNA ≥ 50 | Change in background therapy |
| | 2 this last on-treatment VL occurs during Week 48 but prior to/on the date of change | HIV1-RNA ≥<br>50 | Data in window<br>not below 50 |
| 5. If r | one of the above conditions met | | |
| 5. | 1 VL available during Week 48 | | |
| 5. | 1.1 Last on-treatment VL during Week 48 ≥ 50 c/mL | HIV1-RNA ≥ 50 | Data in window not below 50 |
| 5. | 1.2 Last on-treatment VL during Week 48 <50 c/mL | HIV1-RNA < 50 | |
| 5.2 | No VL during Week 48 | | |
| 5.2 | 2.1 If subjects still on study (i.e. The on-treatment period has not been ended up to the upper bound of Week 48 window. For example, for oral treatment, the on-treatment period ends at permanently IP stop date+1) | No virologic<br>data at Week<br>48 Window | On study but missing data in window |
| 5.2 | 2.2 If subjects withdraw before/during Week 48 due to :- | | |
| 5.2 | 2.2.1 Safety reasons (e.g. AE/death, liver chemistry stopping criteria, renal toxicity withdrawal criteria, QTc withdrawal criteria et al, as recorded in eCRF Study Conclusion form) | No virologic<br>data at Week<br>48 Window | Disc. due to<br>AE/death |
| 5.2 | 2.2.2 Non-safety related reasons (e.g. Lack of efficacy, protocol deviation, withdrew consent, | | |

| loss to follow-up, study closed/terminated, investigator discretion et al, as recorded in eCRF Study Conclusion Form) | | |
|---|---|---|
| 5.2.2.2.1 Last on-treatment VL <50 c/mL OR no on-treatment VL available during study | No virologic<br>Data at Week<br>48 Window | Disc. for other reasons |
| 5.2.2.2.2 Last on-treatment VL ≥ 50 c/mL AND withdrawal due to Lack of efficacy | HIV1-RNA ≥ 50 | Disc. for lack of efficacy |
| 5.2.2.2.3 Last on-treatment VL ≥ 50 c/mL AND withdrawal due to all other non-safety related reasons | HIV1-RNA ≥ 50 | Disc. for other reason while not below 50 |

<sup>1. [</sup>a]: Excluding permitted change in background therapy where change or decision to change is made prior to/on the first on-treatment viral result

Snapshot outcomes are shown below and are to be used in conjunction with the steps in the Snapshot algorithm

Figure 1 Flowchart of Snapshot Outcome



1: Last on-treatment VL in Week 48 window 2: Last on-treatment VL prior to Week 48 Reasons for HIV-1 RNA≥ 50 c/mL 3: Change in background therapy 7: Discontinued for lack of efficacy 8: Discontinued for other reason while not below 50 9: Data in window not below 50 Reasons for 'No Virologic data at Week 48' 4: Discontinued due to AE/death 5: Discontinued for other reasons 6: On study but missing data in window

A dataset will be created based on the Snapshot algorithm, where the dataset contains the following information, as a minimum:

Study identification

Subject identification

Study day and date of last blinded treatment

Virologic outcome based on the snapshot approach (i.e., HIV-1 RNA  $\leq$  50 c/mL, HIV-1 RNA  $\geq$  50 c/mL, discontinued due to AE or death, discontinued for other reasons, on study but missing data during window)

The HIV-1 RNA measurement and the corresponding study day and date used to determine the above virologic outcome if the measurement was not missing

Study day and date when the subject switched to open-label treatment due to lack or loss of virologic suppression, if applicable

Discontinuation study day and date, reason for discontinuation, and last blinded treatment measurement before discontinuation for subjects who discontinued study drug

#### 15.12. Appendix 12: Modified Snapshot Algorithm Details

The below Modified Snapshot Algorithm will be used to determine Snapshot outcomes taking into account COVID-19 related events. The Modified Snapshot Estimand still reports high-level categories (>=50 c/mL, <50 c/mL and No Virologic Data) in exactly the same way as the standard FDA Snapshot Algorithm in Section 15.11, however it reports additional subcategories to account for outcomes related to COVID-19.

- Consider an analysis visit window, Week X (e.g. Week 24, Week 48). The Window for Week 24/48 visit is defined in Appendix 3. e.g. Week 48 (+/- 6 Week: 295 ≤ Study Day ≤ 378)
- Consider an HIV1-RNA threshold (e.g. 40, 50, 200 copies/mL ...) in analysis,
- The analysis window 'Week 48' and HIV1-RNA threshold of '50 c/mL' are used for the purpose of illustration. A subject's Modified Snapshot response and reason at Week 48 are categorized as below.
  - o HIV1-RNA < 50 copies/mL
  - HIV1-RNA  $\geq$  **50** copies/mL

Data in window not below 50

Non-COVID-19 related

Discontinued for lack of efficacy

Discontinued for other reason and HIV-1 RNA >= 50 copies/mL

Change in ART\*

COVID-19 related

Discontinued for lack of efficacy

Discontinued for other and HIV-1 RNA >= 50 copies/mL

Change in background therapy\*

No Virologic Data at Week 48 Window

Non COVID-19 related

Discontinued study due to AE or death

Discontinued study for other reasons

On study but missing data in window

COVID-19 related

Discontinued study due to AE or death

Discontinued study for other reasons

On study but missing data in window

<sup>\*</sup> Note: since changes in ART or dose modification are not permitted in this protocol, all such subjects who change ART during Randomized Phase will be considered 'HIV1-RNA ≥ 50 c/mL' if the change in ART is made prior to an analysis timepoint. For subjects on CAR, a switch from a PI boosted with ritonavir to the same PI boosted with cobicistat (and vice versa) is permitted per protocol and a switch from lamivudine to emtricitabine and vice versa will not be considered 'HIV1-RNA ≥ 50 copies/mL' due to 'change in ART'.

The steps in determining response and reasons are indicated in Table below, in the order stated.

#### **Detailed steps**

- Please note that the following scenarios will NOT be penalized Per Modified Snapshot algorithm (i.e. please excluding these scenarios from Condition 1-4).
- Dose reduction, dropping a component, or change in formulation (e.g. 'Tivicay + Kivexa' to 'Triumeq' with the identical ingredients)
- Permitted Change (if a decision date is not collected in eCRF) / decision to permitted change is made prior to/on the first on-treatment viral load result
- Permitted change is made after the first on-treatment viral load result AND last ontreatment viral load prior to/on the date of change is <50 c/mL</li>

| Condition | Response | Reasons |
|---|---|---|
| ( 'Week 48' indicates Week 48 window) | 110/4 5514 | |
| 1.1 If <i>non-permitted</i> change in background therapy <i>prior</i> to Week XX (Non-COVID-19 switch) | HIV1-RNA ≥ 50 | Change in background therapy (Non-COVID-19 related) |
| 1.2 If <i>non-permitted</i> change in background therapy <i>prior</i> to Week XX (COVID-19 switch) | HIV1-RNA ≥<br>50 | Change in background therapy (COVID-19 related) |
| 2. 1 If <b>permitted</b> change in background therapy <b>prior to</b> Week 48 AND the latest on-treatment VL prior to/on the date of change is ≥ 50 c/mL (not related to COVID-19) [a] | HIV1-RNA ≥ 50 | Change in background therapy(Non-COVID-19 related) |
| 2. 2 If <b>permitted</b> change in background therapy <b>prior to</b> Week 48 AND the latest on-treatment VL prior to/on the date of change is ≥ 50 c/mL(related to COVID-19) [a] | HIV1-RNA ≥ 50 | Change in background therapy(COVID-19 related) |
| 4. If <i>non-permitted</i> change in background therapy | | |
| during Week 48 | | |
| 3.1 Last on-treatment VL during Week 48 prior to/on the date of change ≥ 50 c/mL | HIV1-RNA ≥<br>50 | Data in window not below 50 |
| 3.2 Last on-treatment VL during Week 48 prior to/on the date of change <50 c/mL | HIV1-RNA < 50 | |
| 3.3.1 No VL during Week 48 prior to/on the date of change (non-related to COVID-19) | HIV1-RNA ≥<br>50 | Change in background therapy(Non-COVID-19 related) |

| • | 3.3.2 No VL during Week 48 prior to/on the date of change (related to COVID-19) | HIV1-RNA ≥ 50 | Change in background therapy( COVID-19 related) |
|---|---|---|---|
| V | <b>permitted</b> change in background therapy <b>during</b> /eek 48 AND the last on-treatment VL prior to/on the ate of change is $\geq$ 50 c/mL [a] | | |
| 4. | <ul><li>1.1 this last on-treatment VL occurs prior to Week</li><li>48 (non- COVID-19 related switch)</li></ul> | HIV1-RNA ≥<br>50 | Change in background therapy (Non-COVID-19 related) |
| 4. | <ul><li>1.2 this last on-treatment VL occurs prior to Week</li><li>48 (COVID-19 related switch)</li></ul> | HIV1-RNA ≥<br>50 | Change in background therapy (COVID-19 related) |
| | 2 this last on-treatment VL occurs during Week 48 but prior to/on the date of change | HIV1-RNA ≥<br>50 | Data in window not below 50 |
| | none of the above conditions met | | |
| | 1 VL available during Week 48 | | |
| | 1.1 Last on-treatment VL during Week 48 ≥ 50 c/mL | HIV1-RNA ≥ 50 | Data in window not below 50 |
| 5. | 1.2 Last on-treatment VL during Week 48 <50 c/mL | HIV1-RNA < 50 | |
| 5. | 2 No VL during Week 48 | | |
| 5.: | 2.1 Participants unable to attend Week 48 visit due to COVID-19, but otherwise considered still onstudy (i.e. The on-treatment period continues beyond the upper bound of Week 48 window. For example, for oral treatment, a participant with IP stop date+1> Day 378 of the upper bound of Week 48 window, would be considered 'on study' for Week 48 snapshot assessment) | No virologic<br>data at Week<br>48 Window | On study but<br>missing data in<br>window(COVID-<br>19 related) |
| 5.: | 2.2 If participants still on study but participant has not missed visit due to COVID-19 (i.e. The ontreatment period continues beyond the upper bound of Week 48 window. For example, for oral treatment, a participant with IP stop date+1> Day 378 of the upper bound of Week 48 window, would be considered 'on study' for Week 48 snapshot assessment) | No virologic<br>data at Week<br>48 Window | On study but<br>missing data in<br>window(Non-<br>COVID-19<br>related) |
| 5. | 3.2 If participants withdraw before/during Week 48 due to: | | |

| 5.3.2.1 Non-COVID-19 Safety reasons (e.g. non-COVID-19 AE/death, liver chemistry stopping criteria, renal toxicity withdrawal criteria, QTc withdrawal criteria, as recorded in eCRF Conclusion form) | No virologic<br>data at Week<br>48 Window | Disc. due to<br>AE/death(Non-<br>COVID-19<br>related) |
|---|---|---|
| 5.3.2.2 COVID-19 safety reasons eCRF (e.g. AE/death resulting from COVID-19 as recorded in the eCRF Conclusion form). If subject has AE or death recorded as primary reason for discontinuing (not captured as COVID-19 related), but subject has at least one COVID-19 related AE/death leading to withdrawal per AE eCRF page, the subject will assumed to have discontinued as a result of COVID-19 AE/death and hence will be captured in this Snapshot category. | No virologic<br>data at Week<br>48 Window | Disc. due to<br>AE/death(COVID-<br>19 related) |
| 5.3.2.3 Non-safety and non-COVID-19 related reasons (e.g. Lack of efficacy, protocol deviation, withdrew consent, loss to follow-up, study closed/terminated, investigator discretion et al, as recorded in eCRF Study Conclusion Form) | | |
| 5.3.2.3.1 Last on-treatment VL <50 c/mL OR no on-treatment VL available during study | No virologic<br>Data at Week<br>48 Window | Disc. for other<br>reasons(Non-<br>COVID-19<br>related) |
| 5.3.2.3.2 Last on-treatment VL ≥ 50 c/mL AND withdrawal due to Lack of efficacy | HIV1-RNA ≥<br>50 | Disc. for lack of<br>efficacy(Non-<br>COVID-19<br>related) |
| 5.3.2.3.3 Last on-treatment VL ≥ 50 c/mL AND withdrawal due to all other non-safety related reasons | HIV1-RNA ≥<br>50 | Disc. for other<br>reason while not<br>below 50(Non-<br>COVID-19<br>related) |
| 5.3.2.4 Non-safety and COVID-19 related reasons (e.g. Withdrawal of consent, protocol deviation (where subreason is COVID-19), investigator discretion (where Other text is recorded as 'COVID-19'), as recorded in eCRF Conclusion Form) | | |
| 5.3.2.4.1 Last on-treatment VL <50 c/mL OR no on-treatment VL available during study | No virologic<br>Data at Week<br>48 Window | Disc. for other reasons(COVID-19 related) |
| 5.3.2.4.2 Last on-treatment VL ≥ 50 c/mL AND withdrawal due to all other non-safety related reasons | HIV1-RNA ≥<br>50 | Disc. for other reason while not below 50(COVID-19 related) |

## 15.13. Appendix 13: Abbreviations & Trade Marks

#### 15.13.1. Abbreviations

| Abbreviation | Description |
|---|---|
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| AIC | Akaike's Information Criteria |
| A&R | Analysis and Reporting |
| CAR | Current ART regimen |
| cART | Combination ART |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| CPMS | Clinical Pharmacology Modelling & Simulation |
| CS | Clinical Statistics |
| CSR | Clinical Study Report |
| CTR | Clinical Trial Register |
| CV <sub>b</sub> /CV <sub>w</sub> | Coefficient of Variation (Between) / Coefficient of Variation (Within) |
| DOB | Date of Birth |
| DP | Decimal Places |
| DOV | Date of Visit |
| eCRF | Electronic Case Record Form |
| ERDF | Efficacy Related Discontinuation Failure |
| IA | Interim Analysis |
| ICH | International Conference on Harmonisation |
| IDMC | Independent Data Monitoring Committee |
| IDSL | Integrated Data Standards Library |
| IMMS | International Modules Management System |
| IP | Investigational Product |
| ITT | Intent-To-Treat |
| GUI | Guidance |
| LOC | Last Observation Carries Forward |
| MMRM | Mixed Model Repeated Measures |
| PCI | Potential Clinical Importance |
| PD | Protocol Deviation |
| PDMP | Protocol Deviation Management Plan |
| PK | Pharmacokinetic |
| PP | Per Protocol |
| QC | Quality Control |
| QTcF | Frederica's QT Interval Corrected for Heart Rate |
| RAP | Reporting & Analysis Plan |
| RAMOS | Randomization & Medication Ordering System |
| SAC | Statistical Analysis Complete |
| SDTM | Study Data Tabulation Model |

| Abbreviation | Description |
|--------------|-------------------------------------------|
| SOP | Standard Operation Procedure |
| TA | Therapeutic Area |
| TAF | Tenofovir alafenamide fumarate |
| CAR | Current antiretroviral regimen |
| TFL | Tables, Figures & Listings |
| TRDF | Treatment Related Discontinuation Failure |
| GSK | GlaxoSmithKline |

#### 15.13.2. Trademarks

| Trademarks of the GlaxoSmithKline<br>Group of Companies |
|---------------------------------------------------------|
| Epivir |
| Tivicay |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| Monogram Inc |
| NONMEM |
| SAS |
| WinNonlin |

# 15.14. Appendix 14: Model Checking and Diagnostics for Statistical Analyses

#### 15.14.1. Statistical Analysis Assumptions

| Endpoint(s) | Change from Baseline in bone/renal/inflammatory biomarkers, weight, BMI, HOMA-IR, HbA1c, lipids and health outcomes |
|---|---|
| Analysis | MMRM/ANCOVA |

- Model assumptions will be applied, but appropriate adjustments maybe made based on the data.
- The Kenward and Roger method for approximating the denominator degrees of freedom and correcting for bias in the estimated variance-covariance of the fixed effects will be used for MMRM models.
- An unstructured covariance structure for the R matrix will be estimated by treatment group by specifying 'type=UN' and 'group=treat' on the REPEATED line for MMRM models.
  - o In the event that this model fails to converge, alternative correlation structures may be considered such as CSH or CS.
  - Akaike's Information Criteria (AIC) will be used to assist with the selection of covariance structure.
- Distributional assumptions underlying the model used for analysis will be examined by
  obtaining a normal probability plot of the residuals and a plot of the residuals versus the fitted
  values (i.e. checking the normality assumption and constant variance assumption of the model
  respectively) to gain confidence that the model assumptions are reasonable.
- If there are any departures from the distributional assumptions, alternative models will be explored using appropriate transformed data.

| Endpoint(s) | Change from Baseline in Lipids |
|-------------|--------------------------------|
| Analysis | Multiple Imputation |

- Model assumptions will be applied, but appropriate adjustments maybe made based on the data.
- Distributional assumptions underlying the model used for analysis will be examined by obtaining a normal probability plot of the residuals (i.e. checking the normality assumption) to gain confidence that the model assumptions are reasonable.
- If there are any departures from the distributional assumptions, alternative models will be explored using appropriate transformed data.
- Diagnostic plots (trace and autocorrelation plots) will be checked to verify that the number of burn-in iterations and MCMC steps between imputed datasets are sufficient. If the trace plots show apparent trend or the autocorrelation plots show significant positive or negative autocorrelation, number of iterations will be increased until the diagnostic plots are acceptable.

# 15.15. Appendix 15: Test of Homogeneity: Fleiss, Liu & Kelly Method

# 15.15.1. Statistical Analysis Method for Test of Homogeneity by Fleiss, Liu & Kelly

| Analysis | Test of Homo | Test of Homogeneity by Fleiss, Liu & Kelly | |
|---|---|---|---|
| Subgroup i (i= 1 to K categories) | | | |
| | , | Not | |
| | Outcome of | Outcome of | |
| Treatment <sub>i</sub> (j=1,2) | Interest | Interest | Total |
| • | f both $\widehat{\pi}_{i1}$ or $\widehat{\pi}_{i2}$ (proation is made to count | • | either treatment for level i) is |
| Trt <sub>i</sub> =Trt₁ | $x_{ij} = x_{11}$ | n <sub>ii</sub> - x <sub>ii</sub> | n <sub>ii</sub> = n <sub>11</sub> |
| 7 | | | '''J ''' |
| g -1 | | $= n_{11} - x_{11}$ | 1111 1111 |
| Trt <sub>j</sub> =Trt <sub>2</sub> | $\mathbf{x}_{ij} = \mathbf{x}_{12}$ | , , | n <sub>ij</sub> = n <sub>12</sub> |

#### Sparse cells:

If either  $\widehat{\pi}_{i1}$  or  $\widehat{\pi}_{i2}$  (proportion of outcome in either treatment for level i) is 0 or 1 add 0.5 to each cell in level i (for level i only)

| caon sen in level i (loi level i only) | | | |
|---|---|---|---|
| Trt <sub>j</sub> =Trt₁ | $x_{ij} = x_{11} + 0.5$ | $n_{11} - x_{11} + 0.5$ | n <sub>ij</sub> = n <sub>11</sub> + 1 |
| Trt <sub>i</sub> =Trt <sub>2</sub> | $x_{ij} = x_{12} + 0.5$ | $n_{12} - x_{12} + 0.5$ | n <sub>ii</sub> = n <sub>12</sub> + 1 |

$$\widehat{\pi}_{ij} = \frac{x_{ij}}{n_{ij}}$$

H0: Risk differences in each level are equal.

Test Statistic:  $Q_{\text{wls}} = \sum_{i=1}^K \frac{(Y_{i-\hat{\tau}})^2}{\widehat{w}_I} \sim \text{ChiSq}_{(\text{K-1})}$ 

$$Y_i = \, \widehat{\pi}_{i1} - \, \widehat{\pi}_{i2}$$

$$\widehat{\tau} = \frac{\sum_{i=1}^{K} \frac{Y_i}{\widehat{w}_i}}{\sum_{i=1}^{K} \frac{1}{\widehat{w}_i}}$$

$$w_i = \frac{\widehat{\pi}_{i1} (1 - \widehat{\pi}_{i1})}{n_{i1} - 1} + \frac{\widehat{\pi}_{i2} (1 - \widehat{\pi}_{i2})}{n_{i2} - 1}$$

#### 15.16. Appendix 16: Final (End of Study) Analysis

This appendix provides the details of the planned analyses and data displays for End of Study (EoS) reporting. These analyses may be included in regulatory submissions, study reports and publications

The primary analysis at Week 48 have been completed based on the original RAP. This present appendix is written to cover only analyses included in the final end of study reporting. All derivations described in the study analysis plan will be re-used for end of study reporting and only those definitions and derivations that have changed since the previous interim and primary analysis are described below. This additional appendix summarizes only the key endpoints of interest for the final analysis and explain any deviations from the primary analysis.

The details of the final EOS reporting and analysis plan are described below:

- 1. The analysis for which the data have not been changed since the last interim analysis (Week 48 analysis) will not be reported to avoid redundancy.
- 2. No subgroup analysis, hypotheses testing, or statistical analyses will be performed.
- 3. The Continuation Phase is not applicable for participants in Sweden and Denmark.
- 4. All required disclosure outputs following the FDAAA and EudraCT guidelines will be produced. These outputs will include data from both Randomized and Continuation phase.
- 5. For the purpose of creation of Mexico Final Safety Report and submission to Ministry of Health, some listings at Mexico sites will be reported separately. Such listings are identified in the Programming notes in Section 15.16.9. These listings will include data from both Randomized and Continuation Phase

#### 15.16.1. Study Phases

In the previous analysis (Week 48 analysis), data were summarized for the Randomized Phase of the study. However, when data from the Continuation Phase were available, Continuation Phase was also included. For the EOS reporting, data to be analysed/reported are from Continuation Phase unless specified otherwise, and this will be noted in the title of the output. Listings containing data from both the Randomized and Continuation Phases will have a column added to specify the phase of the study for each record. Continuation Phase is defined as below:

| Phase | Start | End |
|---|---|---|
| Continuation Phase | Date of exposure after Week 52 in the DTG/3TC arm. | Study completion/discontinuation date |

#### 1. Notes:

- A participant enters the Continuation Phase if they have at least one exposure to the Investigational Product after analysis visit Week 52.
- There will be no Continuation Phase in the CAR Treatment arm.

#### 15.16.2. Analysis Populations for the Continuation Phase

In addition to the populations defined in Section 4 of the RAP, the following populations were defined for the End of Study Analysis:

| Population | Definition/ Criteria. | Analysis Evaluated |
|---|---|---|
| Safety - Continuation Phase | Comprises all participants in<br>the Safety Population who<br>receive at least one dose of<br>Investigational Product after<br>entering the Continuation<br>Phase. | • Safety |
| Intent-to-Treat Exposed (ITT-E) - Continuation Phase | Comprises all participants in the ITT-E Population who enter the Continuation Phase. | <ul><li>Efficacy</li><li>Study Population</li><li>Virology</li></ul> |
| CVW- Continuation Phase | Comprises all subjects in the ITT-E- Continuation Phase population who have met the derived CVW criteria | Virology |

#### 15.16.3. Study Population

The study population summaries and data listings will be based on the All Subjects Screened or ITT-E- Continuation Phase population, unless otherwise specified. Demographic and baseline characteristics will be reported only for the subjects who entered the Continuation Phase. Overview of the key planned study population endpoints:

- Study Populations
- Summary of Number of Subjects Enrolled by Country and Site ID for the Continuation Population.
- Concomitant and Antiretroviral Medications
- Protocol deviations
- Full details of the data displays are given in Section 15.16.9

#### 15.16.4. Efficacy Analysis

The efficacy summaries and data listings will be based on the ITT-E-Continuation Phase Population. HIV-1 RNA viral load will be summarized using observed data (i.e., subjects with missing data at a time point are excluded). A figure will be reported to present Individual Plasma HIV-1 RNA and CD4+ Profiles by Visit for Subjects with at least One Confirmed Virologic Withdrawal Visit in the Continuation Phase

Overview of the key planned efficacy endpoints:

- Proportion of Participants with Plasma HIV-1 RNA < 50 c/ mL/ >= 50 c/mLobserved data
- Proportion of Participants with Confirmed Virologic Withdrawal observed data
- Incidence of disease progression and HIV-associated conditions
- Distribution of Quantitative Plasma HIV-1 RNA Results at Suspected and Confirmed Virologic Withdrawal
- Full details of the data displays are given in Section 15.16.9.

#### 15.16.5. Safety Analysis

All safety displays will be based on the Safety population or Safety- Continuation Phase Population. The core adverse event displays for the final report have been identified based on the IDSL library required tables. For AE data (including COVID-19), unless stated otherwise, the summaries and listings will include only those AEs that occurred during Continuation Phase.

Summaries of AE required for the FDAAA and EudraCT will be generated in this reporting effort. Such summaries are identified in the Programming notes. These summaries will include events from both Randomized and Continuation Phase. Common AEs are those with >=1% (without rounding) incidence for any treatment. For drug related grade 2-5 AEs, the common threshold is defined as 0.5%. Overview of the key planned safety endpoints:

- Extent of Exposure
- Adverse Events
- Absolute values and Change from Baseline in Weight and BMI for subjects entering the Continuation Phase.
- Patient profiles for subjects meeting Protocol defined liver stopping criteria in the Continuation Phase.
- Positive Suicidal indication Alerts based on eC-SSRS occurring in the Continuation Phase.
- For subjects at Mexico sites the following listings will be generated in this reporting effort. These listings will include data from both Randomized and Continuation Phase for both DTG/3TC and CAR arms.
  - Listing of Non-Serious AEs of Subjects at Mexico sites
  - Listing of SAEs of Subjects at Mexico sites
  - Full details of the data displays are given in Section 15.16.9.

#### 15.16.6. Virology Analysis

The Virology displays will be based on CVW- Continuation Phase Population and ITT- E Continuation Phase - population. All virology summaries and Listings will include subjects who met Confirmed Virologic Withdrawal criteria during the Continuation phase.

Overview of the key planned virology endpoints: Refer to the Section 9.2.1 of this document.

Full details of the data displays are given in Section 15.16.9.

#### 15.16.7. COVID - 19 analysis

This study was started in 2019 and continued during the COVID -19 pandemic. The information regarding the number of participants affected by COVID-19 and its symptoms will be reported according to GSK core standards. The visits impacted due to the pandemic outbreak will be reported. Protocol deviations or adverse events related to COVID-19 if any, will also be reported according to GSK core standards.

#### 15.16.8. Other Analyses (Health Outcomes)

Overview of the key planned analysis:

• Change from Baseline in SDM for subjects entering the Continuation Phase.

#### 15.16.9. List of Data Displays for End of Study (EOS) Final Report

Outputs that were not reported in previous reporting effort are identified in Programming Notes as 'New output'.

| Study Po | pulation | | | | |
|---|---|---|---|---|---|
| Туре | No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes |
| Table | 1.36 | ITT-E -<br>Continuation<br>Phase | Same shell as<br>week 48, table<br>1.3 | Summary of Number of Subjects<br>Enrolled by Country and Site ID | |
| Table | 1.37 | All Subjects<br>Screened | SA1 | Summary of Study Populations | CS CORE; |
| Table | 1.38 | ITT-E-<br>Continuation<br>Phase | DV1a | Summary of Important Protocol<br>Deviations by relationship to<br>COVID-19 Pandemic-<br>Continuation Phase | CS CORE |
| Table | 1.39 | ITT-E-<br>Continuation<br>Phase | ES1 | Summary of Subject Status and<br>Subject Disposition by relationship<br>to COVID-19 Pandemic-<br>Continuation Phase | FDAAA, EudraCT<br>Summarise by: i)<br>Overall ii) Related to<br>COVID-19, ii) Not<br>related to COVID-19 |
| Table | 1.401 | ITT-E-<br>Continuation<br>Phase | DM1 | Summary of Demographic<br>Characteristics - Continuation<br>Phase | |
| Table | 1.41 | ITT-E-<br>Continuation<br>Phase | CM1 | Summary of Concomitant Medication by ATC Level 1 and Ingredient – Continuation Phase | |

| Study Pop | oulation | | | | |
|---|---|---|---|---|---|
| Listing-<br>ICH | 87 | ITT-E-<br>Continuation<br>Phase | ES2 | Listing of Study Conclusions<br>Reasons for Study Withdrawal –<br>Continuation Phase | |
| Listing-<br>ICH | 88 | ITT-E-<br>Continuation<br>Phase | DV2 | Listing of Important Protocol<br>Deviations – Continuation Phase | |
| Listing-<br>Other | 89 | ITT–E-<br>Continuation<br>Phase | Same shell as<br>week 48,<br>Listing 28 | Listing of Visit Dates -<br>Continuation Phase | |
| Listing -<br>Other | 90 | All Subjects<br>Screened | Same shell as<br>week 48,<br>Listing 29 | Listing of Study Populations | |
| Listing -<br>Other | 91 | ITT-E-<br>Continuation<br>Phase | CM2 | Listing of Concomitant Medications – Continuation Phase | |
| Listing -<br>Other | 92 | ITT-E-<br>Continuation<br>Phase | Same shell as<br>week 48,<br>Listing 39 | Listing of on-treatment Concomitant ART Medications – Continuation phase | |
| Listing -<br>Other | 92.1 | ITT-E-<br>Continuation<br>Phase | Same shell as<br>week 48,<br>Listing 40 | Listing of Antiretroviral Therapy Starting after Treatment Discontinuation - Continuation phase | |
| Efficacy | | | | | |
| Туре | No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes |
| Table | 2.33 | ITT-E-<br>Continuation<br>Phase | gsk3515864/mi<br>d204861/<br>primary_05/Tab<br>le 2.15 | Proportion of Subjects with<br>Plasma HIV-1 RNA <50 c/mL by<br>Visit -Observed Data | |
| Table | 2.34 | ITT-E-<br>Continuation<br>Phase | Same as above | Proportion of Subjects with Plasma HIV-1 RNA >=50 c/mL by Visit -Observed Data | |
| Table | 2.35 | ITT-E<br>Continuation<br>Phase | Same shell as<br>week 48, Table<br>2.14 | Summary of Change from<br>Baseline in Plasma HIV-1 RNA<br>(log10 c/mL) by Visit | |
| Table | 2.36 | ITT-E<br>Continuation<br>Phase | Same shell as<br>week 48, Table<br>2.21 | Proportion of Subjects Meeting<br>Confirmed Virologic Withdrawal<br>Criteria by Visit by Type of Criteria | |
| Table | 2.37 | ITT-E-<br>Continuation<br>Phase | Same shell as<br>week 48, Table<br>2.22 | Distribution of Quantitative Plasma HIV-1 RNA Results at Suspected and Confirmed Virologic Withdrawal | |
| Table | 2.38 | ITT-E-<br>Continuation<br>Phase | Same shell as<br>week 48, Table<br>2.18 | Summary of Post-Baseline HIV-1 Associated Conditions Including Recurrences - Continuation Phase | |

| Study Pop | Study Population | | | | |
|---|---|---|---|---|---|
| Table | | ITT-E- | Same shell as | Summary of Post-Baseline HIV-1 | |
| | | Continuation | week 48, Table | Associated Conditions Excluding | |
| | | Phase | 2.19 | Recurrences – Continuation | |
| | 2.39 | | | Phase | |
| Table | | ITT-E- | Same shell as | Summary of Post-Baseline HIV-1 | |
| | | Continuation | week 48, Table | Disease Progressions - | |
| | 2.40 | Phase | 2.20 | Continuation Phase | |
| | | ITT-E- | Same shell as | Individual Plasma HIV-1 RNA and | |
| | | Continuation | week 48, | CD4+ Profiles by Visit for Subjects | Include all visits |
| | | Phase | Figure 2.2 | with at least One Suspected | IIICIUUE ali VISIIS |
| Figure | 2.5 | | | Virologic Withdrawal Visit | |
| | | ITT-E- | Same shell as | Listing of Quantitative and | |
| Listing - | | Continuation | Week 48, | Qualitative Plasma HIV-1 RNA | |
| ICH | 93 | Phase | Listing 10 | Data- Continuation Phase | |
| | | ITT-E- | Same shell as | Listing of Plasma HIV-1 RNA Data | |
| | | Continuation | week 48, | and CD4+ cell count data for | |
| Listing - | | Phase | Listing 43 | Subjects with Confirmed Virologic | |
| Other | 94 | | | Withdrawal- Continuation Phase | |

| Safety | | | | | |
|---|---|---|---|---|---|
| Туре | No. | Population | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming<br>Notes |
| Table | 3.67 | Safety | EX1 | Summary of Extent of Exposure to Investigational Product | Including all phases |
| | 3.69 | Safety-<br>Continuation<br>Phase | Same shell as<br>Week 48,<br>Table 3.2 | Summary of All Adverse Events by System Organ Class and Preferred Term – Continuation Phase | |
| Table | 3.70 | Safety-<br>Continuation<br>Phase | AE3 | Summary of Common (>=1%) Adverse Events by Preferred Term and Overall Frequency - Continuation Phase | |
| Table | 3.71 | Safety-<br>Continuation<br>Phase | AE3 | Summary of Common (>=1%) Grade 2-5 Adverse Events by Preferred Term and Overall Frequency - Continuation Phase | |
| Table | 3.72 | Safety-<br>Continuation<br>Phase | AE5A | Summary of All Drug-related Adverse Events by System Organ Class, Preferred Term and Maximum Toxicity - Continuation Phase | |
| Table | 3.73 | Safety-<br>Continuation<br>Phase | AE3 | Summary of Common (>=0.5%) Drug-<br>related Grade 2-5 Adverse Events by<br>Overall Frequency - Continuation Phase | |
| Table | 3.74 | Safety-<br>Continuation<br>Phase | AE3 | Summary of Serious Adverse Events by<br>System Organ Class and Preferred Term -<br>Continuation Phase | |
| Table | 3.75 | Safety-<br>Continuation<br>Phase | AE15 | Summary of Serious Adverse Events by<br>System Organ Class and Preferred Term<br>(Number of Subjects and Occurrences) | FDAAA, EudraCT,<br>Ct.gov |

| Safety | | | | | |
|---|---|---|---|---|---|
| <b>,</b> | | | | | |
| Table | | Safety- | | Summary of Non-serious Adverse Events | |
| | | Continuation | | by System Organ Class and Preferred Term | |
| | 3.76 | Phase | AE16 | (Number of Subjects and Occurrences) | FDAAA, EudraCT |
| Table | | Safety- | Same shell as | Number of Subjects with an Adverse Event | |
| | 0.77 | Continuation | week 48, Table | of Suspected, Probable, Confirmed for | |
| T 11 | 3.77 | Phase | 3.18 | COVID-19 Infection – Continuation Phase | |
| Table | | Safety- | Same shell as | | |
| | 3.82 | Continuation<br>Phase | week 48, Table<br>3.42 | Cummony of Woight (kg) by Vioit | |
| Table | 3.02 | | Same shell as | Summary of Weight (kg) by Visit | |
| rable | | Safety-<br>Continuation | week 48, Table | Summary of Change from Baseline in | |
| | 3.83 | Phase | 3.43 | Weight (kg) by Visit | |
| Table | 3.03 | Safety- | Same shell as | Weight (kg) by Visit | |
| Table | | Continuation | week 48, Table | | |
| | 3.84 | Phase | 3.46 | Summary of BMI (kg/m2) by Visit | |
| Table | 0.01 | Safety- | Same shell as | Cummary or Bivii (kg/m2) by visit | |
| Table | | Continuation | week 48, Table | Summary of Change from Baseline in | |
| | 3.85 | Phase | 3.47 | BMI (kg/m2) by Visit | |
| Table | 0.00 | Safety- | Same shell as | Summary of True Positive Suicidal | |
| 1 0010 | | Continuation | week 144, | Indication/ Behaviour Alerts based on | |
| | 3.87 | Phase | Table 3.58 | eCSSRS by Visit – Continuation Phase | |
| Table | | Safety- | Same shell as | Summary of Subjects with Post-Baseline C- | |
| | | Continuation | week 48, Table | SSRS Suicidal Ideation or Behaviour – | |
| | 3.88 | Phase | 3.59 | Continuation Phase | |
| | | Safety- | Same shell as | | |
| Listing - | | Continuation | week 48, | Listing of Investigational Product Exposure | |
| ICH | 95 | Phase | Listing 12 | Data – Continuation Phase | |
| | | Safety- | | | |
| Listing - | | Continuation | AE8 | Listing of All Adverse Events – Continuation | |
| ICH | 96 | Phase | | Phase | |
| | | Safety- | | Listing of Adverse Events Leading to | |
| | | Continuation | | Withdrawal/Permanent Discontinuation of | |
| Listing - | | Phase | | Investigational Product – Continuation | |
| ICH | 97 | | AE8 | Phase | |
| Listing- | | Safety- | | Listing of All Laboratory Data for Subjects | |
| ICH | | Continuation | Same shell as | with Any Value of Potential Clinical | |
| | 00 | Phase | Week 48, | Importance - Continuation Phase | |
| 1 (- 4 | 98 | 0-1-1 | Listing 20 | Lieting of Heineloois Data for O. 11. 4. 19 | |
| Listing- | | Safety- | Same shell as | Listing of Urinalysis Data for Subjects with | |
| ICH | 00.4 | Continuation | Week 48, | Any Value of Potential | |
| Lietine | 98.1 | Phase | Listing 21 | Clinical Importance - Continuation Phase | |
| Listing - | | Safety-<br>Continuation | | Patient Profiles for Subjects Meeting | |
| Other | | Phase | | Patient Profiles for Subjects Meeting Protocol Defined Liver Stopping Criteria – | |
| | 99 | FIIASE | LIVER5 | Continuation Phase | |
| Listing - | 99 | Safety- | Same shell as | Patient Profiles for Subjects Meeting | |
| Other | | Continuation | week 48, | Confirmed Virologic Withdrawal Criteria – | |
| Julion | 100 | Phase | Listing 58 | Continuation Phase | |
| Listing - | | Safety- | | | |
| g | 102 | | PREG1a | Listing of Subjects Who Became Pregnant | |

| Other | | Continuation<br>Phase | | During the Study – Continuation Phase | |
|---|---|---|---|---|---|
| Listing - | | Safety- | Same shell as | Listing of eC-SSRS Suicidal Ideation and | |
| Other | | Continuation | week 48, | Behaviour Positive Alerts (4-9) – | |
| | 103 | Phase | Listing 52 | Continuation Phase | |
| Listing - | | Safety- | Same shell as | | |
| Other | | Continuation | week 48, | Listing of eC-SSRS Suicidal Ideation and | |
| | 104 | Phase | Listing 53 | Behaviour Data Continuation Phase | |
| Listing - | | Safety- | Same shell as | Listing of eC-SSRS False Positive Alerts | |
| Other | | Continuation | week 48, | with Corresponding Reasons – Continuation | |
| | 105 | Phase | Listing 54 | Phase | |
| | | Safety- | Same shell as | | |
| Listing - | | Continuation | week 48, | Listing of all eC-SSRS True Positive Alerts | |
| Other | 106 | Phase | Listing 55 | with AE/SAE status – Continuation Phase | |
| | | Safety- | Same shell as | Listing of Subjects with an Adverse Event of | |
| Listing - | | Continuation | week 48, | Suspected, Probable, Confirmed for | |
| Other | 107 | Phase | Listing 64 | COVID-19 Infection – Continuation Phase | |
| Listing - | | Safety | AE8 | | New Output; |
| Other | | | | Listing of Non-Serious AEs of Subjects at | Mexican Safety |
| | | | | Mexico sites | Report |
| | 108 | | | | requirement |
| Listing - | | Safety | AE8 | | New Output; |
| Other | | , | | | Mexican Safety |
| | | | | Listing of SAEs of Subjects at Mexico sites | Report |
| | 109 | | | Listing of SAES of Subjects at Mexico Siles | requirement |
| Listing - | 103 | Safety- | AE8 | | New Output |
| Other | | Continuation | ALU | Listing of SAEs of Subjects - Continuation | New Output |
| Outer | 110 | Phase | | Phase | |

| Virology | Virology | | | | |
|---|---|---|---|---|---|
| Туре | No. | Population | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming<br>Notes |
| Table | 4.9 | CVW-<br>Continuation<br>Phase | Same shell as week 48, Table 4.7 | Summary of Subject Accountability:<br>Genotypes Available Continuation Phase | |
| Table | 4.10 | CVW-<br>Continuation<br>Phase | Same shell as<br>week 48,<br>Table 4.8 | Summary of Subject Accountability:<br>Phenotypes Available- Continuation<br>Phase | |
| Table | 4.11 | CVW-<br>Continuation<br>Phase | Same shell as<br>week 48,<br>Table 4.1 | Summary of INI Mutations at Baseline and Time of CVW- Continuation Phase | |
| Table | 4.12 | CVW-<br>Continuation<br>Phase | Same shell as<br>week 48,<br>Table 4.2 | Summary of Major Mutations of NRTI,<br>NNRTI and PI Classes by region at<br>Baseline and Time of CVW- Continuation<br>Phase | |
| Table | 4.13 | CVW-<br>Continuation<br>Phase | Same shell as<br>week 48,<br>Table 4.3 | Summary of Genotype at Baseline and Time of CVW by Genotypic Cut-Off-Continuation Phase | |
| Table | 4.14 | CVW-<br>Continuation<br>Phase | Same shell as<br>week 48,<br>Table 4.4 | Summary of Phenotype at Time of CVW by Phenotypic Cut-off- Continuation Phase | |
| Table | 4.15 | CVW-<br>Continuation<br>Phase | Same shell as<br>week 48,<br>Table 4.5 | Summary of Phenotype at Time of CVW by Number of Drugs to Which Subject are Resistant- Continuation Phase | |
| Table | 4.16 | CVW-<br>Continuation<br>Phase | Same shell as<br>week 48,<br>Table 4.6 | Summary of Fold Change to DTG, 3TC at Time of CVW- Continuation Phase | |
| Listing-<br>Other | 111 | ITT-E-<br>Continuation<br>Phase | See Section<br>15.17.16 | Listing of All Genotypic Data – CVWs-<br>Continuation Phase | |
| Listing-<br>Other | 112 | CVW-<br>Continuation<br>Phase | See Section<br>15.17.16 | Listing of All Genotypic Data – pPVWs-<br>Continuation Phase | |
| Listing-<br>Other | 113 | CVW-<br>Continuation<br>Phase | See Section<br>15.17.16 | Listing of Genotype by Genotypic Cut-Off – CVWs- Continuation Phase | |
| Listing-<br>Other | 114 | CVW-<br>Continuation<br>Phase | See Section<br>15.17.16 | Listing of Genotype by Genotypic Cut-Off – pPVWs- Continuation Phase | |
| Listing-<br>Other | 115 | CVW-<br>Continuation<br>Phase | See Section<br>15.17.16 | Listing of All Phenotypic Data - CVWs-<br>Continuation Phase | |

| Virology | Virology | | | |
|---|---|---|---|---|
| Listing-<br>Other | 116 | CVW-<br>Continuation<br>Phase | See Section<br>15.17.16 | Listing of All Phenotypic Data - pPVWs-<br>Continuation Phase |
| Listing-<br>Other | 117 | CVW-<br>Continuation<br>Phase | See Section<br>15.17.16 | Listing of Replication Capacity - CVWs-<br>Continuation Phase |
| Listing-<br>Other | 118 | CVW-<br>Continuation<br>Phase | See Section<br>15.17.16 | Listing of Replication Capacity - pPVWs-<br>Continuation Phase |
| Listing-<br>Other | 119 | CVW-<br>Continuation<br>Phase | See Section<br>15.17.16 | Listing of Net Assessment Score - CVWs-<br>Continuation Phase |
| Listing-<br>Other | 120 | CVW-<br>Continuation<br>Phase | See Section<br>15.17.16 | Listing of Net Assessment Score - pPVWs- Continuation Phase |
| Listing-<br>Other | 121 | CVW-<br>Continuation<br>Phase | See Section<br>15.17.16 | Listing of Genotypic and Phenotypic Data<br>for Subjects with Confirmed Virologic<br>Withdrawal Criteria- Continuation Phase |
| Listing-<br>Other | 122 | CVW-<br>Continuation<br>Phase | See Section<br>15.17.16 | Listing of Genotypic and Phenotypic Data<br>for Subjects with Potential Precautionary<br>Virologic Withdrawal Criteria-<br>Continuation Phase |

| Other analyses (Health Outcomes) | | | | | |
|---|---|---|---|---|---|
| Туре | No. | Population | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming<br>Notes |
| Table | 6.14 | ITT-E -<br>Continuation<br>Phase | Same shell as<br>week 48, Table<br>6.8 | Summary of SDM bother score Change from Baseline by Visit- Continuation Phase | |

#### 15.17. Appendix 17: List of Data Displays

#### 15.17.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------|-------------|-------------|
| Study Population | 1.01 to 1.n | 1.01 to 1.n |
| Efficacy | 2.01 to 2.n | 2.01 to 2.n |
| Safety | 3.01 to 3.n | 3.01 to 3.n |
| Virology | 4.01 to 4.n | 4.01 to 4.n |
| Pharmacokinetic | 5.01 to 5.n | 5.01 to 5.n |
| Health Outcomes | 6.01 to 6.n | 6.01 to 6.n |
| Section Listings | | ings |
| ICH Listings | 1 to x | |
| Other Listings | y t | 0 Z |

#### 15.17.2. Mock Example Shell Referencing

Non- GSK Statistical Display Standard specifications will be referenced as indicated and if required example mock-up displays provided in Appendix 18: Example Mock Shells for Data Displays.

| Section | Figure | Table | Listing |
|------------------------------------|----------|----------|----------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Efficacy | EFF_Fn | EFF_Tn | EFF_Ln |
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |
| Pharmacokinetic | PK_Fn | PK_Tn | PK_Ln |
| Population Pharmacokinetic (PopPK) | POPPK_Fn | POPPK_Tn | POPPK_Ln |
| Pharmacodynamic and / or Biomarker | PD_Fn | PD_Tn | PD_Ln |
| Pharmacokinetic / Pharmacodynamic | PKPD_Fn | PKPD_Tn | PK/PD_Ln |

#### NOTES:

 Non-Standard displays are indicated in the 'GSK Statistical Display Standard/ Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

#### 15.17.3. Deliverables

| Delivery [Priority] [1] | Description |
|-------------------------|------------------------------------------------|
| DS [X] | During Study |
| IA SAC [X] | Interim Analysis Statistical Analysis Complete |
| SAC [X] | Final Statistical Analysis Complete |

#### NOTES:

1. Indicates priority (i.e. order) in which displays will be generated for the reporting effort

## 15.17.4. Study Population Tables

Note that where the Deliverable column states 'All', this refers to all reporting efforts i.e. Weeks 24 and 48.

| Study | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK<br>Statistical<br>Display<br>Standard/<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | | | | |
| 1.1. | ITT-E | ES1 | Summary of Subject Status and Subject Disposition by Relationship to COVID-19 Pandemic | ICH E3, FDAAA, EudraCT Present by "Not Related to COVID-19" and "Related to COVID-19" and Overall | All |
| 1.2. | Screened | ES6 | Summary of Screening Status and Reasons for Screen Failure | Journal Requirements | All |
| 1.3. | Screened | NS1 | Summary of Number of Subjects Enrolled by Country and Site ID | EudraCT/Clinical Operations Repeat by ITT-E population for Disclosure purpose. Add Table 1.3.1 | All |
| 1.4. | ITT-E | POP_T1 | Summary of Reasons for Withdrawal by Visit | ICH E3 | All |
| 1.5. | ITT-E | POP_T13 | Summary of Misrandomized Strata or Treatment | | All |
| 1.6. | ITT-E | POP_T9 | Summary of Number of Subjects Attending Nominal and Actual Analysis Visits | | All |

| Study | Population Ta | bles | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Statistical Display Standard/ Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Protoc | col Deviation | | | | |
| 1.7. | ITT-E | DV1 | Summary of Important Protocol Deviations by Relationship to COVID-19 | ICH E3 Present by "Not Related to COVID-19" and "Related to COVID-19" and Overall | All |
| 1.8. | ITT-E | DV1 | Summary of Protocol Deviations Leading to Exclusion from the Per-Protocol Population | GSK Statistical Display Standard | All |
| 1.9. | | | | Will be combined with Table 1.7 | |
| Popula | ation Analysed | l | | | |
| 1.10. | Screened | SP1 | Summary of Study Populations | GSK Statistical Display Standard | All |
| Demo | graphic and Ba | aseline Characte | eristics | | |
| 1.11. | ITT-E | DM1 | Summary of Demographic Characteristics | ICH E3, FDAAA, EudraCT | All |
| 1.12. | Screened | DM11 | Summary of Age Ranges | EudraCT | All |
| 1.13. | | | | No longer required as it is part of 1.14 | |
| 1.14. | ITT-E | DM6 | Summary of Race and Racial Combinations Details | ICH E3, FDA, FDAAA, EudraCT | All |
| 1.15. | ITT-E | BASELINE3 | Summary of Hepatitis Status at Entry | | All |
| 1.16. | ITT-E | CDC1 | Summary of CDC Classification of HIV Infection at Baseline | | All |
| 1.17. | ITT-E | RF1 | Summary of HIV Risk Factors | | All |

| Study | Population Ta | bles | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Statistical Display Standard/ Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.18. | ITT-E | BASELINE4 | Summary of Screening and Baseline Cardiovascular Risk Assessments | GSK Statistical Display Standard | All |
| 1.19. | ITT-E | BASELINE2 | Summary of Distribution of CD4+ Cell Count (cells/mm^3) Results at Screening and Baseline | | All |
| 1.20. | ITT-E | BASELINE1 | Summary of Distribution of Quantitative Plasma HIV-1 RNA Results at Baseline | | All |
| Prior a | and Concomita | nt Medications, | Medical Conditions | | · |
| 1.21. | ITT-E | MH1 | Summary of Current Medical Conditions | ICH E3 | All |
| 1.22. | ITT-E | MH1 | Summary of Past Medical Conditions | ICH E3 | All |
| 1.23. | ITT-E | CM1 | Summary of Concomitant Medications by Ingredient ATC Level 1 | ICH E3 | All |
| 1.24. | ITT-E | CA1 | Summary of Antiretroviral Therapy Stopped Prior to Screening | | All |
| 1.25. | ITT-E | CA1 | Summary of Antiretroviral Therapy Received at Screening | | All |
| 1.26. | | | | Covered in 1.25 | |
| 1.27. | ITT-E | CA1 | Summary of On-Treatment Antiretroviral Therapy Starting after Day 1 | | All |
| 1.28. | ITT-E | CA1 | Summary of Antiretroviral Therapy Starting after Treatment Discontinuation | | All |

| Study Population Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK<br>Statistical<br>Display<br>Standard/<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.29. | | | | Covered in 1.28 | |
| 1.30. | ITT-E | CA2 | Summary of Baseline Third Agent Class | | All |
| 1.31. | ITT-E | POP_T12 | Summary of Time since First Antiretroviral Therapy until Day 1 | | All |
| 1.32. | ITT-E | POP_T7 | Summary of History of Depression and Anxiety at Baseline | | All |
| Impac | t of COVID-19 | Pandemic | | | |
| 1.33. | ITT-E | PAN4 | Summary of Visits impacted by COVID-19 Pandemic | | All |
| 1.34. | ITT-E | SD4 | Summary of Treatment Status and Reasons for Discontinuation of Study Treatment by Relationship to COVID-19 Pandemic | Summarise by: Related to COVID-19 Not related to COVID-19 | All |
| 1.35. | Screened | NS1 | Summary of Recruitment by Country and Site Before & After Implementation of Pandemic Measures | The dates when implementation of pandemic measures began will be available in HARP dataset and should be used to define before & after implementation of pandemic measures | All |

## 15.17.5. Study Population Figures

| Impact | Impact of COVID-19 Pandemic : Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Statistical Display Standard/ TST ID / Example Shell | Title | Programming<br>Notes | Deliverable<br>[Priority] |
| Visits impacted by COVID-19 Pandemic | | | | | |
| 1.1. | ITT-E | PAN8 | Visits impacted by COVID-19 Pandemic | | All |

15.17.6. Efficacy Tables

| Efficacy: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Populati<br>on | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Primary I | Efficacy Ana | alysis | | | |
| 2.1. | ITT-E | EFF_T1 | Summary of Analysis for Percent of Subjects with Plasma HIV-1 RNA ≥ 50 c/mL at Week X – Snapshot Analysis | | All |
| 2.2. | Per-<br>Protocol | EFF_T1 | Summary of Analysis for Percent of Subjects with Plasma HIV-1 RNA ≥ 50 c/mL at Week X – Snapshot Analysis | | All |
| 2.3. | ITT | EFF_T1 | Summary of Analysis for Percent of Subjects with Plasma HIV-1 RNA ≥ 50 c/mL at Week X – Snapshot Analysis | | All |
| 2.4. | ITT-E | EFF_T1 | Summary of Analysis for Percent of Subjects with Plasma HIV-1 RNA ≥ 50 c/mL at Week X – Snapshot Analysis | | All |

| Efficacy: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Populati<br>on | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| | | | (Sparse Data Sensitivity Analysis) | | |
| Seconda | ary Efficacy | Analyses | | | |
| 2.5. | ITT-E | EFF_T1 | Summary of Analysis for Percent of Subjects with Plasma HIV-1 RNA <50 c/mL at Week X – Snapshot Analysis | | All |
| 2.6. | ITT-E | EFF_T2 | Summary of Study Outcomes (Plasma HIV-1 RNA ≥ / < 50 c/mL) at Week X – Snapshot Analysis | | All |
| 2.7. | Per-<br>Protocol | EFF_T2 | Summary of Study Outcomes (Plasma HIV-1 RNA ≥ / < 50 c/mL) at Week X – Snapshot Analysis | | All |
| 2.8. | ITT | EFF_T2 | Summary of Study Outcomes (Plasma HIV-1 RNA ≥ / < 50 c/mL) at Week X – Snapshot Analysis | | All |
| 2.9. | ITT-E | EFF_T2a | Summary of Study Outcomes (Plasma HIV-1 RNA ≥ / < 50 c/mL) at Week X – Modified Snapshot Analysis | | All |
| 2.10. | ITT-E | EFF_T5 | Summary of Percent of Subjects with Plasma HIV-1 RNA ≥50 c/mL by Visit – Snapshot Analysis | | All |
| 2.11. | ITT-E | EFF_T5 | Summary of Percent of Subjects with Plasma HIV-1 RNA <50 c/mL by Visit – Snapshot Analysis | | All |
| 2.12. | ITT-E | EFF_T6 | Summary of Percent of Subjects with Plasma HIV-1 RNA <50 c/mL at Week X by Subgroup – Snapshot Analysis | | All |
| 2.13. | ITT-E | EFF_T3 | Summary of Study Outcomes (Plasma HIV-1 RNA ≥ / < 50 c/mL) at Week X by Subgroup - Snapshot Analysis | | All |
| 2.14. | ITT-E | EFF_T8 | Summary of Change from Baseline in Plasma HIV-1 RNA (log10 c/mL) by Visit | | All |

| Efficacy | : Tables | | | | |
|---|---|---|---|---|---|
| No. | Populati<br>on | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.15. | ITT-E | EFF_T9 | Summary of Change from Baseline in in CD4+ count (cells/mm3) by Visit | | All |
| 2.16. | ITT-E | EFF_T9 | Summary of Change from Baseline in in CD4+/CD8+ count ratio (cells/mm3) by Visit | | All |
| 2.17. | ITT-E | EFF_T14 | Summary of Change from Baseline in CD4+/CD8+ Count Ratio (cells/mm3) at Week X by Subgroup | | All |
| 2.18. | ITT-E | EFF_T10 | Summary of Post-Baseline HIV-1 Associated Conditions Including Recurrences | | All |
| 2.19. | ITT-E | EFF_T10 | Summary of Post-Baseline HIV-1 Associated Conditions Excluding Recurrences | | All |
| 2.20. | ITT-E | EFF_T11 | Summary of Post-Baseline HIV-1 Disease Progressions | | All |
| 2.21. | ITT-E | EFF_T12 | Cumulative Proportion of Subjects Meeting Confirmed Virologic Withdrawal Criteria by Visit | | All |
| 2.22. | ITT-E | EFF_T13 | Distribution of Quantitative Plasma HIV-1 RNA Results at Suspected and Confirmed Virologic Withdrawal | | All |
| 2.23. | ITT-E | EFF_T14 | Summary of Change from Baseline in in CD4+ count (cells/mm3) at Week X by Subgroup | | All |
| 2.24. | ITT-E | EFF_T15 | Summary of Kaplan-Meier Estimates of Proportion of Subjects Without Confirmed Virologic Withdrawal at Week X - Treatment Related Discontinuation = Failure | | All |
| 2.25. | ITT-E | EFF_T15 | Summary of Kaplan-Meier Estimates of Proportion of Subjects Without Confirmed Virologic Withdrawal at Week X - Efficacy Related Discontinuation = Failure | | All |

| Efficacy | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Populati<br>on | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.26. | ITT-E | EFF_T1 | Summary of Analysis for percent of Subjects with Plasma HIV-1 RNA <40 c/mL at Week X – Snapshot Analysis | | All |
| 2.27. | ITT-E | EFF_T1 | Summary of Analysis for Percent of Subjects with Plasma HIV-1 RNA <40 c/mL and Target Not Detected Status at Week X - Snapshot Analysis - ITT-E | | All |
| 2.28. | ITT-E | EFF_T5 | Summary of Percent of Subjects with Plasma HIV-1 RNA <40 c/mL by Visit - Snapshot Analysis | | All |
| 2.29. | ITT-E | EFF_T5 | Summary of Percent of Subjects with Plasma HIV-1 RNA <40 c/mL and Target Not Detected Status by Visit - Snapshot Analysis | | All |
| 2.30. | ITT-E | EFF_T2 | Summary of Study Outcomes (<40 c/mL and Target Not Detected Status) at Week X - Snapshot | | All |
| 2.31. | ITT-E | EFF_T6 | Summary of Percent of Subjects with Plasma HIV-1 RNA <40 c/mL and Target Not Detected Status at Week X by Baseline Third Agent Class -Snapshot Analysis - ITT-E | | All |
| 2.32. | ITT-E | EFF_T2 | Summary of Study Outcomes (<40 c/mL) at Week X - Snapshot | | |

## 15.17.7. Efficacy Figures

| Efficac | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK<br>Statistical<br>Display<br>Standard/<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Secon | Secondary Efficacy Analyses | | | | |
| 2.1. | ITT-E | EFF_F2 | Unadjusted Treatment Difference in Percent (95% CI) of Subjects with HIV-1 RNA <50 c/mL at Week X by Subgroup – Snapshot Analysis | | All |
| 2.2. | ITT-E | EFF_F3 | Individual Plasma HIV-1 RNA and CD4+ Profiles by Visit for subjects with at least one viral load ≥50 c/mL | | All |
| 2.3. | ITT-E | EFF_F4 | Kaplan-Meier Plot of Time to Failure - Treatment Related Discontinuation = Failure (TRDF) | | All |
| 2.4. | ITT-E | EFF_F4 | Kaplan-Meier Plot of Time to Failure - Efficacy Related Discontinuation = Failure (ERDF) | | All |

## 15.17.8. Safety Tables

| Safety | : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK<br>Statistical<br>Display<br>Standard/<br>Example<br>Shell | Title | Programming<br>Notes | Deliverable<br>[Priority] |
| Expos | ure | | | | |
| 3.1. | Safety | SAFE_T1 | Summary of Extent of Exposure Study Treatment- Randomized Phase | ICH E3 | All |
| Advers | se Events | | | | |
| 3.2. | Safety | AE1 | Summary of All Adverse Events by System Organ Class and Preferred Term | ICH E3 | All |
| 3.3. | Safety | AE5B | Summary of Adverse Events by System Organ Class, Maximum Toxicity and Subgroups | | All |
| 3.4. | Safety | AE5A | Summary of All Adverse Events by Maximum Grade | ICH E3 | All |
| 3.5. | Safety | AE3 | Summary of Common (>=2%) Adverse Events by Overall Frequency | ICH E3 | All |
| 3.6. | Safety | AE3 | Summary of Common (>=2%) Grade 2-5 Adverse Events by Overall Frequency | ICH E3 | All |
| 3.7. | Safety | AE1 | Summary of All Drug-Related Adverse Events by System Organ Class and Preferred Term | ICH E3 | All |

| Safety | Safety: Tables | | | | | | |
|---|---|---|---|---|---|--|--|
| No. | Population | GSK Statistical Display Standard/ Example Shell | Title | Programming<br>Notes | Deliverable<br>[Priority] | | |
| 3.8. | Safety | AE5A | Summary of All Drug-Related Adverse Events by System Organ Class and Preferred Term and Maximum Grade | ICH E3 | All | | |
| 3.9. | Safety | AE15 | Summary of Common (>=2%) Non-serious Adverse Events by System Organ Class and Preferred Term (Number of Subject and Occurrences) | FDAAA, EudraCT | All | | |
| 3.10. | Safety | AE3 | Summary of Common (>=0.5%) Drug-Related Grade 2-5 Adverse Events by Overall Frequency | ICH E3 | All | | |
| 3.11. | Safety | SAFE_T16 | Summary of Subjects with Any Adverse Events by Visit | | All | | |
| 3.12. | Safety | AE20 | Summary of Serious Fatal and Non-Fatal Drug-Related Adverse Events by Overall Frequency | Plain<br>Language<br>Summary<br>requirements | All | | |
| Seriou | s and Other S | ignificant Adver | se Events | | | | |
| 3.13. | Safety | AE16 | Summary of Serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | FDAAA, EudraCT | All | | |
| 3.14. | Safety | AE1 | Summary of Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study by System Organ Class and Preferred Term /by Overall Frequency | GSK Statistical<br>Display Standard | All | | |
| 3.15. | Safety | AE5A | Summary of Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study by Maximum Grade | | All | | |
| Safety | : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK<br>Statistical<br>Display<br>Standard/<br>Example<br>Shell | Title | Programming<br>Notes | Deliverable<br>[Priority] |
| 3.16. | Safety | AE1 | Summary of Serious Drug-Related Adverse Events by System Organ Class | Plain<br>Language<br>Summary<br>requirements. | All |
| 3.17. | Safety | SAFE_T2 | Summary of Cumulative Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study by Visit | | All |
| Impact | of Covid-19 on | Assessment of S | afety Based on COVID-19 eCRF | | |
| 3.18. | Safety | PAN1 | Number of Subjects with an Adverse Event of Suspected, Probable, Confirmed for COVID-19 Infection | GSK Statistical<br>Display Standard | All |
| 3.19. | | | | Covered in 3.18 | |
| Labora | tory: Chemist | try | | | |
| 3.20. | Safety | LB1 | Summary of Chemistry Changes from Baseline by Visit | ICH E3 | All |
| 3.21. | Safety | SAFE_T17 | Summary of Chemistry by Visit | ICH E3 | All |
| 3.22. | Safety | SAFE_T13 | Summary of AST, ALT and Total Bilirubin Maximum Post-Baseline Emergent Toxicity by Baseline Hepatitis C Status | ICH E3 | All |
| 3.23. | Safety | LIVER1 | Summary of Liver Monitoring/Stopping Event Reporting | GSK Statistical<br>Display Standard | |

| opulation | GSK<br>Statistical<br>Display<br>Standard/<br>Example<br>Shell | Title | Programming<br>Notes | Deliverable |
|---|---|---|---|---|
| nu Linida | | | | [Priority] |
| ry: Lipids | | | | |
| Safety | LB1 | Summary of Fasting Lipids by Visit | display both<br>mmol/L and<br>mg/DL | All |
| Safety | LB1 | Summary of Change from Baseline in Fasting Lipids by Visit | display both<br>mmol/L and<br>mg/DL | All |
| Safety | SAFE_T5 | Summary of Changes in NCEP Lipid Baseline Category to Week X Category-Shift Table | display both<br>mmol/L and<br>mg/DL | All |
| Safety | SAFE_T7b | Statistical Analysis of Change from Baseline in Fasting Lipids at Week X - Multiple Imputed Loge Transformed Data - MAR | display both<br>mmol/L and<br>mg/DL | All |
| Safety | SAFE_T7b | Statistical Analysis of Change from Baseline in Fasting Lipids at Week X - Loge Transformed Data – MMRM/ANCOVA | display both<br>mmol/L and<br>mg/DL<br>ANCOVA-<br>Week 24<br>MMRM-Week<br>48 | All |
| | Safety Safety Safety | Safety LB1 Safety SAFE_T5 Safety SAFE_T7b | Safety LB1 Summary of Change from Baseline in Fasting Lipids by Visit Safety SAFE_T5 Summary of Changes in NCEP Lipid Baseline Category to Week X Category-Shift Table Safety SAFE_T7b Statistical Analysis of Change from Baseline in Fasting Lipids at Week X - Multiple Imputed Loge Transformed Data - MAR Safety SAFE_T7b Statistical Analysis of Change from Baseline in Fasting Lipids at Week X - Loge Transformed Data - MMRM/ANCOVA | Safety LB1 Summary of Fasting Lipids by Visit mmol/L and mg/DL Safety LB1 Summary of Change from Baseline in Fasting Lipids by Visit display both mmol/L and mg/DL Safety SAFE_T5 Summary of Changes in NCEP Lipid Baseline Category to Week X Category-Shift Table display both mmol/L and mg/DL Safety SAFE_T7b Statistical Analysis of Change from Baseline in Fasting Lipids at Week X - Multiple Imputed Loge Transformed Data - MAR Safety SAFE_T7b Statistical Analysis of Change from Baseline in Fasting Lipids at Week X - Multiple Imputed Loge Transformed Data - MAR Safety SAFE_T7b Statistical Analysis of Change from Baseline in Fasting Lipids at Week X - Statistical Analysis of Change from Baseline in Fasting Lipids at Week X - Loge Transformed Data - MMRM/ANCOVA Missing Data - Missing Lipids at Week X - Missing Lipids at W |

| Safety | : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Statistical Display Standard/ Example Shell | Title | Programming<br>Notes | Deliverable<br>[Priority] |
| 3.29. | Safety | LB1 | Summary of Hematology Changes from Baseline by Visit | ICH E3 | All |
| 3.30. | Safety | SAFE_T17 | Summary of Hematology by Visit | | All |
| Labora | tory: Urinalys | sis | | | |
| 3.31. | Safety | LB1 | Summary of Urinalysis Changes from Baseline by Visit | ICH E3 | All |
| 3.32. | Safety | SAFE_T17 | Summary of Urinalysis by Visit | | All |
| Labora | tory: Hepatob | oiliary (Liver) | | | |
| 3.33. | Safety | LIVER10 | Summary of Subjects Meeting Hepatobiliary Abnormality Criteria – All Post-<br>Baseline Abnormalities | GSK Statistical<br>Display Standard | All |
| Bioma | rkers (Bone, R | Renal and Inflam | matory) | | |
| 3.34. | Safety | LB1 | Summary of Change from Baseline in Bone Biomarkers by Visit | | All |
| 3.35. | Safety | LB1 | Summary of Change from Baseline in Renal Biomarkers by Visit | | All |
| 3.36. | Safety | LB1 | Summary of Change from Baseline in Renal Biomarkers by Visit- Loge Transformed Data | | All |
| 3.37. | Safety | LB1 | Summary of Change from Baseline in Inflammatory Biomarkers - Loge Transformed Data | | All |
| 3.38. | Safety | SAFE_T7b | Statistical Analysis of Change from Baseline Bone Biomarkers at Week X – MMRM/ANCOVA | ANCOVA-<br>Week 24<br>MMRM-Week<br>48 | All |

| Safety | : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Statistical Display Standard/ Example Shell | Title | Programming<br>Notes | Deliverable<br>[Priority] |
| 3.39. | Safety | SAFE_T7a | Statistical Analysis of Change from Baseline in Renal Biomarkers at Week X – MMRM/ANCOVA | ANCOVA-<br>Week 24<br>MMRM-Week<br>48 | All |
| 3.40. | Safety | SAFE_T7b | Statistical Analysis of Change from Baseline in Renal Biomarkers at Week X - Loge Transformed Data - MMRM /ANCOVA | ANCOVA-<br>Week 24<br>MMRM-Week<br>48 | All |
| 3.41. | Safety | SAFE_T7b | Statistical Analysis of Change from Baseline in Inflammatory Biomarkers at Week X - Loge Transformed Data – MMRM/ANOCVA | ANCOVA-<br>Week 24<br>MMRM-Week<br>48 | All |
| Weight | t, BMI, HOMA- | IR and HbA1c | | | |
| 3.42. | Safety | SAFE_T17 | Summary of Weight (kg) by Visit | | All |
| 3.43. | Safety | LB1 | Summary of Change from Baseline in Weight (kg) by Visit | | All |
| 3.44. | Safety | SAFE_T7 | Statistical Analysis of Change from Baseline in Weight (kg) by Visit- MMRM | | All |
| 3.45. | Safety | SAFE_T18 | Summary of Proportion of Subjects with Change from Baseline in Weight (>=3% and >=10%) at Week X | | All |
| 3.46. | Safety | SAFE_T17 | Summary of BMI (kg/m2) by Visit | | All |

| Safety | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK<br>Statistical<br>Display<br>Standard/<br>Example<br>Shell | Title | Programming<br>Notes | Deliverable<br>[Priority] |
| 3.47. | Safety | LB1 | Summary of Change from Baseline in BMI (kg/m2) by Visit | | All |
| 3.48. | Safety | SAFE_T5 | Summary of Changes in BMI (kg/m2) from Baseline to Week X -Shift Table | | All |
| 3.49. | Safety | SAFE_T7 | Statistical Analysis of Change from Baseline in BMI (kg/m2) by Visit- MMRM | | All |
| 3.50. | Safety | SAFE_T17 | Summary of HOMA-IR by Visit | | All |
| 3.51. | Safety | LB1 | Summary of Change from Baseline in HOMA-IR by Visit - Loge Transformed Data | | All |
| 3.52. | Safety | SAFE_T7 | Statistical Analysis of Change from Baseline in HOMA-IR by Visit- Loge Transformed Data - MMRM | | All |
| 3.53. | Safety | SAFE_T19 | Statistical Analysis of Variables Associated with ≥2 HOMA-IR at Week X – Logistic Regression | | All |
| 3.54. | Safety | SAFE_T19 | Statistical Analysis of Variables Associated with ≥3 HOMA-IR at Week X – Logistic Regression | | All |
| 3.55. | Safety | SAFE_T19 | Statistical Analysis of Variables Associated with ≥4 HOMA-IR at Week X – Logistic Regression | | All |
| 3.56. | Safety | SAFE_T17 | Summary of HbA1c by Visit | | All |
| 3.57. | Safety | LB1 | Summary of Change from Baseline in HbA1c by Visit | | All |
| 3.58. | Safety | SAFE_T7 | Statistical Analysis of Change from Baseline in HbA1c by Visit - MMRM | | All |

| Safety | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK<br>Statistical<br>Display<br>Standard/<br>Example<br>Shell | Title | Programming<br>Notes | Deliverable<br>[Priority] |
| Other | Safety Analys | es | | | |
| 3.59. | Safety | SAFE_T8 | Summary of True Positive Suicidal Indication Alerts Based on eCSSRS by Visit | | All |
| 3.60. | Safety | SAFE_T9 | Summary of Subjects with eCSSRS Suicidal Ideation or Behaviour at Baseline | | All |
| 3.61. | Safety | SAFE_T9 | Summary of Subjects with Post Baseline eCSSRS Suicidal Ideation or Behaviour | | All |
| 3.62. | Safety | SAFE_T10 | Summary of Characteristics of Post Baseline Adverse Events of Special Interest | Present each AESI in a separate table. Table numbering should be from 3.621 to 3.628 | All |

## 15.17.9. Safety Figures

| Safe | Safety: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK<br>Statistical<br>Display<br>Standard/<br>Example<br>Shell | Title | Programming<br>Notes | Deliverable<br>[Priority] |
| Adve | rse Events | | | | |
| 3.1. | Safety | AE10 | Plot of Common (>=2%) Adverse Events and Relative Risk | | All |
| Labo | ratory: Bioma | arkers | | | |
| 3.2. | Safety | LIPID7 | Heatmap Plot of NCEP Categories in Lipids Over Time | | All |
| 3.3. | Safety | SAFE_F2 | Line Plot of Adjusted Mean (95% CI) Change from Baseline in Renal Biomarkers<br>Over Time — MMRM | | All |
| 3.4. | Safety | SAFE_F3 | Line Plot of Ratio of Geometric Means (95% CI) in Renal Biomarkers Over Time - Loge Transformed Data - MMRM | | All |
| 3.5. | Safety | SAFE_F2 | Line Plot of Adjusted Mean (95% CI) of Change from Baseline in Bone Biomarkers Over Time — MMRM | | All |
| 3.6. | Safety | SAFE_F2 | Line Plot of Ratio of Geometric Means (95% of CI) in Inflammatory Biomarkers<br>Over Time - Loge Transformed - MMRM | | All |
| 3.7. | Safety | SAFE_F5 | Line Plot of Adjusted Mean (95% CI) of Change from Baseline in Weight (kg) Over Time — MMRM | | All |
| 3.8. | Safety | SAFE_F5 | Line Plot of Adjusted Mean (95% CI) of Change from Baseline in BMI (kg/m2) Over Time — MMRM | | All |

| Safet | Safety: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK<br>Statistical<br>Display<br>Standard/<br>Example<br>Shell | Title | Programming<br>Notes | Deliverable<br>[Priority] |
| 3.9. | Safety | SAFE_F2 | Line Plot of Ratio of Geometric Means (95% of CI) in HOMA-IR Over Time - Loge Transformed Data – MMRM | | All |
| 3.10. | Safety | SAFE_F5 | Line Plot of Adjusted Mean (95% CI) of Change from Baseline in HbA1c Over Time — MMRM | | All |
| Othe | r Safety | | | | |
| 3.11. | Safety | LIPID7 | Heatmap Plot of BMI (kg/m2) Categories Over Time | | All |
| 3.12. | Safety | LIVER9 | Scatter Plot of Maximum ALT vs. Maximum Total Bilirubin | | All |

## 15.17.10. Virology Tables

| Viro | Virology: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK<br>Statistical<br>Display<br>Standard/<br>TST ID /<br>Example<br>Shell | Title | Programming<br>Notes | Deliverable<br>[Priority] |
| 4.1. | CVW | VIR_T1 | Summary of INI Mutations at Baseline and Time of CVW at or prior to Week X | | All |
| 4.2. | CVW | VIR_T2 | Summary of Major Mutations of NRTI, NNRTI and PI Classes by region at Baseline and Time of CVW at or prior to Week X | | All |
| 4.3. | CVW | VIR_T3 | Summary of Genotype at Baseline and Time of CVW by Genotypic Cut-Off at or prior Week X | | All |
| 4.4. | CVW | VIR_T4 | Summary of Phenotype at Time of CVW by Phenotypic Cut-off at or prior Week X | | All |
| 4.5. | CVW | VIR_T5 | Summary of Phenotype at time of CVW by Number of Drugs to Which Subject are Resistant at or prior Week X | | All |
| 4.6. | CVW | VIR_T6 | Summary of Fold Change to DTG, 3TC at - Time of CVW at or prior to Week X | | All |
| 4.7. | CVW | VIR_T7 | Summary of Subject Accountability: Genotypes Available at or prior to Week X | | All |
| 4.8. | CVW | VIR_T8 | Summary of Subject Accountability: Phenotypes Available at or prior to Week X | | All |

#### 15.17.11. Pharmacokinetic Tables

There is no pharmacokinetic analysis planned in this study.

#### 15.17.12. Pharmacokinetic Figures

There is no pharmacokinetic analysis planned in this study.

#### 15.17.13. Health Outcomes Tables

| Health | Health Outcomes : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK<br>Statistical<br>Display<br>Standard/<br>TST ID /<br>Example<br>Shell | Title | Programming<br>Notes | Deliverable<br>[Priority] |
| Treatm | nent Satisfaction | on (HIVTSQ) | | | |
| 6.1. | ITT-E | THO1 | Summary of HIVTSQ Individual Item Scores by Visit | | All |
| 6.2. | ITT-E | THO2 | Summary of HIVTSQ Total Score, Lifestyle/Ease and General Satisfaction/Clinical Sub-score by Visit | | All |
| 6.3. | ITT-E | THO2 | Summary of Change from Baseline in HIVTSQ Total Score,<br>Lifestyle/Ease and General Satisfaction/Clinical Sub-score by Visit | | All |
| 6.4. | ITT-E | THO3 | Statistical Analysis of HIVTSQ Total Score, Lifestyle/Ease and General Satisfaction/Clinical Sub-score Change from Baseline - MMRM | | All |
| 6.5. | ITT-E | тноз | Statistical Analysis of HIVTSQ Total Score, Lifestyle/Ease and General Satisfaction/Clinical Sub-score Change from Baseline by Subgroups - MMRM | | All |

| Health | Outcomes : | Tables | | | |
|---|---|---|---|---|---|
| No. | Population | GSK<br>Statistical<br>Display<br>Standard/<br>TST ID /<br>Example<br>Shell | Title | Programming<br>Notes | Deliverable<br>[Priority] |
| Sympt | om Distress M | odule | | | |
| 6.6. | ITT-E | THO4 | Summary of SDM Symptom Count by Visit | | All |
| 6.7. | ITT-E | THO4 | Summary of SDM Symptom Bother Score by Visit | | All |
| 6.8. | ITT-E | THO4 | Summary of SDM Symptom Bother Score Change from Baseline by Visit | | All |
| 6.9. | ITT-E | THO5 | Percentage of Subjects with Each Type of Symptom as per the SDM by Visit | | All |
| 6.10. | ITT-E | THO6 | Percentage of Subjects in SDM Symptom Bother Score Categories by Visit | | All |
| 6.11. | ITT-E | THO3 | Statistical Analysis of Change from Baseline in SDM Symptom Bother Score at Week X– MMRM | | All |
| 6.12. | ITT-E | THO3 | Statistical Analysis of Change from Baseline in SDM Symptom Bother Score by Subgroups at Week X– MMRM | | All |
| Willing | Willingness to switch | | | | |
| 6.13. | ITT-E | THO8 | Summary of Reasons for Willingness to Switch | | All |

## 15.17.14. Health Outcomes Figures

| Heal | Health Outcomes : Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK<br>Statistical<br>Display<br>Standard/<br>TST ID /<br>Example<br>Shell | Title | Programming<br>Notes | Deliverable<br>[Priority] |
| Treat | tment Satisfact | tion (HIVTSQ) | | | |
| 6.1. | ITT-E | FHO1 | Line Plot of Adjusted Mean (95% CI) Change from Baseline in HIVTSQ Total Treatment Satisfaction Score, Lifestyle/Ease and General Satisfaction/Clinical Sub-score Over Time | | All |
| Sym | Symptom Distress Module | | | | |
| 6.2. | ITT-E | FHO1 | Line Plot of Adjusted Mean (95% CI) Change from Baseline in SDM Symptom Bother Score Over Time | | All |

## 15.17.15. ICH Listings

| ICH: | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK<br>Statistical<br>Display<br>Standard/<br>Example<br>Shell | Title | Programming<br>Notes | Deliverable [Priority] |
| Subj | ect Dispositio | on | | | |
| 1. | ITT-E | ES2 | Listing of Reasons for Study Withdrawal | ICH E3 | All |
| 2. | ITT-E | SD2 | Listing of Reasons for Study Treatment Discontinuation | ICH E3 | All |
| Prot | Protocol Deviation | | | | |
| 3. | ITT-E | DV2 | Listing of Important Protocol Deviations | ICH E3. Listing to be<br>run regardless of<br>relationship to<br>COVID-19 | All |
| 4. | ITT-E | IE4 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | ICH E3 | All |
| Pop | ulations Analy | /sed | | | |
| 5. | ITT-E | SP3a | Listing of Protocol Deviations Leading to Exclusion from the Per Protocol Population | ICH E3 | All |
| 6. | ITT-E | DV2 | Listing of Protocol Deviations Related to COVID-19 | ICH E3 Include a column to flag Important PDs | All |
| Dem | ographic and | Baseline Ch | naracteristics | | |

| ICH: | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK<br>Statistical<br>Display<br>Standard/<br>Example<br>Shell | Title | Programming<br>Notes | Deliverable [Priority] |
| 7. | ITT-E | DM2 | Listing of Demographic Characteristics | ICH E3 | All |
| 8. | ITT-E | DM10 | Listing of Race | ICH E3 | All |
| Effic | асу | | | | |
| 9. | ITT-E | EFF_L1 | Listing of Study Outcome (≥ / < 50 c/mL) at Week 48 – Snapshot Analysis | | All |
| 10. | ITT-E | EFF_L2 | Listing of Quantitative and Qualitative Plasma HIV-1 RNA Data | | All |
| 11. | ITT-E | EFF_L1 | Listing of Study Outcome (≥ / < 50 c/mL) at Week 48 – Modified Snapshot Analysis | | All |
| Expo | Exposure and Treatment Compliance | | | | |
| 12. | Safety | EX3 | Listing of Exposure Data | ICH E3 | All |
| Adv | erse Events | | | | |
| 13. | Safety | AE8 | Listing of All Adverse Events | ICH E3 | All |
| 14. | Safety | AE14 | Listing of Reasons for Considering as a Serious Adverse Event | ICH E3 | All |
| 15. | Safety | AE8 | Listing of Adverse Events Leading to<br>Withdrawal from Study / Permanent<br>Discontinuation of Study Treatment | ICH E3 | All |

| ICH: | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK<br>Statistical<br>Display<br>Standard/<br>Example<br>Shell | Title | Programming<br>Notes | Deliverable [Priority] |
| 16. | Safety | PSRAE1 | Listing of Possible Suicidality-Related Adverse<br>Event Data: Event and Description (Section 1-<br>Section 2) | ICH E3 | All |
| 17. | Safety | PSRAE3 | Listing of Possible Suicidality-Related Adverse Event Data: Possible Cause(s) (Section 3) | | All |
| 18. | Safety | PSRAE4 | Listing of Possible Suicidality-Related Adverse Event Data (Section 4) | | All |
| 19. | Safety | PSRAE5 | Listing of Possible Suicidality-Related Adverse Event Data (Section 5- Section 8) | | All |
| All L | aboratory | | | | |
| 20. | Safety | LB5 | Listing of All Laboratory Data for Subjects with Any Value of Potential Clinical Importance | Include<br>Chemistry,<br>Hematology and<br>Lipids.<br>ICH E3 | All |
| 21. | Safety | LB5 | Listing of Urinalysis Data for Subjects with Any Value of Potential Clinical Importance | | All |
| Vital | Signs | | | | |
| 22. | Safety | VS4 | Listing of Vital Signs | ICH E3 | All |

## 15.17.16. Non-ICH Listings

| Non-IC | Non-ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Statistical Display<br>Standard/ Example Shell | Title | Programming<br>Notes | Deliverable<br>[Priority] |
| Study | Population | | | | |
| 23. | Screened | ES7 | Listing of Reasons for Screen Failure | Journal Guidelines<br>GSK Statistical Display<br>Standard | All |
| 24. | ITT | TA1 | Listing of Planned Randomized and Actual Strata and Treatment Assignments | | All |
| 25. | ITT | POP_L1 | Listing of Subjects Randomized but not Treated | | All |
| 26. | Screened | POP_L2 | Listing of Subjects Enrolled by Country and Site ID | | All |
| 27. | Screened | ES9 | Listing of Subjects Who Were Rescreened | | All |
| 28. | ITT-E | POP_L3 | Listing of Visit Dates | | All |
| 29. | Screened | POP_L4 | Listing of Study Populations | | All |
| 30. | ITT-E | BASELINE6 | Listing of Hepatitis Test Results at Entry | | All |
| 31. | ITT-E | CDC3 | Listing of CDC Classification of HIV Infection at Baseline | | All |

| Non-IC | Non-ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Statistical Display<br>Standard/ Example Shell | Title | Programming<br>Notes | Deliverable<br>[Priority] |
| 32. | ITT-E | RF2 | Listing of HIV Risk Factors | | All |
| 33. | ITT-E | BASELINE7 | Listing of Screening Cardiovascular Risk<br>Assessment Data | | All |
| 34. | ITT-E | MH2 | Listing of Current and Past Medical Conditions at Baseline | | All |
| 35. | ITT-E | POP_L7 | Listing of Relationship Between Concomitant ATC Level 1, Ingredient and Verbatim Text | | All |
| 36. | ITT-E | CM2 | Listing of Concomitant Medications | GSK Statistical Display<br>Standard | All |
| 37. | ITT-E | CM2 | Listing of Antiretroviral Therapy Stopped Prior to Screening | | All |
| 38. | ITT-E | CM2 | Listing of Antiretroviral Therapy Received at Screening | | All |
| 39. | ITT-E | CM2 | Listing of On-Treatment Antiretroviral Therapy<br>Starting after Day 1 | | All |
| 40. | ITT-E | CM2 | Listing of Antiretroviral Therapy Starting after Treatment Discontinuation | | All |
| 41. | ITT-E | POP_L8 | Listing of Relationship Between Concomitant ATC Level 4, Ingredient and Verbatim Text | | All |
| 42. | ITT-E | POP_L12 | Listing of Menopause History | | All |

| Non-IC | H: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Statistical Display<br>Standard/ Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Efficac | у | | | | • |
| 43. | ITT-E | VF4 | Listing of Plasma HIV-1 RNA data and CD4+ cell count data for subjects with Confirmed Virologic Withdrawal | | All |
| 44. | ITT-E | EFF_L4 | Listing of CD4+ Cell Count Data | | All |
| 45. | ITT-E | EFF_L5 | Listing of CD8+ and CD4+/CD8+ Cell Count Ratio Data | | All |
| 46. | ITT-E | HIV4 | Listing of Stage 3 HIV-1 Associated Conditions | | All |
| 47. | ITT-E | EFF_L6 | Listing of Subjects Treatment-related discontinuation = Failure (TRDF) | | All |
| 48. | ITT-E | EFF_L6 | Listing of Subjects Efficacy-related discontinuation = Failure (ERDF) | | All |
| Safety | | | | | • |
| 49. | Safety | EG3 | Listing of ECG Findings | | All |
| 50. | Safety | SAFE_L1 | Listing of Post Baseline Maximum ALT and Maximum Bilirubin | | All |
| 51. | Safety | SAFE_L2 | Listing of Subjects Meeting Hepatobiliary Abnormality Criteria – All Post-Baseline Abnormalities | | All |
| 52. | Safety | SAFE_L3 | Listing of eCSSRS Suicidal Ideation and Behaviour Data Alerts (4-9) | | All |
| 53. | Safety | SAFE_L4 | Listing of eCSSRS Suicidal Ideation and Behaviour Data | | All |

| Non-ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Statistical Display<br>Standard/ Example Shell | Title | Programming<br>Notes | Deliverable<br>[Priority] |
| 54. | Safety | SAFE_L5 | Listing of eCSSRS False Positive Alerts with Corresponding Reasons | | All |
| 55. | Safety | SAFE_L5 | Listing of all eCSSRS True Positives, with Corresponding Reasons and AE or SAE status | | All |
| 56. | Safety | SAFE_L6 | Listing of Subjects Who Became Pregnant During the Study | | All |
| 57. | Safety | SAFE_L7 | Patient Profiles for Subjects Meeting Protocol<br>Defined Liver Stopping Criteria | | All |
| 58. | Safety | SAFE_L7 | Patient Profiles for Subjects Meeting Confirmed Virologic Withdrawal Criteria | | All |
| 59. | Safety | SAFE_L7 | Patient Profiles for Subject Excluded from Safety Population Due to Non-Study Treatment Ongoing at Randomisation | | All |
| 60. | Safety | SAFE_L8 | Listing of Cardiovascular Events | | All |
| 61. | Safety | AE7 | Listing of Subject Numbers for Individual Adverse Events | | All |
| 62. | Safety | AE2 | Listing of Relationship Between Adverse Event<br>System Organ Classes, Preferred Terms, and<br>Verbatim Text | | All |
| 63. | Safety | LB14 | Listing of Laboratory Data with Character Results | | All |
| 64. | Safety | PAN12 | Listing of Subjects with an Adverse Event of Suspected, Probable, Confirmed for COVID-19 Infection | | All |

| Non-IC | H: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Statistical Display<br>Standard/ Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 65. | | | | Covered in 64 | |
| Hepato | biliary (Liver) | | | • | |
| 66. | Safety | MH2 | Listing of Medical Conditions for Subjects with Liver Stopping Events | | All |
| 67. | Safety | SU2 | Listing of Substance Use for Subjects with Liver Stopping Events | | All |
| 68. | Safety | PK07 | Listing of Plasma DTG Pharmacokinetic for Subjects with Liver Stopping Events | | All |
| Virolog | У | | | | 1 |
| 69. | CVW | VIR_L1 | Listing of All Genotypic Data – CVWs | | All |
| 70. | pPVW | VIR_L1 | Listing of All Genotypic Data – pPVWs | | All |
| 71. | CVW | VIR_L2 | Listing of Genotype by Genotypic Cut-Off – CVWs | | All |
| 72. | pPVW | VIR_L2 | Listing of Genotype by Genotypic Cut-Off – pPVWs | | All |
| 73. | CVW | VIR_L3 | Listing of All Phenotypic Data – CVWs | | All |
| 74. | pPVW | VIR_L3 | Listing of All Phenotypic Data – pPVWs | | All |
| 75. | CVW | VIR_L4 | Listing of Replication Capacity – CVWs | | All |
| 76. | pPVW | VIR_L4 | Listing of Replication Capacity – pPVWs | | All |

| Non-IC | H: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Statistical Display<br>Standard/ Example Shell | Title | Programming<br>Notes | Deliverable<br>[Priority] |
| 77. | CVW | VIR_L5 | Listing of Net Assessment Score – CVWs | | All |
| 78. | pPVW | VIR_L5 | Listing of Net Assessment Score – pPVWs | | All |
| 79. | CVW | VIR_L7 | Listing of Genotypic and Phenotypic Data for Subjects with Confirmed Virologic Withdrawal Criteria | | All |
| 80. | pPVW | VIR_L7 | Listing of Genotypic and Phenotypic Data for<br>Subjects with Potential Precautionary Virologic<br>Withdrawal Criteria | | All |
| 80.1 | ITT-E | VIR_L7 | Listing of Genotypic and Phenotypic Data for<br>Subjects Last on Study HIV-1 RNA >400 c/mL<br>with Resistance Testing | | Week 48 |
| 81. | pPVW | VF4 | Listing of Plasma HIV-1 RNA data and CD4+ cell count data for subjects with Potential Precautionary Virologic Withdrawal Criteria | | All |
| Health | Outcomes | | | | |
| 82. | ITT-E | LHO1 | Listing of HIV Treatment Satisfaction Questionnaire Scores (HIVTSQ) | | All |
| 83. | ITT-E | LHO2 | Listing of Symptom Distress Module Outcome | | All |
| 84. | ITT-E | LHO3 | Listing of Willingness to Switch | | All |

| Non-IC | Non-ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Statistical Display<br>Standard/ Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Impact | Impact of COVID-19 Pandemic | | | | |
| 85. | ITT-E | PAN7 | Listing of All Subjects with Visits and Assessments Impacted by COVID-19 Pandemic | | |
| 86. | Screened | PAN5 | Listing of Country Level Start Dates of COVID-19 Pandemic Measures | | |

# **15.18.** Appendix 18: Example Mock Shells for Data Displays Available Upon Request.

## Signature Page for $\,208090$ TMF-15022019 v1.0 $\,$

| Reason for signing: Approved | Name: PPD |
|---|---|
| | Role: A |
| | Date of signature: 29-Sep-2022 16:35:55 GMT+0000 |

Signature Page for TMF-15022019 v1.0